CLINICAL TRIAL: NCT03816891
Title: A Phase 2a/b, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy, Safety, Tolerability and Pharmacokinetics of KPL-716 in Reducing Pruritus in Subjects With Prurigo Nodularis
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of Vixarelimab in Reducing Pruritus in Prurigo Nodularis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Kiniksa Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPL-716-C201; GS45044 (Other: Genentech, Inc.)
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Prurigo Nodularis; Pruritis
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Intervention Model Description: Phase 2a: 2 arms; Phase 2b: 5 arms (4 arms during Double Blind Period and 1 arm during Open Label Extension)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 2a - Vixarelimab 360 mg SC Weekly (QW) (Experimental): Vixarelimab 720 mg loading dose followed by 360 mg weekly for 8 weeks (Protocol Version 3) or 16 weeks (Protocol Version 2)
  Interventions: Drug: Vixarelimab
- Phase 2a - Placebo SC QW (Placebo Comparator): Placebo loading dose followed by placebo weekly for 8 weeks (Protocol Version 3) or 16 weeks (Protocol Version 2)
  Interventions: Drug: Placebo
- Phase 2b - Vixarelimab 540 mg SC Every 4 Weeks (Q4W; DBL) (Experimental): Vixarelimab 540 mg SC, every 4 weeks (Q4W) for 16 weeks during Double Blind Period
  Interventions: Drug: Vixarelimab
- Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) (Experimental): Vixarelimab 360 mg SC, every 4 weeks (Q4W) for 16 weeks during Double Blind Period
  Interventions: Drug: Vixarelimab
- Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) (Experimental): Vixarelimab 120 mg SC, every 4 weeks (Q4W) for 16 weeks during Double Blind Period
  Interventions: Drug: Vixarelimab
- Phase 2b - Placebo SC, Q4W (DBL) (Placebo Comparator): Placebo SC, every 4 weeks (Q4W) for 16 weeks during Double Blind Period
  Interventions: Drug: Placebo
- Phase 2b - Vixarelimab 360 mg SC, Every 2 Weeks (Q2W; OLE) (Experimental): Vixarelimab 360 mg SC, every 2 weeks for 36 weeks during Open Label Extension
  Interventions: Drug: Vixarelimab

INTERVENTIONS:
Drug: Vixarelimab — solution for injection
  Other Names: KPL-716; RG6536
  Arms: Phase 2a - Vixarelimab 360 mg SC Weekly (QW); Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL); Phase 2b - Vixarelimab 360 mg SC, Every 2 Weeks (Q2W; OLE); Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL); Phase 2b - Vixarelimab 540 mg SC Every 4 Weeks (Q4W; DBL)
Drug: Placebo — solution for injection
  Arms: Phase 2a - Placebo SC QW; Phase 2b - Placebo SC, Q4W (DBL)

SUMMARY:
Study of the efficacy, safety, tolerability, pharmacokinetics (PK), and immunogenicity of Vixarelimab (KPL-716) in subjects with prurigo nodularis (PN).

DETAILED DESCRIPTION:
This is a Phase 2a/b randomized, double-blind, placebo-controlled study to investigate the efficacy, safety, tolerability, PK and immunogenicity of Vixarelimab administered subcutaneously (SC) in subjects with prurigo nodularis experiencing pruritus.

Phase 2a portion:

Forty-nine subjects with moderate to severe PN experiencing moderate to severe pruritus are treated in the Phase 2a portion of the study. At Baseline, subjects are randomized 1:1 to receive double-blind (DBL) vixarelimab or placebo: vixarelimab 720 mg loading dose followed by 360 mg every week; placebo loading dose followed by placebo every week. The treatment period is 8 weeks or 16 weeks (treatment duration was reduced from 16 weeks to 8 weeks in a protocol amendment [Protocol Version 3]).

Phase 2b portion:

The Phase 2b study consists of a 4-week Screening Period and a 16-week Double-Blind Period, followed by a 36-week Open-Label-Extension (OLE) Period. Approximately 180 subjects with PN, experiencing severe pruritus, are randomized (at 1:1:1:1 ratio) into one of 4 arms (3 active arms and one placebo arm). A total of 4 doses of study drug are administered during the Double-Blind Period to measure the efficacy, safety, and PK of Vixarelimab. After the Double-Blind Period, all subjects have the option to receive vixarelimab during the OLE Period to evaluate the long-term safety and PK.

ELIGIBILITY:
Inclusion Criteria (apply to both Phase 2a and Phase 2b unless otherwise specified):

1. Male or female aged 18 to 75 years (Phase 2a), 18 to 80 years (Phase 2b)
2. Have clinical diagnosis of prurigo nodularis for at least 6 months
3. Have at least 10 nodules (Phase 2a), 20 nodules (Phase 2b) at the Screening Visit and Day 1
4. Moderate to severe pruritus (Phase 2a); severe pruritus (Phase 2b)
5. Female subjects of childbearing potential must have a negative pregnancy test, be nonlactating, and having agreed to use a highly effective method of contraception, as specified in the protocol, from the Screening Visit until 16 weeks after final study drug administration
6. Able to comprehend and willing to sign an Informed Consent Form and able to abide by the study restrictions and comply with all study procedures for the duration of the study

Exclusion Criteria (apply to both Phase 2a and Phase 2b unless otherwise specified):

1. Use of prohibited medications within the indicated timeframe from Day 1
2. Is currently using medication known to cause pruritus
3. Presence of any inflammatory, pruritic, and/or fibrotic skin condition other than moderate to severe prurigo nodularis or atopic dermatitis unless approved by the Sponsor
4. Laboratory abnormalities that fall outside the windows specified in the protocol at the Screening Visit
5. Has an active infection, including skin infection
6. Any medical or psychiatric condition which, in the opinion of the Investigator or the Sponsor, may place the subject at increased risk as a result of study participation, interfere with study participation or study assessments, affect compliance with study requirements, or complicate interpretation of study results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (86):
- United States (40):
  - Arizona Research Center, Phoenix, Arizona
  - Investigate MD, LLC, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Wallace Medical Group, Inc., Los Angeles, California
  - Velocity Clinical Research - North Hollywood, North Hollywood, California
  - Colorado Center for Dermatology, PLLC, Centennial, Colorado
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Rybear, Inc., Fort Lauderdale, Florida
  - University of Florida, Department of Dermatology, Gainesville, Florida
  - Olympian Clinical Research, Largo, Florida
  - University of Miami Itch Center, Miami, Florida
  - Riverchase Dermatology, Pembroke Pines, Florida
  - Olympian Clinical Research, St. Petersburg, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - Palm Harbor Dermatology, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - Integrated Clinical Research, West Palm Beach, Florida
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - DS Research, New Albany, Indiana
  - DS Research, Louisville, Kentucky
  - ALLCUTIS Research, LLC, Beverly, Massachusetts
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Skin Specialists, PC, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Bobby Buka MD, PC, New York, New York
  - University of Rochester Dermatology at College Town, Rochester, New York
  - Wright State Physicians, Fairborn, Ohio
  - Paddington Testing Co., Inc., Philadelphia, Pennsylvania
  - Medical University of South Carolina, Department of Dermatology and Dermatological Surgery, Charleston, South Carolina
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Dermatology Specialists of Spokane, Spokane, Washington
- Australia (4):
  - Premier Specialists Pty Ltd, Kogarah, New South Wales
  - St. George Dermatology & Skin Cancer Centre, Kogarah, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - The Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Medical University of Graz, Graz
  - Medical University of Vienna, Vienna
- Belgium (2):
  - Cliniques Universitaires Saint-Luc (UCL St-Luc), Brussels
  - CHU de Liège, Liège
- Canada (8):
  - Stratica Medical, Edmonton, Alberta
  - Alberta DermaSurgery Centre, Edmonton, Alberta
  - Central Alberta Research Clinic (CARe Clinic), Red Deer, Alberta
  - Brunswick Dermatology Center, Fredericton, New Brunswick
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Drc Angélique Gagné-Henley MD Inc., Saint-Jérôme, Quebec
- Czechia (2):
  - CCR Czech a.s., Pardubice
  - CLINTRIAL s.r.o., Prague
- France (3):
  - Hôpital Saint André - CHU de Bordeaux, Bordeaux
  - Hôpital Morvan - CHU Brest, Brest
  - CHU Nantes - Service de Dermatologie, Nantes
- Germany (8):
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Klinikum Bielefeld Rosenhöhe, Bielefeld, North Rhine-Westphalia
  - University Hospital Dresden, Dresden
  - Studienzentrale Entzündliche Hauterkrankungen, Erlangen
  - George-August-Universität Göttingen, Göttingen
  - University Hospital Muenster, Department of Dermatology, Münster
  - Eberhard-Karls-University, Tübingen
  - Hautarztpraxis Dr. Hoffmann, Witten
- Italy (2):
  - A.O.U. Policlinico Vittorio Emanuele, Catania, Sicily
  - Asst Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
- Poland (3):
  - Grażyna Pulka Centrum Medyczne All-Med, Krakow
  - Kliniczny Szpital Wojewódzki Nr 1 im. Fryderyka Chopina w Rzeszowie, Klinika Dermatologii, Rzeszów
  - Kyclinic Przychodnia Lekarsko-Psychologiczna Matusiak Spółka Partnerska, Wroclaw
- South Korea (4):
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Taiwan (4):
  - Taipei Medical University Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan
- United Kingdom (4):
  - Royal Infirmary of Edinburgh at Little France, Edinburgh
  - Barts Health NHS Trust, Whipps Cross Hospital, Leytonstone
  - Broadgreen Hospital, Liverpool
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stander S, Yosipovitch G, Sofen H, Abramzon D, Galanter J, Wang S, Paolini JF. Vixarelimab in Patients With Prurigo Nodularis: A Randomized Clinical Trial. JAMA Dermatol. 2025 Dec 17:e254950. doi: 10.1001/jamadermatol.2025.4950. Online ahead of print. PMID 41405882
- [Derived] Ma DX, Neerumalla S, Baird A, Whitehead RA, Filip P, Tajudeen BA, Batra PS, Papagiannopoulos P. Impact of Obesity on the Structured Histopathology of Chronic Rhinosinusitis Patients. Laryngoscope. 2025 Oct 6. doi: 10.1002/lary.70177. Online ahead of print. PMID 41051123
- [Derived] Sofen H, Bissonnette R, Yosipovitch G, Silverberg JI, Tyring S, Loo WJ, Zook M, Lee M, Zou L, Jiang GL, Paolini JF. Efficacy and safety of vixarelimab, a human monoclonal oncostatin M receptor beta antibody, in moderate-to-severe prurigo nodularis: a randomised, double-blind, placebo-controlled, phase 2a study. EClinicalMedicine. 2023 Feb 3;57:101826. doi: 10.1016/j.eclinm.2023.101826. eCollection 2023 Mar. PMID 36816342

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized 1:1 to receive vixarelimab or placebo in Phase 2a. In Phase 2b, participants were randomized 1:1:1:1:1 to receive 4 different dosing regimens of vixarelimab or placebo in a 16-week Double-Blind Period followed by a 36-week Open-Label-Extension (OLE) Period.
Groups:
- Phase 2a - Vixarelimab 360 mg SC QW: Vixarelimab 720 mg loading dose followed by 360 mg subcutaneously (SC) weekly (QW) for 8 weeks (Protocol Version 3) or 16 weeks (Protocol Version 2).
- Phase 2a - Placebo SC QW: Placebo loading dose followed by placebo SC QW for 8 weeks (Protocol Version 3) or 16 weeks (Protocol Version 2).
- Phase 2b - Vixarelimab 540 mg SC Q4W (DBL): Vixarelimab 540 mg SC, every 4 weeks (Q4W) for 16 weeks during the double blind (DBL) period. Vixarelimab 360 mg SC, every 2 weeks for 36 weeks during open label extension (OLE).
- Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL): Vixarelimab 360 mg SC, Q4W for 16 weeks during the double blind (DBL) period. Vixarelimab 360 mg SC, every 2 weeks for 36 weeks during open label extension (OLE).
- Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL): Vixarelimab 120 mg SC, Q4W for 16 weeks during double blind (DBL) period. Vixarelimab 360 mg SC, every 2 weeks for 36 weeks during open label extension (OLE).
- Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE): Placebo SC, Q4W for 16 weeks during double blind (DBL) period. Vixarelimab 360 mg SC, every 2 weeks for 36 weeks during open label extension (OLE).
Period: Double-Blind Period
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Started (Randomized) | 24 | 26 | 47 | 47 | 47 | 49
Randomized and Treated | 23 | 26 | 47 | 47 | 47 | 48
Completed Treatment | 23 | 23 | 45 | 44 | 47 | 47
Completed | 20 | 24 | 45 | 44 | 47 | 47
Not Completed | 4 | 2 | 2 | 3 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Coronavirus Disease (COVID-19) | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Period (Phase 2b Only)
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Started (Entered Phase 2b Open-Label Period) | 0 | 0 | 45 | 43 | 47 | 46
Completed Treatment | 0 | 0 | 38 | 38 | 38 | 43
Completed | 0 | 0 | 38 | 38 | 39 | 43
Not Completed | 0 | 0 | 7 | 5 | 8 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 3 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 2 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (mITT) Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE) | Total
Number analyzed (Participants) | 23 | 26 | 47 | 47 | 47 | 48 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Phase 2a and Phase 2b populations were analyzed separately.
  years
    Phase 2a: number analyzed (Participants) | 23 | 26 | 0 | 0 | 0 | 0 | 49
    Phase 2a | 52.0 (15.56) | 64.1 (7.86) |  |  |  |  | 58.4 (13.41)
    Phase 2b: number analyzed (Participants) | 0 | 0 | 47 | 47 | 47 | 48 | 189
    Phase 2b |  |  | 56.7 (12.18) | 55.9 (13.73) | 54.4 (16.11) | 54.8 (13.35) | 55.4 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Phase 2a and Phase 2b populations were analyzed separately.
  Participants
    Phase 2a: number analyzed (Participants) | 23 | 26 | 0 | 0 | 0 | 0 | 49
    Phase 2a: Female | 13 | 16 |  |  |  |  | 29
    Phase 2a: Male | 10 | 10 |  |  |  |  | 20
    Phase 2b: number analyzed (Participants) | 0 | 0 | 47 | 47 | 47 | 48 | 189
    Phase 2b: Female |  |  | 29 | 28 | 28 | 29 | 114
    Phase 2b: Male |  |  | 18 | 19 | 19 | 19 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Phase 2a and Phase 2b populations were analyzed separately.
  Participants
    Phase 2a: number analyzed (Participants) | 23 | 26 | 0 | 0 | 0 | 0 | 49
    Phase 2a: Hispanic or Latino | 2 | 0 |  |  |  |  | 2
    Phase 2a: Not Hispanic or Latino | 21 | 26 |  |  |  |  | 47
    Phase 2a: Unknown or Not Reported | 0 | 0 |  |  |  |  | 0
    Phase 2b: number analyzed (Participants) | 0 | 0 | 47 | 47 | 47 | 48 | 189
    Phase 2b: Hispanic or Latino |  |  | 0 | 5 | 4 | 3 | 12
    Phase 2b: Not Hispanic or Latino |  |  | 47 | 42 | 43 | 45 | 177
    Phase 2b: Unknown or Not Reported |  |  | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Phase 2a and Phase 2b populations were analyzed separately.
  Participants
    Phase 2a: number analyzed (Participants) | 23 | 26 | 0 | 0 | 0 | 0 | 49
    Phase 2a: American Indian or Alaska Native | 0 | 1 |  |  |  |  | 1
    Phase 2a: Asian | 2 | 0 |  |  |  |  | 2
    Phase 2a: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  |  | 0
    Phase 2a: Black or African American | 5 | 3 |  |  |  |  | 8
    Phase 2a: White | 15 | 21 |  |  |  |  | 36
    Phase 2a: More than one race | 1 | 0 |  |  |  |  | 1
    Phase 2a: Unknown or Not Reported | 0 | 1 |  |  |  |  | 1
    Phase 2b: number analyzed (Participants) | 0 | 0 | 47 | 47 | 47 | 48 | 189
    Phase 2b: American Indian or Alaska Native |  |  | 0 | 1 | 1 | 2 | 4
    Phase 2b: Asian |  |  | 9 | 11 | 3 | 11 | 34
    Phase 2b: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0 | 0 | 0
    Phase 2b: Black or African American |  |  | 3 | 5 | 8 | 6 | 22
    Phase 2b: White |  |  | 31 | 27 | 34 | 29 | 121
    Phase 2b: More than one race |  |  | 1 | 1 | 0 | 0 | 2
    Phase 2b: Unknown or Not Reported |  |  | 3 | 2 | 1 | 0 | 6
Weekly Average Worst Itch-Numeric Rating Scale (WI-NRS) Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — Participants rated pruritus daily on Worst Itch [pruritis]-Numeric Rating Scale (WI-NRS: 0=no pruritus; 10=worst imaginable pruritus) at baseline (from Day -6 to Day 1 of the study). Population: The Phase 2a and Phase 2b populations were analyzed separately.
  score on a scale
    Phase 2a: number analyzed (Participants) | 23 | 26 | 0 | 0 | 0 | 0 | 49
    Phase 2a | 8.7 (0.88) | 8.0 (1.09) |  |  |  |  | 8.3 (1.05)
    Phase 2b: number analyzed (Participants) | 0 | 0 | 47 | 47 | 47 | 48 | 189
    Phase 2b |  |  | 8.4 (0.93) | 8.7 (0.91) | 8.4 (1.17) | 8.6 (0.89) | 8.5 (0.98)

OUTCOME MEASURES:

1. Primary Outcome: Phase 2a & 2b: Percent Change From Baseline in Weekly Average Worst Itch-Numeric Rating Scale (WI-NRS) Score
Description: Participants rated pruritus daily on the Worst Itch [pruritis] Numeric Rating Scale (WI-NRS: 0=no pruritus; 10=worst imaginable pruritus). The least squares mean (LSM) and LSM difference were rounded up or down to the nearest single decimal place.
Time Frame: at Week 8 (Phase 2a); at Week 16 (Phase 2b)
Population: Modified Intent to Treat (mITT) Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period. Part 2a: Last Observation Carried Forward (LOCF); Part 2b: Multiple imputation (WI)
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 23 | 26 | 47 | 47 | 47 | 48
percentage change | -50.6 (6.99) | -29.4 (6.80) | -56.2 (4.84) | -51.0 (4.83) | -33.0 (4.86) | -14.5 (4.76)
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Test type: Superiority; p = 0.0347, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -21.2, 95% CI 2-sided [-40.82 to -1.60], Standard Error of Mean 9.73
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p < 0.0001, ANCOVA — Estimated from ANCOVA model with treatment and randomization stratification factors of sex and years since the first nodule observed (i.e., ≥10 vs. <10 years) as fixed effect factors, baseline as covariate; LS Mean Difference = -41.7, 95% CI 2-sided [-54.9 to -28.5], Standard Error of Mean 6.73
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -36.4, 95% CI 2-sided [-49.6 to 23.3], Standard Error of Mean 6.70
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p = 0.0061, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -18.4, 95% CI 2-sided [-31.6 to -5.3], Standard Error of Mean 6.72

2. Secondary Outcome: Phase 2a: Percentage of Participants Achieving at Least a 4-point Reduction From Baseline in Weekly Average WI-NRS at Week 8
Description: Participants rated pruritus daily on the Worst Itch [pruritis]-Numeric Rating Scale (WI-NRS; 0=no pruritus; 10=worst imaginable pruritus).
Time Frame: Baseline, Week 8
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period; LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage of participants | 52.2 [30.6 to 73.2] | 30.8 [14.3 to 51.8]
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Test type: Superiority; p = 0.1093, Cochran-Mantel-Haenszel — Calculated from Cochran-Mantel-Haenszel (CMH) test with sex and atopy as stratification factors and placebo as reference within corresponding cohort; Odds Ratio (OR) = 2.76, 95% CI 2-sided [0.81 to 9.44]

3. Secondary Outcome: Phase 2a: Percent Change From Baseline in Pruritus Visual Analog Scale (VAS) at Week 8
Description: At every visit, participants rated the intensity of their average pruritus over previous 3 days on VAS 0-10 line scale (0=no pruritis, 10=worst imaginable pruritis)
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage change | -54.4 (7.03) | -32.6 (6.96)
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Test type: Superiority; p = 0.0325, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -21.8, 95% CI 2-sided [-41.62 to -1.90], Standard Error of Mean 9.86

4. Secondary Outcome: Phase 2a: Change From Baseline in Weekly Average of WI-NRS Over Time
Description: as for outcome 2
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period. Baseline through Week 16: LOCF; Weeks 17-24: participants with an assessment at given time point.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
score on a scale
  Week 1 | -1.6 (0.36) | -0.8 (0.29)
  Week 2 | -2.4 (0.47) | -1.3 (0.30)
  Week 3 | -2.9 (0.52) | -1.9 (0.37)
  Week 4 | -3.7 (0.62) | -2.3 (0.42)
  Week 5 | -4.2 (0.66) | -2.6 (0.39)
  Week 6 | -4.3 (0.64) | -2.6 (0.37)
  Week 7 | -4.5 (0.68) | -2.8 (0.44)
  Week 8 | -4.5 (0.68) | -2.7 (0.43)
  Week 9 | -4.2 (0.65) | -2.8 (0.41)
  Week 10 | -4.2 (0.62) | -2.9 (0.41)
  Week 11 | -4.0 (0.65) | -3.2 (0.43)
  Week 12 | -3.9 (0.63) | -2.9 (0.41)
  Week 13 | -4.2 (0.67) | -2.8 (0.43)
  Week 14 | -4.4 (0.69) | -2.7 (0.45)
  Week 15 | -4.3 (0.69) | -2.9 (0.44)
  Week 16 | -4.3 (0.64) | -3.0 (0.42)
  Week 17: number analyzed (Participants) | 11 | 12
  Week 17 | -3.8 (1.04) | -3.1 (0.64)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -4.3 (1.05) | -3.2 (0.61)
  Week 19: number analyzed (Participants) | 10 | 12
  Week 19 | -4.4 (1.02) | -3.3 (0.62)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -4.3 (1.04) | -3.6 (0.69)
  Week 21: number analyzed (Participants) | 10 | 12
  Week 21 | -4.3 (1.03) | -3.4 (0.74)
  Week 22: number analyzed (Participants) | 10 | 12
  Week 22 | -4.4 (1.00) | -3.1 (0.66)
  Week 23: number analyzed (Participants) | 10 | 12
  Week 23 | -4.4 (1.04) | -3.1 (0.72)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -4.3 (1.03) | -2.9 (0.74)

5. Secondary Outcome: Phase 2a: Percent Change From Baseline in Weekly Average of WI-NRS Over Time
Description: Participants rated pruritus daily on the Worst Itch [pruritis]-Numeric Rating Scale (WI-NRS; 0=no pruritus; 10=worst imaginable pruritus). The least squares mean (LSM) and LSM difference were rounded up or down to the nearest single decimal place.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage change
  Week 1 | -20.2 (4.21) | -9.1 (4.09)
  Week 2 | -27.3 (5.00) | -13.9 (4.86)
  Week 3 | -33.6 (5.39) | -18.1 (5.24)
  Week 4 | -42.3 (6.27) | -22.8 (6.10)
  Week 5 | -46.6 (6.48) | -28.0 (6.29)
  Week 6 | -48.3 (6.27) | -27.9 (6.10)
  Week 7 | -50.5 (7.01) | -29.7 (6.81)
  Week 8 | -50.6 (6.99) | -29.4 (6.80)
  Week 9 | -47.0 (6.69) | -29.7 (6.50)
  Week 10 | -47.9 (6.42) | -30.8 (6.24)
  Week 11 | -44.8 (6.84) | -34.0 (6.65)
  Week 12 | -43.9 (6.59) | -29.9 (6.41)
  Week 13 | -46.3 (6.59) | -28.1 (6.41)
  Week 14 | -48.9 (6.97) | -27.6 (6.78)
  Week 15 | -48.8 (6.93) | -29.6 (6.74)
  Week 16 | -50.4 (6.43) | -31.3 (6.25)
  Week 17: number analyzed (Participants) | 11 | 12
  Week 17 | -47.0 (10.96) | -36.5 (10.40)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -50.9 (10.83) | -38.1 (9.84)
  Week 19: number analyzed (Participants) | 10 | 12
  Week 19 | -51.2 (10.51) | -39.6 (9.55)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -50.1 (10.76) | -43.9 (9.77)
  Week 21: number analyzed (Participants) | 10 | 26
  Week 21 | -50.2 (11.09) | -41.0 (10.07)
  Week 22: number analyzed (Participants) | 10 | 12
  Week 22 | -50.3 (10.52) | -38.0 (9.55)
  Week 23: number analyzed (Participants) | 10 | 12
  Week 23 | -51.7 (11.24) | -37.5 (10.21)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -51.8 (11.76) | -33.8 (10.68)
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 1; Test type: Superiority; p = 0.0657, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -11.1, 95% CI 2-sided [-22.85 to 0.75], Standard Error of Mean 5.85
Statistical Analysis 2: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 2; Test type: Superiority; p = 0.0595, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -13.5, 95% CI 2-sided [-27.48 to 0.56], Standard Error of Mean 6.96
Statistical Analysis 3: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 3; Test type: Superiority; p = 0.0455, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -15.4, 95% CI 2-sided [-30.55 to -0.33], Standard Error of Mean 7.50
Statistical Analysis 4: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 4; Test type: Superiority; p = 0.0305, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -19.5, 95% CI 2-sided [-37.11 to -1.93], Standard Error of Mean 8.73
Statistical Analysis 5: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 5; Test type: Superiority; p = 0.0456, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -18.5, 95% CI 2-sided [-36.69 to -0.38], Standard Error of Mean 9.01
Statistical Analysis 6: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 6; Test type: Superiority; p = 0.0236, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -20.5, 95% CI 2-sided [-38.06 to -2.88], Standard Error of Mean 8.73
Statistical Analysis 7: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 7; Test type: Superiority; p = 0.0385, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -20.8, 95% CI 2-sided [-40.45 to -1.15], Standard Error of Mean 9.75
Statistical Analysis 8: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 8; Test type: Superiority; p = 0.0347, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -21.2, 95% CI 2-sided [-40.82 to -1.60], Standard Error of Mean 9.73
Statistical Analysis 9: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 9; Test type: Superiority; p = 0.0694, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -17.3, 95% CI 2-sided [-36.06 to 1.44], Standard Error of Mean 9.30
Statistical Analysis 10: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 10; Test type: Superiority; p = 0.0621, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -17.1, 95% CI 2-sided [-35.08 to 0.90], Standard Error of Mean 8.93
Statistical Analysis 11: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 11; Test type: Superiority; p = 0.2619, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -10.8, 95% CI 2-sided [-30.0 to 8.37], Standard Error of Mean 9.52
Statistical Analysis 12: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 12; Test type: Superiority; p = 0.1344, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -14.0, 95% CI 2-sided [-32.48 to 4.50], Standard Error of Mean 9.17
Statistical Analysis 13: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 13; Test type: Superiority; p = 0.0533, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -18.2, 95% CI 2-sided [-36.71 to 0.27], Standard Error of Mean 9.17
Statistical Analysis 14: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 14; Test type: Superiority; p = 0.0335, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -21.3, 95% CI 2-sided [-40.82 to -1.74], Standard Error of Mean 9.70
Statistical Analysis 15: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 15; Test type: Superiority; p = 0.0536, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -19.1, 95% CI 2-sided [-38.58 to 0.31], Standard Error of Mean 9.65
Statistical Analysis 16: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 16; Test type: Superiority; p = 0.0388, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -19.1, 95% CI 2-sided [-37.11 to -1.03], Standard Error of Mean 8.95
Statistical Analysis 17: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 17; Test type: Superiority; p = 0.5181, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -10.5, 95% CI 2-sided [-43.94 to 22.95], Standard Error of Mean 15.92
Statistical Analysis 18: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 18; Test type: Superiority; p = 0.4142, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -12.8, 95% CI 2-sided [-45.08 to 19.47], Standard Error of Mean 15.30
Statistical Analysis 19: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 19; Test type: Superiority; p = 0.4450, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -11.6, 95% CI 2-sided [-42.94 to 19.72], Standard Error of Mean 14.85
Statistical Analysis 20: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 20; Test type: Superiority; p = 0.6897, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -6.2, 95% CI 2-sided [-38.23 to 25.89], Standard Error of Mean 15.20
Statistical Analysis 21: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 21; Test type: Superiority; p = 0.5636, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -9.2, 95% CI 2-sided [-42.25 to 23.81], Standard Error of Mean 15.66
Statistical Analysis 22: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 22; Test type: Superiority; p = 0.4190, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -12.3, 95% CI 2-sided [-43.64 to 19.04], Standard Error of Mean 14.85
Statistical Analysis 23: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 23; Test type: Superiority; p = 0.3818, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -14.3, 95% CI 2-sided [-47.76 to 19.24], Standard Error of Mean 15.88
Statistical Analysis 24: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 24; Test type: Superiority; p = 0.2957, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -17.9, 95% CI 2-sided [-52.97 to 17.13], Standard Error of Mean 16.61

6. Secondary Outcome: Phase 2a: Change From Baseline in Pruritis Visual Analog Scale (VAS) Over Time
Description: Participants rated intensity of their average pruritus over previous 3 days on VAS 0-10 line scale (0=no pruritis, 10=worst imaginable pruritis)
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 24
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period. Baseline through Week 8: LOCF; Weeks 9-24: participants with an assessment at given time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
units on a scale
  Week 1 | -1.9 (0.55) | -1.4 (0.33)
  Week 2 | -2.9 (0.62) | -1.8 (0.51)
  Week 3 | -3.5 (0.63) | -2.2 (0.52)
  Week 4 | -4.5 (0.72) | -3.3 (0.58)
  Week 5 | -4.5 (0.70) | -2.7 (0.50)
  Week 6 | -4.7 (0.75) | -2.9 (0.54)
  Week 7 | -5.0 (0.69) | -3.2 (0.56)
  Week 8 | -5.0 (0.72) | -3.0 (0.48)
  Week 9: number analyzed (Participants) | 10 | 14
  Week 9 | -4.3 (1.08) | -3.8 (0.61)
  Week 10: number analyzed (Participants) | 22 | 26
  Week 10 | -5.0 (0.71) | -3.7 (0.49)
  Week 11: number analyzed (Participants) | 10 | 14
  Week 11 | -4.7 (1.27) | -4.3 (0.58)
  Week 12: number analyzed (Participants) | 22 | 26
  Week 12 | -4.8 (0.66) | -3.8 (0.46)
  Week 13: number analyzed (Participants) | 10 | 14
  Week 13 | -4.6 (1.20) | -3.5 (0.64)
  Week 14: number analyzed (Participants) | 10 | 14
  Week 14 | -4.8 (1.10) | -3.7 (0.68)
  Week 15: number analyzed (Participants) | 10 | 14
  Week 15 | -4.5 (1.16) | -3.9 (0.69)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -5.1 (0.70) | -3.3 (0.50)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -4.8 (1.14) | -3.0 (0.67)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -4.6 (1.19) | -2.9 (0.74)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -4.9 (1.19) | -2.9 (0.80)

7. Secondary Outcome: Phase 2a: Percent Change From Baseline in Pruritis Visual Analog Scale (VAS) Over Time
Description: Participants rated intensity of their average pruritus over previous 3 days on VAS 0-10 line scale (0=no pruritis, 10=worst imaginable pruritis). The least squares mean (LSM) and LSM difference were rounded up or down to the nearest single decimal place.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage change
  Week 1 | -18.4 (5.45) | -15.8 (5.40)
  Week 2 | -28.2 (6.74) | -18.3 (6.67)
  Week 3 | -36.8 (6.53) | -19.2 (6.46)
  Week 4 | -48.9 (7.60) | -33.1 (7.52)
  Week 5 | -47.5 (6.88) | -27.9 (6.81)
  Week 6 | -50.0 (7.81) | -31.8 (7.73)
  Week 7 | -54.3 (7.41) | -33.6 (7.33)
  Week 8 | -54.4 (7.03) | -32.6 (6.96)
  Week 9: number analyzed (Participants) | 10 | 14
  Week 9 | -42.5 (9.51) | -47.2 (8.10)
  Week 10: number analyzed (Participants) | 22 | 26
  Week 10 | -54.0 (6.92) | -40.0 (6.71)
  Week 11: number analyzed (Participants) | 10 | 14
  Week 11 | -50.5 (10.59) | -51.2 (9.02)
  Week 12: number analyzed (Participants) | 22 | 26
  Week 12 | -53.4 (6.19) | -40.2 (6.00)
  Week 13: number analyzed (Participants) | 10 | 14
  Week 13 | -48.3 (10.88) | -43.0 (9.26)
  Week 14: number analyzed (Participants) | 10 | 14
  Week 14 | -50.4 (10.25) | -44.2 (8.73)
  Week 15: number analyzed (Participants) | 10 | 14
  Week 15 | -46.0 (10.66) | -47.6 (9.08)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -56.5 (6.70) | -35.6 (6.50)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -50.2 (11.56) | -39.3 (10.44)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -48.8 (12.47) | -37.1 (11.26)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -50.4 (12.32) | -36.6 (11.11)
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 1; Test type: Superiority; p = 0.7379, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -2.6, 95% CI 2-sided [-17.98 to 12.83], Standard Error of Mean 7.64
Statistical Analysis 2: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 2; Test type: Superiority; p = 0.3022, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -9.9, 95% CI 2-sided [-28.90 to 9.17], Standard Error of Mean 9.45
Statistical Analysis 3: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 3; Test type: Superiority; p = 0.0606, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -17.6, 95% CI 2-sided [-36.07 to 0.82], Standard Error of Mean 9.15
Statistical Analysis 4: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 4; Test type: Superiority; p = 0.1448, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -15.8, 95% CI 2-sided [-37.28 to 5.66], Standard Error of Mean 10.65
Statistical Analysis 5: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 5; Test type: Superiority; p = 0.0480, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -19.6, 95% CI 2-sided [-39.06 to -0.18], Standard Error of Mean 9.65
Statistical Analysis 6: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 6; Test type: Superiority; p = 0.1032, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -18.2, 95% CI 2-sided [-40.30 to 3.85], Standard Error of Mean 10.95
Statistical Analysis 7: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 7; Test type: Superiority; p = 0.0523, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -20.7, 95% CI 2-sided [-41.66 to 0.22], Standard Error of Mean 10.39
Statistical Analysis 8: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 8; Test type: Superiority; p = 0.0325, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -21.8, 95% CI 2-sided [-41.62 to -1.90], Standard Error of Mean 9.86
Statistical Analysis 9: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 9; Test type: Superiority; p = 0.7274, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = 4.6, 95% CI 2-sided [-22.83 to 32.12], Standard Error of Mean 13.13
Statistical Analysis 10: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 10; Test type: Superiority; p = 0.1523, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -14.0, 95% CI 2-sided [-33.47 to 5.39], Standard Error of Mean 9.63
Statistical Analysis 11: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 11; Test type: Superiority; p = 0.9649, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = 0.7, 95% CI 2-sided [-29.93 to 31.24], Standard Error of Mean 14.61
Statistical Analysis 12: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 12; Test type: Superiority; p = 0.1351, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -13.1, 95% CI 2-sided [-30.48 to 4.25], Standard Error of Mean 8.61
Statistical Analysis 13: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 13; Test type: Superiority; p = 0.7258, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -5.3, 95% CI 2-sided [-36.75 to 26.07], Standard Error of Mean 15.01
Statistical Analysis 14: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 14; Test type: Superiority; p = 0.6646, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -6.2, 95% CI 2-sided [-35.81 to 23.36], Standard Error of Mean 14.14
Statistical Analysis 15: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 15; Test type: Superiority; p = 0.9151, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = 1.6, 95% CI 2-sided [-29.20 to 32.38], Standard Error of Mean 14.71
Statistical Analysis 16: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 16; Test type: Superiority; p = 0.0304, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -20.9, 95% CI 2-sided [-39.66 to -2.07], Standard Error of Mean 9.32
Statistical Analysis 17: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 18; Test type: Superiority; p = 0.5209, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -10.9, 95% CI 2-sided [-45.96 to 24.17], Standard Error of Mean 16.62
Statistical Analysis 18: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 20; Test type: Superiority; p = 0.5254, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -11.6, 95% CI 2-sided [-49.46 to 26.20], Standard Error of Mean 17.93
Statistical Analysis 19: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 24; Test type: Superiority; p = 0.4458, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -13.8, 95% CI 2-sided [-51.16 to 23.53], Standard Error of Mean 17.70

8. Secondary Outcome: Phase 2a: Change From Baseline in 5-D Pruritus Total Score Over Time
Description: Administered every 2 visits, the 5-D Pruritus Scale evaluates pruritus in 5 domains: duration, degree, direction, disability and distribution. The scores from each domain are added together to obtain a total 5-D score ranging from 5 (no pruritus) to 25 (most severe pruritus).
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period. Baseline through Week 8: LOCF; Weeks 10-24: participants with an assessment at given time point.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
score on a scale
  Week 2 | -5.8 (0.95) | -2.7 (0.57)
  Week 4 | -6.7 (1.12) | -3.9 (0.76)
  Week 6 | -7.2 (1.09) | -4.2 (0.76)
  Week 8 | -7.7 (1.17) | -4.3 (0.78)
  Week 10: number analyzed (Participants) | 22 | 26
  Week 10 | -7.7 (1.18) | -5.0 (0.77)
  Week 12: number analyzed (Participants) | 22 | 26
  Week 12 | -7.4 (1.16) | -4.8 (0.83)
  Week 14: number analyzed (Participants) | 10 | 14
  Week 14 | -7.1 (1.72) | -4.7 (1.13)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -7.5 (1.26) | -4.6 (0.72)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -6.8 (1.60) | -3.4 (1.42)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -6.8 (1.67) | -3.5 (1.40)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -7.9 (1.82) | -3.7 (1.57)

9. Secondary Outcome: Phase 2a: Percent Change From Baseline in 5-D Pruritus Total Score Over Time
Description: Administered every 2 visits, the 5-D Pruritus Scale evaluates pruritus in five domains: duration, degree, direction, disability and distribution. The scores from each domain are added together to obtain a total 5-D score ranging from 5 (no pruritus) to 25 (most severe pruritus). The least squares mean (LSM) and LSM difference were rounded up or down to the nearest single decimal place.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage change
  Week 2 | -26.8 (3.83) | -13.3 (3.75)
  Week 4 | -31.8 (4.83) | -21.7 (4.74)
  Week 6 | -34.2 (4.65) | -23.6 (4.56)
  Week 8 | -36.8 (5.04) | -24.2 (4.95)
  Week 10: number analyzed (Participants) | 22 | 26
  Week 10 | -36.2 (4.69) | -26.4 (4.52)
  Week 12: number analyzed (Participants) | 22 | 26
  Week 12 | -33.7 (4.90) | -25.0 (4.71)
  Week 14: number analyzed (Participants) | 10 | 14
  Week 14 | -35.1 (7.28) | -26.0 (6.21)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -35.0 (4.66) | -24.5 (4.49)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -30.5 (7.71) | -18.1 (7.08)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -34.1 (8.05) | -19.4 (7.39)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -36.6 (8.92) | -20.5 (8.19)
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 2; Test type: Superiority; p = 0.0149, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -13.5, 95% CI 2-sided [-24.22 to -2.76], Standard Error of Mean 5.33
Statistical Analysis 2: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 4; Test type: Superiority; p = 0.1399, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -10.1, 95% CI 2-sided [-23.67 to 3.44], Standard Error of Mean 6.73
Statistical Analysis 3: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 6; Test type: Superiority; p = 0.1078, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -10.6, 95% CI 2-sided [-23.68 to 2.42], Standard Error of Mean 6.47
Statistical Analysis 4: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 8; Test type: Superiority; p = 0.0798, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -12.6, 95% CI 2-sided [-26.72 to 1.56], Standard Error of Mean 7.02
Statistical Analysis 5: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 10; Test type: Superiority; p = 0.1405, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -9.7, 95% CI 2-sided [-22.83 to 3.34], Standard Error of Mean 6.49
Statistical Analysis 6: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 12; Test type: Superiority; p = 0.2026, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -8.8, 95% CI 2-sided [-22.43 to 4.90], Standard Error of Mean 6.77
Statistical Analysis 7: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 14; Test type: Superiority; p = 0.3646, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -9.1, 95% CI 2-sided [-29.52 to 11.37], Standard Error of Mean 9.77
Statistical Analysis 8: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 16; Test type: Superiority; p = 0.1106, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -10.5, 95% CI 2-sided [-23.52 to 2.50], Standard Error of Mean 6.45
Statistical Analysis 9: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 18; Test type: Superiority; p = 0.2623, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -12.5, 95% CI 2-sided [-35.11 to 10.20], Standard Error of Mean 10.74
Statistical Analysis 10: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 20; Test type: Superiority; p = 0.2095, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -14.6, 95% CI 2-sided [-38.27 to 9.03], Standard Error of Mean 11.21
Statistical Analysis 11: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 24; Test type: Superiority; p = 0.2127, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -16.1, 95% CI 2-sided [-42.30 to 10.13], Standard Error of Mean 12.43

10. Secondary Outcome: Phase 2a: Percentage of Participants Achieving at Least a 4-point Reduction From Baseline in Weekly Average WI-NRS Over Time
Description: as for outcome 2
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period; Baseline through Week 16: LOCF; Weeks 17-24: participants with an assessment at given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage of participants
  Week 1 | 17.4 [5.0 to 38.8] | 7.7 [0.9 to 25.1]
  Week 2 | 26.1 [10.2 to 48.4] | 7.7 [0.9 to 25.1]
  Week 3 | 39.1 [19.7 to 61.5] | 11.5 [2.4 to 30.2]
  Week 4 | 52.2 [30.6 to 73.2] | 23.1 [9.0 to 43.6]
  Week 5 | 52.2 [30.6 to 73.2] | 23.1 [9.0 to 43.6]
  Week 6 | 52.2 [30.6 to 73.2] | 26.9 [11.6 to 47.8]
  Week 7 | 52.2 [30.6 to 73.2] | 34.6 [17.2 to 55.7]
  Week 8 | 52.2 [30.6 to 73.2] | 30.8 [14.3 to 51.8]
  Week 9 | 52.2 [30.6 to 73.2] | 30.8 [14.3 to 51.8]
  Week 10 | 47.8 [26.8 to 69.4] | 34.6 [17.2 to 55.7]
  Week 11 | 47.8 [26.8 to 69.4] | 34.6 [17.2 to 55.7]
  Week 12 | 47.8 [26.8 to 69.4] | 34.6 [17.2 to 55.7]
  Week 13 | 52.2 [30.6 to 73.2] | 26.9 [11.6 to 47.8]
  Week 14 | 52.2 [30.6 to 73.2] | 30.8 [14.3 to 51.8]
  Week 15 | 52.2 [30.6 to 73.2] | 30.8 [14.3 to 51.8]
  Week 16 | 52.2 [30.6 to 73.2] | 42.3 [23.4 to 63.1]
  Week 17: number analyzed (Participants) | 11 | 12
  Week 17 | 36.4 [10.9 to 69.2] | 41.7 [15.2 to 72.3]
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | 50.0 [18.7 to 81.3] | 33.3 [9.9 to 65.1]
  Week 19: number analyzed (Participants) | 10 | 12
  Week 19 | 60.0 [26.2 to 87.8] | 33.3 [9.9 to 65.1]
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | 60.0 [26.2 to 87.8] | 41.7 [15.2 to 72.3]
  Week 21: number analyzed (Participants) | 10 | 12
  Week 21 | 60.0 [26.2 to 87.8] | 50.0 [21.1 to 78.9]
  Week 22: number analyzed (Participants) | 10 | 12
  Week 22 | 50.0 [18.7 to 81.3] | 25.0 [5.5 to 57.2]
  Week 23: number analyzed (Participants) | 10 | 12
  Week 23 | 60.0 [26.2 to 87.8] | 33.3 [9.9 to 65.1]
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | 60.0 [26.2 to 87.8] | 41.7 [15.2 to 72.3]
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 1; Test type: Superiority; p = 0.2474, Cochran-Mantel-Haenszel — Calculated from CMH test with sex and atopy as stratification factors and placebo as reference within corresponding cohort; Odds Ratio (OR) = 2.96, 95% CI 2-sided [0.43 to 20.56]
Statistical Analysis 2: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 2; Test type: Superiority; p = 0.0687, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 4.49, 95% CI 2-sided [0.83 to 24.27]
Statistical Analysis 3: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 3; Test type: Superiority; p = 0.0145, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 6.89, 95% CI 2-sided [1.38 to 34.48]
Statistical Analysis 4: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 4; Test type: Superiority; p = 0.0235, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 4.85, 95% CI 2-sided [1.24 to 18.89]
Statistical Analysis 5: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 5; Test type: Superiority; p = 0.0334, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 3.81, 95% CI 2-sided [1.09 to 13.26]
Statistical Analysis 6: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 6; Test type: Superiority; p = 0.0618, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 3.27, 95% CI 2-sided [0.95 to 11.32]
Statistical Analysis 7: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 7; Test type: Superiority; p = 0.1748, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.38, 95% CI 2-sided [0.70 to 8.15]
Statistical Analysis 8: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 8; Test type: Superiority; p = 0.1093, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [0.81 to 9.44]
Statistical Analysis 9: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 9; Test type: Superiority; p = 0.1093, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [0.81 to 9.44]
Statistical Analysis 10: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 10; Test type: Superiority; p = 0.2610, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.60 to 6.80]
Statistical Analysis 11: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 11; Test type: Superiority; p = 0.2867, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.59 to 5.71]
Statistical Analysis 12: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 12; Test type: Superiority; p = 0.2874, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.59 to 6.01]
Statistical Analysis 13: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 13; Test type: Superiority; p = 0.0527, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 3.07, 95% CI 2-sided [0.94 to 10.05]
Statistical Analysis 14: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 14; Test type: Superiority; p = 0.0936, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.67, 95% CI 2-sided [0.82 to 8.73]
Statistical Analysis 15: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 15; Test type: Superiority; p = 0.0830, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.92, 95% CI 2-sided [0.84 to 10.21]
Statistical Analysis 16: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 16; Test type: Superiority; p = 0.3786, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.53 to 5.33]
Statistical Analysis 17: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 17; Test type: Superiority; p = 0.6949, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.12 to 3.99]
Statistical Analysis 18: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 18; Test type: Superiority; p = 0.5288, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.31 to 10.66]
Statistical Analysis 19: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 19; Test type: Superiority; p = 0.2613, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 3.18, 95% CI 2-sided [0.43 to 23.37]
Statistical Analysis 20: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 20; Test type: Superiority; p = 0.4208, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.34 to 14.81]
Statistical Analysis 21: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 21; Test type: Superiority; p = 0.7884, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.20 to 8.76]
Statistical Analysis 22: Comparison: Phase 2a - Vixarelimab 360 mg SC QW; Week 22; Test type: Superiority; p = 0.2982, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.68, 95% CI 2-sided [0.45 to 16.04]
Statistical Analysis 23: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 23; Test type: Superiority; p = 0.2613, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 3.18, 95% CI 2-sided [0.43 to 23.37]
Statistical Analysis 24: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 24; Test type: Superiority; p = 0.4208, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.34 to 14.81]

11. Secondary Outcome: Phase 2a: Change From Baseline in Sleep Loss VAS Over Time
Description: Participants rated intensity of their average sleeplessness over previous 3 days on 0-10 line scale (0=no sleeplessness, 10=worst imaginable sleeplessness).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24
Population: as for outcome 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
units on a scale
  Week 1 | -2.0 (0.54) | -1.5 (0.42)
  Week 2 | -2.8 (0.58) | -1.2 (0.50)
  Week 3 | -3.3 (0.63) | -1.4 (0.61)
  Week 4 | -3.9 (0.71) | -2.5 (0.57)
  Week 5 | -4.2 (0.71) | -2.3 (0.59)
  Week 6 | -4.1 (0.73) | -1.7 (0.61)
  Week 7 | -4.8 (0.73) | -2.4 (0.61)
  Week 8 | -4.5 (0.68) | -2.5 (0.53)
  Week 9: number analyzed (Participants) | 10 | 14
  Week 9 | -4.3 (1.16) | -3.1 (0.74)
  Week 10: number analyzed (Participants) | 22 | 26
  Week 10 | -4.8 (0.74) | -2.7 (0.57)
  Week 11: number analyzed (Participants) | 10 | 14
  Week 11 | -4.0 (1.23) | -3.8 (0.74)
  Week 12: number analyzed (Participants) | 22 | 26
  Week 12 | -4.3 (0.64) | -3.1 (0.55)
  Week 13: number analyzed (Participants) | 10 | 14
  Week 13 | -4.1 (1.27) | -2.7 (0.82)
  Week 14: number analyzed (Participants) | 10 | 14
  Week 14 | -4.1 (1.24) | -3.1 (0.85)
  Week 15: number analyzed (Participants) | 10 | 14
  Week 15 | -3.9 (1.21) | -3.2 (0.90)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -4.4 (0.70) | -2.8 (0.59)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -4.3 (1.20) | -2.9 (0.81)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -4.0 (1.27) | -2.8 (0.97)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -4.3 (1.20) | -2.6 (1.07)

12. Secondary Outcome: Phase 2a: Percent Change From Baseline in Sleep Loss VAS Over Time
Description: Participants rated intensity of their average sleeplessness over previous 3 days on 0-10 line scale (0=no sleeplessness, 10=worst imaginable sleeplessness). The least squares mean (LSM) and LSM difference were rounded up or down to the nearest single decimal place.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage change
  Week 1 | -22.0 (9.95) | -13.1 (9.66)
  Week 2 | -25.5 (10.77) | -2.2 (10.46)
  Week 3 | -25.1 (19.68) | 2.5 (19.11)
  Week 4 | -44.9 (9.02) | -25.7 (8.75)
  Week 5 | -48.5 (9.02) | -22.6 (8.75)
  Week 6 | -40.1 (16.09) | -7.5 (15.62)
  Week 7 | -53.8 (9.25) | -25.7 (8.98)
  Week 8 | -56.3 (7.72) | -30.0 (7.50)
  Week 9: number analyzed (Participants) | 10 | 14
  Week 9 | -45.1 (12.13) | -38.0 (10.37)
  Week 10: number analyzed (Participants) | 22 | 26
  Week 10 | -56.9 (8.25) | -29.7 (7.87)
  Week 11: number analyzed (Participants) | 10 | 14
  Week 11 | -50.6 (13.53) | -43.5 (11.57)
  Week 12: number analyzed (Participants) | 22 | 26
  Week 12 | -50.4 (7.85) | -35.9 (7.48)
  Week 13: number analyzed (Participants) | 10 | 14
  Week 13 | -54.2 (14.30) | -29.4 (12.23)
  Week 14: number analyzed (Participants) | 10 | 14
  Week 14 | -50.0 (13.52) | -34.8 (11.56)
  Week 15: number analyzed (Participants) | 10 | 14
  Week 15 | -44.2 (16.22) | -31.4 (13.88)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -52.4 (9.11) | -27.1 (8.69)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -54.3 (12.93) | -37.7 (11.84)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -42.9 (15.26) | -34.8 (13.97)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -50.2 (19.88) | -24.6 (18.20)
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 1; Test type: Superiority; p = 0.5172, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -8.9, 95% CI 2-sided [-36.42 to 18.60], Standard Error of Mean 13.65
Statistical Analysis 2: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 2; Test type: Superiority; p = 0.1228, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -23.2, 95% CI 2-sided [-53.02 to 6.53], Standard Error of Mean 14.77
Statistical Analysis 3: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 3; Test type: Superiority; p = 0.3129, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -27.6, 95% CI 2-sided [-81.95 to 26.84], Standard Error of Mean 26.99
Statistical Analysis 4: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 4; Test type: Superiority; p = 0.1277, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -19.2, 95% CI 2-sided [-44.11 to 5.72], Standard Error of Mean 12.36
Statistical Analysis 5: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 5; Test type: Superiority; p = 0.0424, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -25.8, 95% CI 2-sided [-50.76 to -0.92], Standard Error of Mean 12.36
Statistical Analysis 6: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 6; Test type: Superiority; p = 0.1465, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -32.6, 95% CI 2-sided [-77.08 to 11.85], Standard Error of Mean 22.06
Statistical Analysis 7: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 7; Test type: Superiority; p = 0.0316, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -28.2, 95% CI 2-sided [-53.71 to -2.59], Standard Error of Mean 12.68
Statistical Analysis 8: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 8; Test type: Superiority; p = 0.0169, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -26.3, 95% CI 2-sided [-47.63 to -4.95], Standard Error of Mean 10.59
Statistical Analysis 9: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 9; Test type: Superiority; p = 0.6641, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -7.1, 95% CI 2-sided [-40.80 to 26.59], Standard Error of Mean 16.10
Statistical Analysis 10: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 10; Test type: Superiority; p = 0.0199, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -27.2, 95% CI 2-sided [-49.94 to -4.53], Standard Error of Mean 11.26
Statistical Analysis 11: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 11; Test type: Superiority; p = 0.6980, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -7.1, 95% CI 2-sided [-44.67 to 30.51], Standard Error of Mean 17.96
Statistical Analysis 12: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 12; Test type: Superiority; p = 0.1838, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -14.5, 95% CI 2-sided [-36.05 to 7.13], Standard Error of Mean 10.70
Statistical Analysis 13: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 13; Test type: Superiority; p = 0.2078, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -24.8, 95% CI 2-sided [-64.50 to 14.98], Standard Error of Mean 18.99
Statistical Analysis 14: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 14; Test type: Superiority; p = 0.4090, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -15.2, 95% CI 2-sided [-52.72 to 22.41], Standard Error of Mean 17.95
Statistical Analysis 15: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 15; Test type: Superiority; p = 0.5580, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -12.8, 95% CI 2-sided [-57.92 to 32.23], Standard Error of Mean 21.54
Statistical Analysis 16: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 16; Test type: Superiority; p = 0.0486, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -25.2, 95% CI 2-sided [-50.30 to -0.16], Standard Error of Mean 12.43
Statistical Analysis 17: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 18; Test type: Superiority; p = 0.3613, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -16.6, 95% CI 2-sided [-54.06 to 20.78], Standard Error of Mean 17.73
Statistical Analysis 18: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 20; Test type: Superiority; p = 0.7042, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -8.1, 95% CI 2-sided [-52.24 to 36.08], Standard Error of Mean 20.93
Statistical Analysis 19: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 24; Test type: Superiority; p = 0.3602, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -25.6, 95% CI 2-sided [-83.17 to 31.89], Standard Error of Mean 27.27

13. Secondary Outcome: Phase 2a: Change From Baseline in Weekly Average of Difficulty Falling Asleep NRS Over Time
Description: Participants rate difficulty falling asleep daily on Numerical Rating Scale (0=no difficulty, 10=extremely difficult).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
units on a scale
  Week 1 | -1.3 (0.37) | -0.9 (0.30)
  Week 2 | -1.9 (0.46) | -1.7 (0.34)
  Week 3 | -2.6 (0.54) | -2.1 (0.41)
  Week 4 | -3.2 (0.63) | -2.4 (0.43)
  Week 5 | -3.5 (0.67) | -2.7 (0.42)
  Week 6 | -3.7 (0.70) | -2.9 (0.40)
  Week 7 | -3.7 (0.73) | -3.0 (0.43)
  Week 8 | -3.8 (0.74) | -3.1 (0.45)
  Week 9 | -3.6 (0.72) | -3.2 (0.43)
  Week 10 | -3.6 (0.68) | -3.3 (0.39)
  Week 11 | -3.5 (0.69) | -3.4 (0.44)
  Week 12 | -3.4 (0.69) | -3.2 (0.41)
  Week 13 | -3.6 (0.68) | -3.2 (0.44)
  Week 14 | -3.5 (0.69) | -3.0 (0.44)
  Week 15 | -3.6 (0.70) | -3.1 (0.44)
  Week 16 | -3.6 (0.69) | -3.2 (0.45)
  Week 17: number analyzed (Participants) | 11 | 12
  Week 17 | -3.0 (1.14) | -2.9 (0.74)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -3.3 (1.16) | -2.9 (0.78)
  Week 19: number analyzed (Participants) | 10 | 12
  Week 19 | -3.3 (1.16) | -2.9 (0.76)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -3.4 (1.16) | -3.0 (0.83)
  Week 21: number analyzed (Participants) | 10 | 12
  Week 21 | -3.4 (1.18) | -3.1 (0.83)
  Week 22: number analyzed (Participants) | 10 | 12
  Week 22 | -3.4 (1.17) | -2.8 (0.78)
  Week 23: number analyzed (Participants) | 10 | 12
  Week 23 | -3.4 (1.18) | -3.1 (0.83)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -3.3 (1.18) | -3.2 (0.84)

14. Secondary Outcome: Phase 2a: Percent Change From Baseline in Weekly Average of Difficulty Falling Asleep NRS Over Time
Description: Participants rate difficulty falling asleep daily on Numerical Rating Scale (0=no difficulty, 10=extremely difficult). The least squares mean (LSM) and LSM difference were rounded up or down to the nearest single decimal place.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage change
  Week 1 | -17.2 (5.20) | -13.5 (5.02)
  Week 2 | -24.2 (5.78) | -22.5 (5.58)
  Week 3 | -31.6 (6.15) | -25.8 (5.94)
  Week 4 | -39.2 (6.98) | -30.8 (6.74)
  Week 5 | -43.1 (7.58) | -35.1 (7.32)
  Week 6 | -44.0 (7.87) | -37.9 (7.60)
  Week 7 | -44.2 (8.04) | -39.0 (7.77)
  Week 8 | -45.4 (8.13) | -39.1 (7.85)
  Week 9 | -42.1 (8.10) | -41.0 (7.83)
  Week 10 | -43.3 (7.53) | -43.3 (7.27)
  Week 11 | -41.2 (7.78) | -43.7 (7.51)
  Week 12 | -40.8 (7.72) | -40.0 (7.45)
  Week 13 | -44.5 (7.26) | -39.2 (7.01)
  Week 14 | -45.3 (7.33) | -36.5 (7.08)
  Week 15 | -46.2 (7.30) | -37.2 (7.05)
  Week 16 | -46.3 (7.51) | -40.4 (7.25)
  Week 17: number analyzed (Participants) | 11 | 12
  Week 17 | -41.5 (12.68) | -39.0 (12.18)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -44.3 (12.62) | -37.8 (11.61)
  Week 19: number analyzed (Participants) | 10 | 12
  Week 19 | -44.7 (12.66) | -38.6 (11.65)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -44.0 (12.84) | -40.3 (11.81)
  Week 21: number analyzed (Participants) | 10 | 12
  Week 21 | -46.1 (13.37) | -41.4 (12.30)
  Week 22: number analyzed (Participants) | 10 | 12
  Week 22 | -44.1 (12.68) | -36.9 (11.67)
  Week 23: number analyzed (Participants) | 10 | 12
  Week 23 | -43.9 (13.02) | -40.1 (11.98)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -42.9 (12.82) | -41.5 (11.80)
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 1; Test type: Superiority; p = 0.5896, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -3.8, 95% CI 2-sided [-17.83 to 10.26], Standard Error of Mean 6.97
Statistical Analysis 2: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 2; Test type: Superiority; p = 0.8292, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -1.7, 95% CI 2-sided [-17.29 to 13.93], Standard Error of Mean 7.75
Statistical Analysis 3: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 3; Test type: Superiority; p = 0.4852, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -5.8, 95% CI 2-sided [-22.39 to 10.80], Standard Error of Mean 8.23
Statistical Analysis 4: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 4; Test type: Superiority; p = 0.3731, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -8.4, 95% CI 2-sided [-27.24 to 10.42], Standard Error of Mean 9.34
Statistical Analysis 5: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 5; Test type: Superiority; p = 0.4360, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -8.0, 95% CI 2-sided [-28.44 to 12.48], Standard Error of Mean 10.15
Statistical Analysis 6: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 6; Test type: Superiority; p = 0.5655, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -6.1, 95% CI 2-sided [-27.36 to 15.15], Standard Error of Mean 10.54
Statistical Analysis 7: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 7; Test type: Superiority; p = 0.6302, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -5.2, 95% CI 2-sided [-26.93 to 16.49], Standard Error of Mean 10.77
Statistical Analysis 8: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 8; Test type: Superiority; p = 0.5671, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -6.3, 95% CI 2-sided [-28.23 to 15.67], Standard Error of Mean 10.89
Statistical Analysis 9: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 9; Test type: Superiority; p = 0.935, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -1.0, 95% CI 2-sided [-22.93 to 29.83], Standard Error of Mean 10.86
Statistical Analysis 10: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 10; Test type: Superiority; p = 0.9982, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = 0.0, 95% CI 2-sided [-20.30 to 20.34], Standard Error of Mean 10.08
Statistical Analysis 11: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 11; Test type: Superiority; p = 0.8102, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = 2.5, 95% CI 2-sided [-18.48 to 23.51], Standard Error of Mean 10.42
Statistical Analysis 12: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 12; Test type: Superiority; p = 0.9334, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -0.9, 95% CI 2-sided [-21.70 to 19.97], Standard Error of Mean 10.34
Statistical Analysis 13: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 13; Test type: Superiority; p = 0.5873, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -5.3, 95% CI 2-sided [-24.92 to 14.29], Standard Error of Mean 9.73
Statistical Analysis 14: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 14; Test type: Superiority; p = 0.3737, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -8.8, 95% CI 2-sided [-28.61 to 10.96], Standard Error of Mean 9.82
Statistical Analysis 15: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 15; Test type: Superiority; p = 0.3631, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -9.0, 95% CI 2-sided [-28.70 to 10.72], Standard Error of Mean 9.78
Statistical Analysis 16: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 16; Test type: Superiority; p = 0.5585, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -5.9, 95% CI 2-sided [-26.20 to 14.34], Standard Error of Mean 10.06
Statistical Analysis 17: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 17; Test type: Superiority; p = 0.8889, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -2.5, 95% CI 2-sided [-39.58 to 34.58], Standard Error of Mean 17.65
Statistical Analysis 18: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 18; Test type: Superiority; p = 0.7099, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -6.5, 95% CI 2-sided [-42.67 to 29.70], Standard Error of Mean 17.15
Statistical Analysis 19: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 19; Test type: Superiority; p = 0.7270, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -6.1, 95% CI 2-sided [-42.40 to 30.19], Standard Error of Mean 17.20
Statistical Analysis 20: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 20; Test type: Superiority; p = 0.8366, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -3.7, 95% CI 2-sided [-40.47 to 33.16], Standard Error of Mean 17.45
Statistical Analysis 21: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 21; Test type: Superiority; p = 0.8013, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -4.6, 95% CI 2-sided [-42.99 to 33.69], Standard Error of Mean 18.17
Statistical Analysis 22: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 22; Test type: Superiority; p = 0.6810, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -7.2, 95% CI 2-sided [-43.56 to 29.15], Standard Error of Mean 17.23
Statistical Analysis 23: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 23; Test type: Superiority; p = 0.8347, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -3.7, 95% CI 2-sided [-41.08 to 33.58], Standard Error of Mean 17.69
Statistical Analysis 24: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 24; Test type: Superiority; p = 0.9358, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -1.4, 95% CI 2-sided [-38.18 to 35.33], Standard Error of Mean 17.42

15. Secondary Outcome: Phase 2a: Change From Baseline in Weekly Average of Sleep Quality NRS Over Time
Description: Participants rated daily sleep quality on Numerical Rating Scale (0=best possible sleep, 10=worst possible sleep).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
units on a scale
  Week 1 | -1.4 (0.38) | -0.8 (0.26)
  Week 2 | -1.9 (0.45) | -1.5 (0.33)
  Week 3 | -2.6 (0.55) | -1.7 (0.35)
  Week 4 | -3.1 (0.67) | -2.1 (0.36)
  Week 5 | -3.4 (0.68) | -2.2 (0.39)
  Week 6 | -3.6 (0.67) | -2.4 (0.39)
  Week 7 | -3.8 (0.71) | -2.5 (0.41)
  Week 8 | -3.8 (0.71) | -2.6 (0.42)
  Week 9 | -3.5 (0.67) | -2.8 (0.41)
  Week 10 | -3.6 (0.66) | -2.8 (0.43)
  Week 11 | -3.4 (0.68) | -3.1 (0.42)
  Week 12 | -3.3 (0.67) | -2.9 (0.41)
  Week 13 | -3.5 (0.70) | -3.0 (0.43)
  Week 14 | -3.6 (0.71) | -2.9 (0.46)
  Week 15 | -3.7 (0.71) | -3.0 (0.46)
  Week 16 | -3.7 (0.68) | -3.1 (0.45)
  Week 17: number analyzed (Participants) | 11 | 12
  Week 17 | -2.6 (1.10) | -2.7 (0.79)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -3.1 (1.16) | -2.9 (0.79)
  Week 19: number analyzed (Participants) | 10 | 12
  Week 19 | -3.2 (1.17) | -2.8 (0.77)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -3.0 (1.14) | -2.9 (0.84)
  Week 21: number analyzed (Participants) | 10 | 12
  Week 21 | -3.3 (1.18) | -2.8 (0.86)
  Week 22: number analyzed (Participants) | 10 | 12
  Week 22 | -3.2 (1.17) | -2.8 (0.78)
  Week 23: number analyzed (Participants) | 10 | 12
  Week 23 | -3.2 (1.18) | -2.8 (0.84)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -3.3 (1.16) | -2.7 (0.78)

16. Secondary Outcome: Phase 2a: Percent Change From Baseline in Weekly Average of Sleep Quality NRS Over Time
Description: Participants rated daily sleep quality on Numerical Rating Scale (0=best possible sleep, 10=worst possible sleep). The least squares mean (LSM) and LSM difference were rounded up or down to the nearest single decimal place.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage change
  Week 1 | -11.0 (5.98) | -12.0 (5.78)
  Week 2 | -21.9 (5.59) | -20.6 (5.40)
  Week 3 | -29.6 (5.94) | -20.9 (5.74)
  Week 4 | -33.6 (7.04) | -26.1 (6.80)
  Week 5 | -39.6 (7.24) | -28.8 (6.99)
  Week 6 | -42.8 (7.23) | -30.9 (6.99)
  Week 7 | -45.3 (7.40) | -31.1 (7.14)
  Week 8 | -46.1 (7.52) | -33.5 (7.27)
  Week 9 | -42.0 (7.52) | -37.0 (7.26)
  Week 10 | -42.8 (7.38) | -36.0 (7.12)
  Week 11 | -41.5 (7.49) | -39.2 (7.23)
  Week 12 | -40.1 (7.37) | -36.1 (7.11)
  Week 13 | -40.9 (7.66) | -37.5 (7.40)
  Week 14 | -40.3 (8.40) | -36.9 (8.12)
  Week 15 | -44.0 (7.94) | -37.0 (7.67)
  Week 16 | -45.7 (7.71) | -38.8 (7.45)
  Week 17: number analyzed (Participants) | 11 | 12
  Week 17 | -33.2 (12.43) | -35.8 (11.94)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -38.8 (12.59) | -37.1 (11.59)
  Week 19: number analyzed (Participants) | 10 | 12
  Week 19 | -41.4 (12.76) | -36.3 (11.74)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -37.3 (12.79) | -37.6 (11.77)
  Week 21: number analyzed (Participants) | 10 | 12
  Week 21 | -42.3 (13.40) | -36.5 (12.33)
  Week 22: number analyzed (Participants) | 10 | 12
  Week 22 | -39.7 (12.70) | -35.9 (11.68)
  Week 23: number analyzed (Participants) | 10 | 12
  Week 23 | -41.2 (13.42) | -34.8 (12.34)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -42.4 (13.00) | -35.0 (11.96)
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 1; Test type: Superiority; p = 0.8948, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week. Program:; LS Mean Difference = 1.1, 95% CI 2-sided [-15.20 to 17.35], Standard Error of Mean 8.08
Statistical Analysis 2: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 2; Test type: Superiority; p = 0.8581, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -1.4, 95% CI 2-sided [-16.58 to 13.86], Standard Error of Mean 7.55
Statistical Analysis 3: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 3; Test type: Superiority; p = 0.2797, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -8.8, 95% CI 2-sided [-24.93 to 7.38], Standard Error of Mean 8.02
Statistical Analysis 4: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 4; Test type: Superiority; p = 0.4333, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -7.5, 95% CI 2-sided [-26.67 to 11.64], Standard Error of Mean 9.50
Statistical Analysis 5: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 5; Test type: Superiority; p = 0.2774, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -10.7, 95% CI 2-sided [-30.44 to 8.95], Standard Error of Mean 9.77
Statistical Analysis 6: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 6; Test type: Superiority; p = 0.2308, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -11.9, 95% CI 2-sided [-31.55 to 7.82], Standard Error of Mean 9.77
Statistical Analysis 7: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 7; Test type: Superiority; p = 0.1617, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -14.2, 95% CI 2-sided [-34.34 to 5.91], Standard Error of Mean 9.99
Statistical Analysis 8: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 8; Test type: Superiority; p = 0.2220, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -12.6, 95% CI 2-sided [-33.05 to 7.89], Standard Error of Mean 10.16
Statistical Analysis 9: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 9; Test type: Superiority; p = 0.6195, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -5.1, 95% CI 2-sided [-25.54 to 15.38], Standard Error of Mean 10.15
Statistical Analysis 10: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 10; Test type: Superiority; p = 0.4984, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -6.8, 95% CI 2-sided [-26.86 to 13.27], Standard Error of Mean 9.96
Statistical Analysis 11: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 11; Test type: Superiority; p = 0.8147, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -2.4, 95% CI 2-sided [-22.75 to 17.99], Standard Error of Mean 10.11
Statistical Analysis 12: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 12; Test type: Superiority; p = 0.6917, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -4.0, 95% CI 2-sided [-24.01 to 16.07], Standard Error of Mean 9.94
Statistical Analysis 13: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 13; Test type: Superiority; p = 0.7437, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -3.4, 95% CI 2-sided [-24.24 to 17.43], Standard Error of Mean 10.34
Statistical Analysis 14: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 14; Test type: Superiority; p = 0.7663, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -3.4, 95% CI 2-sided [-26.26 to 19.47], Standard Error of Mean 11.34
Statistical Analysis 15: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 15; Test type: Superiority; p = 0.5157, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -7.0, 95% CI 2-sided [-28.61 to 14.75], Standard Error of Mean 10.71
Statistical Analysis 16: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 16; Test type: Superiority; p = 0.5115, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -6.9, 95% CI 2-sided [-27.86 to 14.09], Standard Error of Mean 10.41
Statistical Analysis 17: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 17; Test type: Superiority; p = 0.8795, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = 2.7, 95% CI 2-sided [-33.68 to 39.00], Standard Error of Mean 17.30
Statistical Analysis 18: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 18; Test type: Superiority; p = 0.9254, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -1.6, 95% CI 2-sided [-37.73 to 34.48], Standard Error of Mean 17.11
Statistical Analysis 19: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 19; Test type: Superiority; p = 0.7718, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -5.1, 95% CI 2-sided [-41.68 to 31.47], Standard Error of Mean 17.34
Statistical Analysis 20: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 20; Test type: Other; p = 0.9855, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = 0.3, 95% CI 2-sided [-36.34 to 36.98], Standard Error of Mean 17.38
Statistical Analysis 21: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 21; Test type: Superiority; p = 0.7508, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -5.9, 95% CI 2-sided [-44.29 to 32.54], Standard Error of Mean 18.21
Statistical Analysis 22: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 22; Test type: Superiority; p = 0.8260, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -3.9, 95% CI 2-sided [-40.26 to 32.55], Standard Error of Mean 17.26
Statistical Analysis 23: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 23; Test type: Superiority; p = 0.7259, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -6.5, 95% CI 2-sided [-44.95 to 31.96], Standard Error of Mean 18.23
Statistical Analysis 24: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 24; Test type: Superiority; p = 0.6826, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -7.3, 95% CI 2-sided [-44.61 to 29.92], Standard Error of Mean 17.66

17. Secondary Outcome: Phase 2a: Change From Baseline in Quality of Life (QoL) Measure Dermatology QoL Index (DLQI) Over Time
Description: QoL was assessed at designated visits and includes the DLQI whereby 0=no effect on quality of life; 30= extremely large effect on QoL.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 16, 24
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period. Baseline through Week 8: LOCF; Weeks 12-24: participants with an assessment at given time point.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
score on a scale
  Week 2 | -6.7 (1.23) | -2.8 (0.82)
  Week 4 | -8.3 (1.45) | -4.5 (0.87)
  Week 6 | -8.9 (1.45) | -6.1 (0.85)
  Week 8 | -9.4 (1.62) | -6.3 (0.94)
  Week 12: number analyzed (Participants) | 10 | 14
  Week 12 | -6.8 (2.22) | -7.3 (1.33)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -8.1 (1.64) | -6.9 (0.88)
  Week 24: number analyzed (Participants) | 9 | 12
  Week 24 | -7.0 (2.71) | -7.3 (1.92)

18. Secondary Outcome: Phase 2a: Percent Change From Baseline in QoL Measure DLQI Over Time
Description: as for outcome 17
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 16, 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage change
  Week 2 | -40.0 (6.26) | -12.0 (6.09)
  Week 4 | -50.4 (6.09) | -29.1 (5.93)
  Week 6 | -54.1 (6.34) | -41.7 (6.16)
  Week 8 | -55.4 (7.15) | -43.0 (6.95)
  Week 12: number analyzed (Participants) | 10 | 14
  Week 12 | -46.9 (10.33) | -46.1 (8.80)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -49.6 (6.51) | -45.2 (6.23)
  Week 24: number analyzed (Participants) | 9 | 12
  Week 24 | -54.6 (12.86) | -46.0 (11.12)
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 2; Test type: Superiority; p = 0.0018, ANCOVA — from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -28.0, 95% CI 2-sided [-44.96 to -10.97], Standard Error of Mean 8.43
Statistical Analysis 2: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 4; Test type: Superiority; p = 0.0127, ANCOVA — from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -21.3, 95% CI 2-sided [-37.83 to -4.77], Standard Error of Mean 8.20
Statistical Analysis 3: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 6; Test type: Superiority; p = 0.1547, ANCOVA — from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -12.4, 95% CI 2-sided [-29.54 to 4.84], Standard Error of Mean 8.53
Statistical Analysis 4: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 8; Test type: Superiority; p = 0.2048, ANCOVA — from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -12.4, 95% CI 2-sided [-31.78 to 7.01], Standard Error of Mean 9.62
Statistical Analysis 5: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 12; Test type: Superiority; p = 0.9508, ANCOVA — from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -0.8, 95% CI 2-sided [-29.28 to 27.58], Standard Error of Mean 13.58
Statistical Analysis 6: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 16; Test type: Superiority; p = 0.6140, ANCOVA — from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -4.4, 95% CI 2-sided [-22.07 to 13.19], Standard Error of Mean 8.74
Statistical Analysis 7: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 24; Test type: Superiority; p = 0.6207, ANCOVA — from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -8.6, 95% CI 2-sided [-44.94 to 27.66], Standard Error of Mean 17.12

19. Secondary Outcome: Phase 2a: Change From Baseline in QoL Measure Itchy Quality of Life (ItchyQoL) Over Time
Description: ItchyQoL focuses on impact of pruritus on daily activities and on the level of psychological stress. It contains 22 items. The frequency items are scored using a 5-point Likert scale ranging from "never" to "all the time". The bother items are scored from 1 (not bothered) to 5 (severely bothered). The recall period in ItchyQoL is the past week. The ItchyQoL total score is defined as the sum of all 22-items scores. Total scores can be classified as little (0-30), mild (31-50), moderate (51-80), and severe (81-110).
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 16, 24
Population: as for outcome 17
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
units on a scale
  Week 2 | -16.3 (3.18) | -6.2 (1.08)
  Week 4 | -25.3 (4.32) | -11.0 (2.22)
  Week 6 | -27.6 (4.60) | -14.5 (2.50)
  Week 8 | -30.0 (4.80) | -16.0 (2.54)
  Week 12: number analyzed (Participants) | 10 | 14
  Week 12 | -26.0 (7.57) | -18.1 (3.51)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -29.6 (4.96) | -15.8 (2.49)
  Week 24: number analyzed (Participants) | 9 | 12
  Week 24 | -26.3 (8.44) | -19.1 (5.15)

20. Secondary Outcome: Phase 2a: Percent Change From Baseline in QoL Measure Itchy QoL Over Time
Description: ItchyQoL focuses on impact of pruritus on daily activities and on the level of psychological stress. It contains 22 items. The frequency items are scored using a 5-point Likert scale ranging from "never" to "all the time". The bother items are scored from 1 (not bothered) to 5 (severely bothered). The recall period in ItchyQoL is the past week. The ItchyQoL total score is defined as the sum of all 22-items scores. Total scores can be classified as little (0-30), mild (31-50), moderate (51-80), and severe (81-110). The least squares mean (LSM) and LSM difference were rounded up or down to the nearest single decimal place.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 16, 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage change
  Week 2 | -16.4 (2.60) | -6.6 (2.53)
  Week 4 | -27.5 (3.78) | -14.1 (3.68)
  Week 6 | -29.6 (3.99) | -17.7 (3.89)
  Week 8 | -32.6 (4.25) | -18.8 (4.14)
  Week 12: number analyzed (Participants) | 10 | 14
  Week 12 | -29.7 (6.26) | -21.1 (5.37)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -32.2 (4.26) | -17.1 (4.07)
  Week 24: number analyzed (Participants) | 9 | 12
  Week 24 | -29.8 (7.56) | -22.0 (6.57)
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 2; Test type: Superiority; p = 0.0079, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -9.8, 95% CI 2-sided [-16.89 to -2.71], Standard Error of Mean 3.52
Statistical Analysis 2: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 4; Test type: Superiority; p = 0.0122, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -13.4, 95% CI 2-sided [-23.69 to -3.06], Standard Error of Mean 5.12
Statistical Analysis 3: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 6; Test type: Superiority; p = 0.0328, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -11.9, 95% CI 2-sided [-22.80 to -1.02], Standard Error of Mean 5.40
Statistical Analysis 4: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 8; Test type: Superiority; p = 0.0212, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -13.8, 95% CI 2-sided [-25.36 to -2.15], Standard Error of Mean 5.76
Statistical Analysis 5: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 12; Test type: Superiority; p = 0.3112, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -8.6, 95% CI 2-sided [-25.95 to 8.72], Standard Error of Mean 8.28
Statistical Analysis 6: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 16; Test type: Superiority; p = 0.0113, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -15.2, 95% CI 2-sided [-26.75 to -3.61], Standard Error of Mean 5.74
Statistical Analysis 7: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 24; Test type: Superiority; p = 0.4540, ANCOVA — Calculated from ANCOVA models including treatment as fixed effect, sex, atopy and baseline value as covariates by week; LS Mean Difference = -7.8, 95% CI 2-sided [-29.20 to 13.68], Standard Error of Mean 10.11

21. Secondary Outcome: Phase 2a: Change From Baseline in Prurigo Nodularis Nodule Assessment Tool (PN-NAT) Over Time: Number of Nodules Over the Whole Body Score
Description: PN-NAT, assessed at designated visits, is a novel exploratory tool for the evaluation of disease severity based on estimate of the number of nodules over the whole body, estimate of hardness of nodules over the whole body, estimate of extent of excoriation over the whole body, distribution of nodules, exact number of nodules in the representative area. The first three components (number of nodules over the whole body, estimate of hardness of nodules over the whole body, estimate of extent of excoriations over the whole body) were analyzed as secondary endpoints. For the Number of Nodules over the Whole Body score: 0=0 nodules; 1=1 to 9 nodules; 2=10 to 50 nodules; and 3=more than 50 nodules. A higher score indicates worse disease.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24
Population: as for outcome 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
score on a scale
  Week 2 | -0.2 (0.08) | -0.1 (0.08)
  Week 4 | -0.4 (0.14) | -0.2 (0.08)
  Week 6 | -0.5 (0.14) | -0.2 (0.12)
  Week 8 | -0.5 (0.16) | -0.3 (0.11)
  Week 10: number analyzed (Participants) | 22 | 26
  Week 10 | -0.5 (0.16) | -0.3 (0.09)
  Week 12: number analyzed (Participants) | 22 | 26
  Week 12 | -0.7 (0.18) | -0.4 (0.11)
  Week 14: number analyzed (Participants) | 10 | 14
  Week 14 | -0.9 (0.28) | -0.5 (0.14)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -1.0 (0.19) | -0.3 (0.09)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -0.9 (0.28) | -0.5 (0.15)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -0.9 (0.28) | -0.4 (0.15)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -0.9 (0.28) | -0.5 (0.15)

22. Secondary Outcome: Phase 2a: Change From Baseline in PN-NAT Over Time: Estimate of Hardness of Nodules Over the Whole Body
Description: PN-NAT, assessed at designated visits, is a novel exploratory tool for the evaluation of disease severity based on estimate of the number of nodules over the whole body, estimate of hardness of nodules over the whole body, estimate of extent of excoriation over the whole body, distribution of nodules, exact number of nodules in the representative area. The first three components (number of nodules over the whole body, estimate of hardness of nodules over the whole body, estimate of extent of excoriations over the whole body) were analyzed as secondary endpoints. For the Estimate of Hardness of Nodules Over the Whole Body score: 0=No nodules are hard; 1=Up to one-third of nodules are hard; 2=One-third to two-thirds of nodules are hard; and 3=More than two-thirds of nodules are hard. A higher score indicates worse disease.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24
Population: as for outcome 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
score on a scale
  Week 2 | -0.2 (0.12) | -0.2 (0.12)
  Week 4 | -0.5 (0.19) | -0.4 (0.15)
  Week 6 | -0.6 (0.23) | -0.5 (0.16)
  Week 8 | -0.7 (0.23) | -0.6 (0.17)
  Week 10: number analyzed (Participants) | 22 | 26
  Week 10 | -1.1 (0.23) | -0.8 (0.17)
  Week 12: number analyzed (Participants) | 22 | 26
  Week 12 | -1.0 (0.22) | -0.8 (0.19)
  Week 14: number analyzed (Participants) | 10 | 14
  Week 14 | -1.2 (0.39) | -0.9 (0.25)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -1.1 (0.24) | -0.8 (0.20)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -1.2 (0.42) | -0.9 (0.26)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -1.3 (0.45) | -1.2 (0.24)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -1.2 (0.39) | -0.8 (0.18)

23. Secondary Outcome: Phase 2a: Change From Baseline in PN-NAT Over Time: Extent of Excoriations Over the Whole Body
Description: PN-NAT, assessed at designated visits, is a novel exploratory tool for the evaluation of disease severity based on estimate of the number of nodules over the whole body, estimate of hardness of nodules over the whole body, estimate of extent of excoriation over the whole body, distribution of nodules, exact number of nodules in the representative area. The first three components (number of nodules over the whole body, estimate of hardness of nodules over the whole body, estimate of extent of excoriations over the whole body) were analyzed as secondary endpoints. For the Extent of Excoriations over the Whole Body score: 0=No nodules are excoriated; 1=Up to one-third of nodules are excoriated; 2=One-third to two-thirds of nodules are excoriated; and 3=More than two-thirds of nodules are excoriated. A higher score indicates worse disease.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24
Population: as for outcome 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
score on a scale
  Week 2 | -0.2 (0.14) | -0.2 (0.10)
  Week 4 | -0.5 (0.23) | -0.7 (0.16)
  Week 6 | -0.6 (0.27) | -0.7 (0.17)
  Week 8 | -0.4 (0.26) | -0.7 (0.17)
  Week 10: number analyzed (Participants) | 22 | 26
  Week 10 | -0.7 (0.23) | -0.8 (0.16)
  Week 12: number analyzed (Participants) | 22 | 26
  Week 12 | -0.8 (0.23) | -0.8 (0.16)
  Week 14: number analyzed (Participants) | 10 | 14
  Week 14 | -1.0 (0.37) | -1.0 (0.23)
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | -1.1 (0.19) | -0.7 (0.16)
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | -1.0 (0.37) | -1.0 (0.25)
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | -1.0 (0.33) | -1.1 (0.26)
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | -0.8 (0.29) | -0.8 (0.27)

24. Secondary Outcome: Phase 2a: Percentage of Participants With Improvement in Prurigo Nodularis Investigator Global Assessment (PN-IGA) by 2 Categories Over Time
Description: PN-IGA, assessed at designated visits, is a novel exploratory tool for the overall investigator assessment of PN disease severity based on the presence/absence of nodules and the size of the nodules as defined by their elevation. The IGA utilizes a 5-point scale that ranges from 0 (clear) to 4 (severe disease).
Time Frame: Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period; Baseline through Week 8: LOCF; Weeks 10-24: participants with an assessment at given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW
Number analyzed (Participants) | 23 | 26
percentage of participants
  Week 2 | 8.7 [1.1 to 28.0] | 7.7 [0.9 to 25.1]
  Week 4 | 13.0 [2.8 to 33.6] | 7.7 [0.9 to 25.1]
  Week 6 | 43.5 [23.2 to 65.5] | 11.5 [2.4 to 30.2]
  Week 8 | 43.5 [23.2 to 65.5] | 15.4 [4.4 to 34.9]
  Week 10: number analyzed (Participants) | 22 | 26
  Week 10 | 40.9 [20.7 to 63.6] | 19.2 [6.6 to 39.4]
  Week 12: number analyzed (Participants) | 22 | 26
  Week 12 | 50.0 [28.2 to 71.8] | 23.1 [9.0 to 43.6]
  Week 14: number analyzed (Participants) | 10 | 14
  Week 14 | 60.0 [26.2 to 87.8] | 35.7 [12.8 to 64.9]
  Week 16: number analyzed (Participants) | 22 | 26
  Week 16 | 59.1 [36.4 to 79.3] | 26.9 [11.6 to 47.8]
  Week 18: number analyzed (Participants) | 10 | 12
  Week 18 | 60.0 [26.2 to 87.8] | 16.7 [2.1 to 48.4]
  Week 20: number analyzed (Participants) | 10 | 12
  Week 20 | 70.0 [34.8 to 93.3] | 16.7 [2.1 to 48.4]
  Week 24: number analyzed (Participants) | 10 | 12
  Week 24 | 50.0 [18.7 to 81.3] | 8.3 [0.2 to 38.5]
Statistical Analysis 1: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 2; Test type: Superiority; p = 0.8436, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.16 to 9.64]
Statistical Analysis 2: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 4; Test type: Superiority; p = 0.4922, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.29 to 13.75]
Statistical Analysis 3: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 6; Test type: Superiority; p = 0.0064, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 7.70, 95% CI 2-sided [1.61 to 36.91]
Statistical Analysis 4: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 8; Test type: Superiority; p = 0.0201, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 5.14, 95% CI 2-sided [1.26 to 20.91]
Statistical Analysis 5: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 10; Test type: Superiority; p = 0.0841, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.95, 95% CI 2-sided [0.82 to 10.55]
Statistical Analysis 6: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 12; Test type: Superiority; p = 0.0292, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 4.14, 95% CI 2-sided [1.12 to 15.22]
Statistical Analysis 7: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 14; Test type: Superiority; p = 0.2259, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [0.51 to 15.00]
Statistical Analysis 8: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 16; Test type: Superiority; p = 0.0104, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 5.44, 95% CI 2-sided [1.41 to 20.95]
Statistical Analysis 9: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 18; Test type: Other; p = 0.0434, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 13.80, 95% CI 2-sided [0.89 to 214.44]
Statistical Analysis 10: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 20; Test type: Superiority; p = 0.0093, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 11: Comparison: Phase 2a - Vixarelimab 360 mg SC QW vs Phase 2a - Placebo SC QW; Week 24; Test type: Superiority; p = 0.0290, Cochran-Mantel-Haenszel — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 14.40, 95% CI 2-sided [1.10 to 189.25]

25. Secondary Outcome: Phase 2b: Percentage of Participants Achieving at Least a 6-Point Reduction From Baseline in Weekly Average WI-NRS at Week 16
Description: Participants rated pruritus daily on the Worst Itch [pruritis]-Numeric Rating Scale (0=no pruritus; 10=worst imaginable pruritus).
Time Frame: Baseline, Week 16
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period. Non-responder imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage of participants | 42.6 [28.3 to 57.8] | 23.4 [12.3 to 38.0] | 17.4 [7.8 to 31.4] | 2.1 [0.1 to 11.1]
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Calculated from CMH tests adjusted by the randomization stratification variables: sex and years since the first nodule observed (≥10 vs. <10 years); Odds Ratio (OR) = 71.24, 95% CI 2-sided [5.35 to 948.31]
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p = 0.0019, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 11.62, 95% CI 2-sided [1.62 to 83.47]
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p = 0.0117, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 8.84, 95% CI 2-sided [1.14 to 68.26]

26. Secondary Outcome: Phase 2b: Percentage of Participants Achieving at Least a 4-point Reduction From Baseline in Weekly Average WI-NRS at Week 16
Description: as for outcome 25
Time Frame: Baseline, Week 16
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage of participants | 66.0 [50.7 to 79.1] | 61.7 [46.4 to 75.5] | 29.8 [17.3 to 44.9] | 16.7 [7.5 to 30.2]
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 8.60, 95% CI 2-sided [3.34 to 22.14]
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 7.60, 95% CI 2-sided [2.91 to 19.79]
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p = 0.1252, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.14, 95% CI 2-sided [0.80 to 5.75]

27. Secondary Outcome: Phase 2b: Percentage of Participants Achieving a Score of 0 or 1 in PN-IGA at Week 16
Description: PN-IGA, assessed at designated visits, is a novel exploratory tool for the overall investigator assessment of PN disease severity based on the presence/absence of nodules and the size of the nodules as defined by their elevation. The IGA utilizes a 5-point scale that ranges from 0 (clear) to 4 (severe disease); 0 (clear) indicates no nodules and 1 (almost clear) indicates nodules are present, few of the nodules are moderately raised.
Time Frame: Week 16
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage of participants | 38.3 [24.5 to 53.6] | 29.8 [17.3 to 44.9] | 14.9 [6.2 to 28.3] | 10.4 [3.5 to 22.7]
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.65, 95% CI 2-sided [1.83 to 17.47]
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p = 0.0196, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.61, 95% CI 2-sided [1.19 to 10.99]
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Test type: Superiority; p = 0.6213, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.40 to 4.69]

28. Secondary Outcome: Phase 2b: Change From Baseline in Weekly Average of WI-NRS Over Time
Description: as for outcome 5
Time Frame: Baseline, Weeks 1 through 52
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period. Participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
units on a scale
  Week 1 | -1.7 (0.21) | -1.1 (0.21) | -0.9 (0.21) | -0.4 (0.21)
  Week 2: number analyzed (Participants) | 46 | 47 | 47 | 48
  Week 2 | -2.8 (0.30) | -1.9 (0.29) | -1.9 (0.30) | -0.7 (0.29)
  Week 3 | -3.4 (0.32) | -2.2 (0.32) | -1.8 (0.32) | -0.7 (0.31)
  Week 4: number analyzed (Participants) | 46 | 47 | 47 | 48
  Week 4 | -3.8 (0.33) | -2.5 (0.33) | -1.5 (0.33) | -0.8 (0.33)
  Week 5: number analyzed (Participants) | 46 | 47 | 47 | 48
  Week 5 | -4.0 (0.33) | -2.9 (0.33) | -2.0 (0.33) | -0.8 (0.33)
  Week 6: number analyzed (Participants) | 45 | 47 | 47 | 48
  Week 6 | -4.2 (0.35) | -3.2 (0.34) | -2.4 (0.34) | -0.9 (0.33)
  Week 7: number analyzed (Participants) | 45 | 47 | 47 | 47
  Week 7 | -4.3 (0.36) | -3.5 (0.35) | -2.3 (0.36) | -0.9 (0.35)
  Week 8: number analyzed (Participants) | 45 | 47 | 47 | 47
  Week 8 | -4.4 (0.37) | -3.6 (0.36) | -2.3 (0.37) | -1.0 (0.36)
  Week 9: number analyzed (Participants) | 45 | 47 | 47 | 47
  Week 9 | -4.6 (0.38) | -3.9 (0.37) | -2.7 (0.38) | -1.1 (0.37)
  Week 10: number analyzed (Participants) | 45 | 46 | 47 | 46
  Week 10 | -4.7 (0.39) | -4.2 (0.39) | -3.1 (0.39) | -1.2 (0.39)
  Week 11: number analyzed (Participants) | 45 | 45 | 47 | 46
  Week 11 | -4.8 (0.40) | -4.2 (0.40) | -2.8 (0.40) | -1.2 (0.40)
  Week 12: number analyzed (Participants) | 45 | 45 | 47 | 46
  Week 12 | -4.8 (0.41) | -3.9 (0.41) | -2.5 (0.40) | -1.3 (0.40)
  Week 13: number analyzed (Participants) | 45 | 45 | 47 | 46
  Week 13 | -4.9 (0.41) | -4.4 (0.41) | -3.1 (0.41) | -1.5 (0.41)
  Week 14: number analyzed (Participants) | 45 | 45 | 47 | 46
  Week 14 | -4.9 (0.42) | -4.5 (0.42) | -3.2 (0.41) | -1.3 (0.41)
  Week 15: number analyzed (Participants) | 45 | 45 | 47 | 46
  Week 15 | -5.0 (0.41) | -4.4 (0.41) | -3.1 (0.41) | -1.2 (0.40)
  Week 16: number analyzed (Participants) | 45 | 45 | 47 | 47
  Week 16 | -4.9 (0.41) | -4.3 (0.42) | -2.9 (0.41) | -1.2 (0.40)
  Week 17: number analyzed (Participants) | 45 | 43 | 46 | 46
  Week 17 | -5.2 (0.43) | -4.9 (0.44) | -3.7 (0.43) | -2.1 (0.42)
  Week 18: number analyzed (Participants) | 45 | 42 | 47 | 46
  Week 18 | -5.3 (0.43) | -4.9 (0.44) | -3.9 (0.42) | -2.7 (0.42)
  Week 19: number analyzed (Participants) | 45 | 42 | 46 | 46
  Week 19 | -5.4 (0.43) | -5.1 (0.44) | -4.4 (0.43) | -3.3 (0.43)
  Week 20: number analyzed (Participants) | 45 | 42 | 47 | 46
  Week 20 | -5.4 (0.43) | -5.0 (0.45) | -4.4 (0.43) | -3.5 (0.43)
  Week 21: number analyzed (Participants) | 43 | 41 | 47 | 46
  Week 21 | -5.5 (0.44) | -5.3 (0.46) | -4.7 (0.43) | -3.9 (0.43)
  Week 22: number analyzed (Participants) | 42 | 41 | 47 | 46
  Week 22 | -5.5 (0.45) | -5.3 (0.46) | -4.6 (0.44) | -4.1 (0.43)
  Week 23: number analyzed (Participants) | 41 | 41 | 47 | 46
  Week 23 | -5.5 (0.46) | -5.3 (0.47) | -4.8 (0.44) | -4.4 (0.44)
  Week 24: number analyzed (Participants) | 42 | 41 | 46 | 46
  Week 24 | -5.5 (0.46) | -5.5 (0.46) | -4.8 (0.44) | -4.4 (0.44)
  Week 25: number analyzed (Participants) | 41 | 41 | 45 | 45
  Week 25 | -5.6 (0.45) | -5.6 (0.46) | -4.9 (0.44) | -4.6 (0.44)
  Week 26: number analyzed (Participants) | 42 | 40 | 45 | 46
  Week 26 | -5.6 (0.45) | -5.7 (0.46) | -4.9 (0.44) | -4.5 (0.43)
  Week 27: number analyzed (Participants) | 42 | 39 | 43 | 46
  Week 27 | -5.5 (0.44) | -5.6 (0.46) | -5.2 (0.44) | -4.5 (0.42)
  Week 28: number analyzed (Participants) | 41 | 40 | 41 | 46
  Week 28 | -5.8 (0.45) | -5.6 (0.46) | -5.1 (0.45) | -4.5 (0.43)
  Week 29: number analyzed (Participants) | 41 | 39 | 43 | 45
  Week 29 | -5.8 (0.43) | -5.8 (0.45) | -5.2 (0.43) | -4.7 (0.42)
  Week 30: number analyzed (Participants) | 41 | 39 | 43 | 46
  Week 30 | -5.9 (0.44) | -5.8 (0.45) | -5.2 (0.44) | -4.5 (0.42)
  Week 31: number analyzed (Participants) | 40 | 39 | 43 | 45
  Week 31 | -6.1 (0.44) | -5.9 (0.45) | -5.3 (0.43) | -4.8 (0.42)
  Week 32: number analyzed (Participants) | 40 | 40 | 42 | 46
  Week 32 | -6.1 (0.44) | -5.8 (0.44) | -5.2 (0.43) | -4.7 (0.41)
  Week 33: number analyzed (Participants) | 39 | 40 | 44 | 46
  Week 33 | -6.0 (0.44) | -5.8 (0.44) | -5.2 (0.42) | -4.8 (0.41)
  Week 34: number analyzed (Participants) | 40 | 40 | 43 | 46
  Week 34 | -6.2 (0.44) | -5.9 (0.44) | -5.3 (0.43) | -4.8 (0.41)
  Week 35: number analyzed (Participants) | 39 | 40 | 43 | 46
  Week 35 | -6.2 (0.45) | -5.7 (0.44) | -5.4 (0.43) | -4.9 (0.41)
  Week 36: number analyzed (Participants) | 39 | 39 | 44 | 46
  Week 36 | -6.2 (0.45) | -5.8 (0.45) | -5.4 (0.43) | -4.9 (0.41)
  Week 37: number analyzed (Participants) | 38 | 39 | 44 | 45
  Week 37 | -6.4 (0.45) | -5.9 (0.45) | -5.5 (0.43) | -5.0 (0.42)
  Week 38: number analyzed (Participants) | 38 | 39 | 44 | 44
  Week 38 | -6.4 (0.45) | -5.9 (0.44) | -5.5 (0.42) | -5.1 (0.42)
  Week 39: number analyzed (Participants) | 38 | 38 | 43 | 45
  Week 39 | -6.4 (0.44) | -6.1 (0.44) | -5.7 (0.42) | -5.1 (0.41)
  Week 40: number analyzed (Participants) | 38 | 38 | 43 | 45
  Week 40 | -6.4 (0.44) | -6.1 (0.44) | -5.7 (0.42) | -5.1 (0.41)
  Week 41: number analyzed (Participants) | 38 | 38 | 41 | 44
  Week 41 | -6.4 (0.43) | -6.1 (0.44) | -5.9 (0.42) | -5.4 (0.41)
  Week 42: number analyzed (Participants) | 38 | 37 | 41 | 43
  Week 42 | -6.5 (0.42) | -6.1 (0.43) | -5.8 (0.41) | -5.4 (0.41)
  Week 43: number analyzed (Participants) | 37 | 38 | 40 | 43
  Week 43 | -6.3 (0.43) | -6.2 (0.43) | -5.9 (0.42) | -5.4 (0.40)
  Week 44: number analyzed (Participants) | 37 | 37 | 40 | 43
  Week 44 | -6.5 (0.43) | -6.0 (0.44) | -5.9 (0.42) | -5.5 (0.41)
  Week 45: number analyzed (Participants) | 38 | 37 | 40 | 43
  Week 45 | -6.6 (0.41) | -6.3 (0.43) | -5.6 (0.41) | -5.4 (0.40)
  Week 46: number analyzed (Participants) | 38 | 38 | 40 | 43
  Week 46 | -6.5 (0.42) | -6.3 (0.43) | -5.6 (0.42) | -5.5 (0.40)
  Week 47: number analyzed (Participants) | 38 | 38 | 40 | 43
  Week 47 | -6.7 (0.43) | -6.2 (0.44) | -5.7 (0.43) | -5.6 (0.41)
  Week 48: number analyzed (Participants) | 38 | 37 | 39 | 44
  Week 48 | -6.7 (0.42) | -6.4 (0.43) | -5.8 (0.42) | -5.6 (0.40)
  Week 49: number analyzed (Participants) | 38 | 35 | 36 | 43
  Week 49 | -6.7 (0.44) | -6.3 (0.46) | -5.6 (0.46) | -5.8 (0.42)
  Week 50: number analyzed (Participants) | 36 | 35 | 36 | 39
  Week 50 | -6.8 (0.45) | -6.2 (0.46) | -5.9 (0.46) | -5.7 (0.44)
  Week 51: number analyzed (Participants) | 36 | 31 | 36 | 39
  Week 51 | -6.6 (0.44) | -6.5 (0.48) | -6.0 (0.44) | -5.5 (0.43)
  Week 52: number analyzed (Participants) | 36 | 30 | 36 | 40
  Week 52 | -6.8 (0.45) | -6.2 (0.49) | -5.6 (0.45) | -5.7 (0.43)
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p < 0.0001, ANCOVA — Estimated from ANCOVA models with treatment and randomization stratification factors of sex and years since the first nodule observed ( ≥ 10 vs. <10 years) as fixed effect factors, baseline as covariate; LS Mean Difference = -1.2, 95% CI 2-sided [-1.8 to -0.7], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p = 0.0287, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.2 to -0.1], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p = 0.1123, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.0 to 0.1], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.1, 95% CI 2-sided [-3.0 to -1.3], Standard Error of Mean 0.41
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0044, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.0 to -0.4], Standard Error of Mean 0.41
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0046, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.0 to -0.4], Standard Error of Mean 0.41
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.7, 95% CI 2-sided [-3.6 to -1.8], Standard Error of Mean 0.44
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p = 0.0011, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-2.3 to -0.6], Standard Error of Mean 0.44
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p = 0.0171, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-1.9 to -0.2], Standard Error of Mean 0.44
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -2.1], Standard Error of Mean 0.46
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.7, 95% CI 2-sided [-2.6 to -0.8], Standard Error of Mean 0.46
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.1146, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.6 to 0.2], Standard Error of Mean 0.46
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.2, 95% CI 2-sided [-4.2 to -2.3], Standard Error of Mean 0.46
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.1, 95% CI 2-sided [-3.0 to -1.2], Standard Error of Mean 0.46
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p = 0.0087, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.1 to -0.3], Standard Error of Mean 0.46
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.3, 95% CI 2-sided [-4.3 to -2.4], Standard Error of Mean 0.48
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.4, 95% CI 2-sided [-3.3 to -1.4], Standard Error of Mean 0.47
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p = 0.0013, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-2.5 to -0.6], Standard Error of Mean 0.47
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.4, 95% CI 2-sided [-4.4 to -2.4], Standard Error of Mean 0.50
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.6, 95% CI 2-sided [-3.6 to -1.6], Standard Error of Mean 0.49
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p = 0.0048, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.4 to -0.4], Standard Error of Mean 0.50
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.5, 95% CI 2-sided [-4.5 to -2.4], Standard Error of Mean 0.51
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.6, 95% CI 2-sided [-3.6 to -1.6], Standard Error of Mean 0.51
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0124, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.3 to -0.3], Standard Error of Mean 0.51
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.5, 95% CI 2-sided [-4.5 to -2.5], Standard Error of Mean 0.53
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.8, 95% CI 2-sided [-3.8 to -1.7], Standard Error of Mean 0.52
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p = 0.0021, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.6, 95% CI 2-sided [-2.7 to -0.6], Standard Error of Mean 0.52
Statistical Analysis 28: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.5, 95% CI 2-sided [-4.6 to -2.4], Standard Error of Mean 0.55
Statistical Analysis 29: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -1.9], Standard Error of Mean 0.54
Statistical Analysis 30: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p = 0.0005, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-3.0 to -0.9], Standard Error of Mean 0.54
Statistical Analysis 31: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.5, 95% CI 2-sided [-4.6 to -2.4], Standard Error of Mean 0.56
Statistical Analysis 32: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.0, 95% CI 2-sided [-4.1 to -1.8], Standard Error of Mean 0.56
Statistical Analysis 33: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Other; p = 0.0044, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.6, 95% CI 2-sided [-2.7 to -0.5], Standard Error of Mean 0.56
Statistical Analysis 34: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.6, 95% CI 2-sided [-4.7 to -2.4], Standard Error of Mean 0.57
Statistical Analysis 35: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.7, 95% CI 2-sided [-3.8 to -1.6], Standard Error of Mean 0.56
Statistical Analysis 36: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0231, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.4 to -0.2], Standard Error of Mean 0.56
Statistical Analysis 37: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.3, 95% CI 2-sided [-4.5 to -2.2], Standard Error of Mean 0.57
Statistical Analysis 38: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.8, 95% CI 2-sided [-4.0 to -1.7], Standard Error of Mean 0.57
Statistical Analysis 39: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p = 0.0074, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-2.7 to -0.4], Standard Error of Mean 0.57
Statistical Analysis 40: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.6, 95% CI 2-sided [-4.8 to -2.5], Standard Error of Mean 0.58
Statistical Analysis 41: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.2, 95% CI 2-sided [-4.3 to -2.1], Standard Error of Mean 0.58
Statistical Analysis 42: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p = 0.0013, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-3.0 to -0.7], Standard Error of Mean 0.58
Statistical Analysis 43: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.7, 95% CI 2-sided [-4.8 to -2.6], Standard Error of Mean 0.57
Statistical Analysis 44: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.2, 95% CI 2-sided [-4.3 to -2.1], Standard Error of Mean 0.57
Statistical Analysis 45: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p = 0.0010, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-3.0 to -0.8], Standard Error of Mean 0.57
Statistical Analysis 46: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.6, 95% CI 2-sided [-4.8 to -2.5], Standard Error of Mean 0.57
Statistical Analysis 47: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.1, 95% CI 2-sided [-4.2 to -2.0], Standard Error of Mean 0.57
Statistical Analysis 48: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0040, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.7, 95% CI 2-sided [-2.8 to -0.5], Standard Error of Mean 0.57
Statistical Analysis 49: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -3.1, 95% CI 2-sided [-4.2 to -1.9], Standard Error of Mean 0.59
Statistical Analysis 50: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.7, 95% CI 2-sided [-3.9 to -1.6], Standard Error of Mean 0.60
Statistical Analysis 51: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p = 0.0087, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.6, 95% CI 2-sided [-2.7 to -0.4], Standard Error of Mean 0.59
Statistical Analysis 52: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.6, 95% CI 2-sided [-3.8 to -1.4], Standard Error of Mean 0.60
Statistical Analysis 53: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0003, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.2, 95% CI 2-sided [-3.4 to -1.0], Standard Error of Mean 0.60
Statistical Analysis 54: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.359, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.4 to -0.1], Standard Error of Mean 0.59
Statistical Analysis 55: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.0005, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.1, 95% CI 2-sided [-3.3 to -0.9], Standard Error of Mean 0.60
Statistical Analysis 56: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.0027, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-3.1 to -0.6], Standard Error of Mean 0.61
Statistical Analysis 57: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.0657, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.3 to 0.1], Standard Error of Mean 0.60
Statistical Analysis 58: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0021, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-3.1 to -0.7], Standard Error of Mean 0.60
Statistical Analysis 59: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0172, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-2.7 to -0.3], Standard Error of Mean 0.61
Statistical Analysis 60: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.1344, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-2.1 to -0.3], Standard Error of Mean 0.60
Statistical Analysis 61: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.0134, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-2.7 to -0.3], Standard Error of Mean 0.61
Statistical Analysis 62: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.0260, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.6 to -0.2], Standard Error of Mean 0.62
Statistical Analysis 63: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.2150, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.9 to 0.4], Standard Error of Mean 0.60
Statistical Analysis 64: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.0271, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.6 to -0.2], Standard Error of Mean 0.62
Statistical Analysis 65: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.0502, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.5 to 0.0], Standard Error of Mean 0.62
Statistical Analysis 66: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.4138, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.7], Standard Error of Mean 0.61
Statistical Analysis 67: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.0738, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.4 to 0.1], Standard Error of Mean 0.63
Statistical Analysis 68: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.1247, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.2 to 0.3], Standard Error of Mean 0.63
Statistical Analysis 69: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.4572, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.8], Standard Error of Mean 0.61
Statistical Analysis 70: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.0617, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.4 to 0.1], Standard Error of Mean 0.62
Statistical Analysis 71: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.677, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.4 to 0.1], Standard Error of Mean 0.63
Statistical Analysis 72: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.4688, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.7 to 0.8], Standard Error of Mean 0.61
Statistical Analysis 73: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.1093, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.2 to 0.2], Standard Error of Mean 0.62
Statistical Analysis 74: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.1196, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.2 to 0.3], Standard Error of Mean 0.62
Statistical Analysis 75: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.5763, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-1.5 to 0.9], Standard Error of Mean 0.61
Statistical Analysis 76: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.0661, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.4 to 0.1], Standard Error of Mean 0.62
Statistical Analysis 77: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.0622, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.4 to 0.1], Standard Error of Mean 0.62
Statistical Analysis 78: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.4677, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.6 to 0.8], Standard Error of Mean 0.61
Statistical Analysis 79: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.0854, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.2 to 0.1], Standard Error of Mean 0.61
Statistical Analysis 80: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.0768, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.3 to 0.1], Standard Error of Mean 0.62
Statistical Analysis 81: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.2560, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.9 to 0.5], Standard Error of Mean 0.60
Statistical Analysis 82: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.0337, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.5 to -0.1], Standard Error of Mean 0.61
Statistical Analysis 83: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.0778, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.3 to 0.1], Standard Error of Mean 0.62
Statistical Analysis 84: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.3218, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.8 to 0.6], Standard Error of Mean 0.61
Statistical Analysis 85: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.0549, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.3 to 0.0], Standard Error of Mean 0.59
Statistical Analysis 86: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.0543, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.4 to 0.0], Standard Error of Mean 0.60
Statistical Analysis 87: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.3759, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.6], Standard Error of Mean 0.59
Statistical Analysis 88: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.0286, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.5 to -0.1], Standard Error of Mean 0.60
Statistical Analysis 89: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.0477, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.4 to 0.0], Standard Error of Mean 0.61
Statistical Analysis 90: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.2699, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.8 to 0.5], Standard Error of Mean 0.60
Statistical Analysis 91: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.0294, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.5 to -0.1], Standard Error of Mean 0.60
Statistical Analysis 92: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.0702, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.3 to 0.1], Standard Error of Mean 0.60
Statistical Analysis 93: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.3636, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.6], Standard Error of Mean 0.59
Statistical Analysis 94: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.0273, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.5 to -0.1], Standard Error of Mean 0.59
Statistical Analysis 95: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.0785, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.2 to 0.1], Standard Error of Mean 0.59
Statistical Analysis 96: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.4111, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.6 to 0.7], Standard Error of Mean 0.59
Statistical Analysis 97: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.0471, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.4 to 0.0], Standard Error of Mean 0.60
Statistical Analysis 98: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.0891, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.2 to 0.2], Standard Error of Mean 0.59
Statistical Analysis 99: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.4820, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.6 to 0.7], Standard Error of Mean 0.58
Statistical Analysis 100: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.0222, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.6 to -0.2], Standard Error of Mean 0.60
Statistical Analysis 101: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.0682, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.3 to 0.1], Standard Error of Mean 0.60
Statistical Analysis 102: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.4112, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.7], Standard Error of Mean 0.59
Statistical Analysis 103: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.0307, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.5 to -0.1], Standard Error of Mean 0.60
Statistical Analysis 104: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.1538, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-2.0 to 0.3], Standard Error of Mean 0.60
Statistical Analysis 105: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.4047, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.7], Standard Error of Mean 0.59
Statistical Analysis 106: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.0260, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.5 to -0.2], Standard Error of Mean 0.60
Statistical Analysis 107: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.1223, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-2.1 to 0.3], Standard Error of Mean 0.60
Statistical Analysis 108: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.3641, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.6], Standard Error of Mean 0.59
Statistical Analysis 109: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.0284, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.6 to -0.1], Standard Error of Mean 0.61
Statistical Analysis 110: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.1534, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-2.1 to 0.3], Standard Error of Mean 0.61
Statistical Analysis 111: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.3914, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.7], Standard Error of Mean 0.59
Statistical Analysis 112: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.0265, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.6 to -0.2], Standard Error of Mean 0.61
Statistical Analysis 113: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.1682, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-2.0 to 0.4], Standard Error of Mean 0.60
Statistical Analysis 114: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.4699, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.6 to 0.7], Standard Error of Mean 0.59
Statistical Analysis 115: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.0241, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.5 to -0.2], Standard Error of Mean 0.59
Statistical Analysis 116: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.1064, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.1 to 0.2], Standard Error of Mean 0.1064
Statistical Analysis 117: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.2948, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.7 to 0.5], Standard Error of Mean 0.58
Statistical Analysis 118: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.0282, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.5 to -0.1], Standard Error of Mean 0.59
Statistical Analysis 119: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.1074, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.1 to 0.2], Standard Error of Mean 0.59
Statistical Analysis 120: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.3061, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.7 to 0.5], Standard Error of Mean 0.58
Statistical Analysis 121: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.0705, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.2 to 0.1], Standard Error of Mean 0.59
Statistical Analysis 122: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.2405, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.9 to 0.5], Standard Error of Mean 0.59
Statistical Analysis 123: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.3726, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.6], Standard Error of Mean 0.58
Statistical Analysis 124: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.0554, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.3 to 0.0], Standard Error of Mean 0.58
Statistical Analysis 125: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.2386, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.8 to 0.5], Standard Error of Mean 0.58
Statistical Analysis 126: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.5147, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.5 to 0.8], Standard Error of Mean 0.57
Statistical Analysis 127: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.1116, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-2.1 to 0.2], Standard Error of Mean 0.58
Statistical Analysis 128: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.1266, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-2.0 to 0.3], Standard Error of Mean 0.58
Statistical Analysis 129: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.3822, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.6 to 0.6], Standard Error of Mean 0.57
Statistical Analysis 130: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.0720, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.2 to 0.1], Standard Error of Mean 0.59
Statistical Analysis 131: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.3434, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.7 to 0.6], Standard Error of Mean 0.58
Statistical Analysis 132: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.5061, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.5 to 0.8], Standard Error of Mean 0.58
Statistical Analysis 133: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.0366, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.2, 95% CI 2-sided [-2.3 to -0.1], Standard Error of Mean 0.57
Statistical Analysis 134: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.1181, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-2.0 to 0.2], Standard Error of Mean 0.57
Statistical Analysis 135: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.7078, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.3 to 0.9], Standard Error of Mean 0.56
Statistical Analysis 136: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.0868, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.1 to 0.1], Standard Error of Mean 0.58
Statistical Analysis 137: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.1683, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-1.9 to 0.3], Standard Error of Mean 0.57
Statistical Analysis 138: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.8909, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-1.2 to 1.1], Standard Error of Mean 0.57
Statistical Analysis 139: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Other; p = 0.0671, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.3 to 0.1], Standard Error of Mean 0.59
Statistical Analysis 140: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Superiority; p = 0.3325, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.7 to 0.6], Standard Error of Mean 0.59
Statistical Analysis 141: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Other; p = 0.8912, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-1.2 to 1.1], Standard Error of Mean 0.59
Statistical Analysis 142: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.0612, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.2 to 0.1], Standard Error of Mean 0.58
Statistical Analysis 143: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.1879, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-1.9 to 0.4], Standard Error of Mean 0.58
Statistical Analysis 144: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.7696, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.3 to 1.0], Standard Error of Mean 0.58
Statistical Analysis 145: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.1211, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-2.1 to 0.2], Standard Error of Mean 0.60
Statistical Analysis 146: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.3908, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.7], Standard Error of Mean 0.61
Statistical Analysis 147: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.8036, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-1.1 to 1.4], Standard Error of Mean 0.61
Statistical Analysis 148: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.0928, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.3 to 0.2], Standard Error of Mean 0.63
Statistical Analysis 149: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.4439, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = 0.63, 95% CI 2-sided [-1.7 to 0.8], Standard Error of Mean 0.63
Statistical Analysis 150: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.7769, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.4 to 1.1], Standard Error of Mean 0.63
Statistical Analysis 151: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.0742, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.3 to 0.1], Standard Error of Mean 0.61
Statistical Analysis 152: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.1496, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-2.2 to 0.3], Standard Error of Mean 0.63
Statistical Analysis 153: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.4901, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.6 to 0.8], Standard Error of Mean 0.61
Statistical Analysis 154: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.0895, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.3 to 0.2], Standard Error of Mean 0.62
Statistical Analysis 155: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.4572, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.8 to 0.8], Standard Error of Mean 0.65
Statistical Analysis 156: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.8157, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-1.1 to 1.4], Standard Error of Mean 0.62

29. Secondary Outcome: Phase 2b: Percent Change From Baseline in Weekly Average of WI-NRS Over Time
Description: as for outcome 5
Time Frame: Baseline, Weeks 1 through 52
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage change
  Week 1 | -19.6 (2.56) | -12.5 (2.56) | -10.0 (2.60) | -5.1 (2.53)
  Week 2: number analyzed (Participants) | 46 | 47 | 47 | 48
  Week 2 | -33.2 (3.60) | -21.9 (3.57) | -21.4 (3.62) | -7.9 (3.52)
  Week 3 | -40.2 (3.83) | -25.4 (3.83) | -19.9 (3.88) | -8.2 (3.78)
  Week 4: number analyzed (Participants) | 46 | 47 | 47 | 48
  Week 4 | -45.1 (4.00) | -29.7 (3.96) | -16.9 (4.01) | -9.1 (3.91)
  Week 5: number analyzed (Participants) | 46 | 47 | 47 | 48
  Week 5 | -47.8 (3.98) | -34.2 (3.94) | -23.2 (3.99) | -9.6 (3.89)
  Week 6: number analyzed (Participants) | 45 | 47 | 47 | 48
  Week 6 | -49.5 (4.10) | -38.2 (4.02) | -28.0 (4.08) | -10.5 (3.97)
  Week 7: number analyzed (Participants) | 45 | 47 | 47 | 47
  Week 7 | -50.1 (4.26) | -41.3 (4.18) | -27.1 (4.24) | -11.0 (4.17)
  Week 8: number analyzed (Participants) | 45 | 47 | 47 | 47
  Week 8 | -51.7 (4.39) | -42.1 (4.30) | -26.0 (4.37) | -11.7 (4.30)
  Week 9: number analyzed (Participants) | 45 | 47 | 47 | 47
  Week 9 | -54.0 (4.58) | -45.9 (4.48) | -31.1 (4.55) | -13.3 (4.48)
  Week 10: number analyzed (Participants) | 45 | 46 | 47 | 46
  Week 10 | -55.0 (4.63) | -49.4 (4.59) | -36.0 (4.61) | -14.3 (4.58)
  Week 11: number analyzed (Participants) | 45 | 45 | 47 | 46
  Week 11 | -55.2 (4.77) | -49.5 (4.79) | -32.5 (4.75) | -14.3 (4.72)
  Week 12: number analyzed (Participants) | 45 | 45 | 47 | 46
  Week 12 | -56.0 (4.76) | -46.8 (4.78) | -29.2 (4.74) | -14.6 (4.71)
  Week 13: number analyzed (Participants) | 45 | 45 | 47 | 46
  Week 13 | -56.6 (4.80) | -51.6 (4.82) | -35.6 (4.78) | -17.9 (4.74)
  Week 14: number analyzed (Participants) | 45 | 45 | 47 | 46
  Week 14 | -57.1 (4.91) | -52.9 (4.93) | -36.7 (4.89) | -15.3 (4.85)
  Week 15: number analyzed (Participants) | 45 | 45 | 47 | 46
  Week 15 | -57.5 (4.81) | -52.1 (4.83) | -36.2 (4.79) | -14.9 (4.75)
  Week 16: number analyzed (Participants) | 45 | 45 | 47 | 47
  Week 16 | -56.5 (4.88) | -51.2 (4.90) | -33.3 (4.85) | -14.8 (4.77)
  Week 17: number analyzed (Participants) | 45 | 43 | 46 | 46
  Week 17 | -60.3 (5.02) | -57.2 (5.14) | -43.0 (5.04) | -25.1 (4.98)
  Week 18: number analyzed (Participants) | 45 | 42 | 47 | 46
  Week 18 | -61.3 (5.03) | -57.9 (5.20) | -45.5 (5.00) | -31.4 (4.99)
  Week 19: number analyzed (Participants) | 45 | 42 | 46 | 46
  Week 19 | -62.3 (5.06) | -59.9 (5.24) | -50.8 (5.08) | -38.1 (5.02)
  Week 20: number analyzed (Participants) | 45 | 42 | 47 | 46
  Week 20 | -62.2 (5.10) | -58.2 (5.27) | -50.9 (5.07) | -40.6 (5.06)
  Week 21: number analyzed (Participants) | 43 | 41 | 47 | 46
  Week 21 | -63.1 (5.23) | -62.2 (5.37) | -54.3 (5.09) | -45.7 (5.07)
  Week 22: number analyzed (Participants) | 42 | 41 | 47 | 46
  Week 22 | -63.3 (5.32) | -62.3 (5.40) | -53.3 (5.12) | -47.4 (5.10)
  Week 23: number analyzed (Participants) | 41 | 41 | 47 | 46
  Week 23 | -63.7 (5.47) | -62.7 (5.49) | -56.2 (5.21) | -50.6 (5.18)
  Week 24: number analyzed (Participants) | 42 | 41 | 46 | 48
  Week 24 | -64.2 (5.39) | -64.3 (7.41) | -55.6 (5.23) | -50.5 (5.16)
  Week 25: number analyzed (Participants) | 41 | 41 | 45 | 45
  Week 25 | -64.8 (5.35) | -65.0 (5.37) | -57.2 (5.18) | -53.0 (5.13)
  Week 26: number analyzed (Participants) | 42 | 40 | 45 | 46
  Week 26 | -65.4 (5.30) | -66.2 (5.44) | -57.4 (5.19) | -51.8 (5.08)
  Week 27: number analyzed (Participants) | 42 | 39 | 43 | 46
  Week 27 | -64.2 (5.25) | -65.3 (5.46) | -59.7 (5.23) | -51.9 (5.03)
  Week 28: number analyzed (Participants) | 41 | 40 | 41 | 46
  Week 28 | -67.1 (5.31) | -65.0 (5.40) | -58.3 (5.35) | -51.6 (5.03)
  Week 29: number analyzed (Participants) | 41 | 39 | 43 | 45
  Week 29 | -67.8 (5.17) | -68.4 (5.30) | -59.9 (5.10) | -54.1 (4.95)
  Week 30: number analyzed (Participants) | 41 | 39 | 43 | 46
  Week 30 | -68.5 (5.25) | -67.5 (5.39) | -60.3 (5.18) | -52.7 (4.98)
  Week 31: number analyzed (Participants) | 40 | 39 | 43 | 45
  Week 31 | -70.8 (5.23) | -68.5 (5.30) | -61.3 (5.09) | -55.1 (4.95)
  Week 32: number analyzed (Participants) | 40 | 40 | 42 | 46
  Week 32 | -70.7 (5.21) | -67.9 (5.21) | -60.3 (5.12) | -54.9 (4.88)
  Week 33: number analyzed (Participants) | 39 | 40 | 44 | 46
  Week 33 | -70.3 (5.26) | -68.3 (5.19) | -60.5 (5.00) | -56.1 (4.85)
  Week 34: number analyzed (Participants) | 40 | 40 | 43 | 46
  Week 34 | -72.2 (5.31) | -68.9 (5.30) | -60.4 (5.16) | -55.5 (4.96)
  Week 35: number analyzed (Participants) | 39 | 40 | 43 | 46
  Week 35 | -72.3 (5.29) | -67.2 (5.23) | -61.8 (5.10) | -56.5 (4.90)
  Week 36: number analyzed (Participants) | 39 | 39 | 44 | 46
  Week 36 | -72.7 (5.27) | -68.2 (5.29) | -62.5 (5.03) | -56.3 (4.88)
  Week 37: number analyzed (Participants) | 38 | 39 | 44 | 45
  Week 37 | -73.9 (5.34) | -68.8 (5.30) | -64.0 (5.04) | -58.0 (4.96)
  Week 38: number analyzed (Participants) | 38 | 39 | 44 | 44
  Week 38 | -75.2 (5.29) | -69.5 (5.25) | -63.6 (4.99) | -59.1 (4.97)
  Week 39: number analyzed (Participants) | 38 | 38 | 43 | 45
  Week 39 | -75.2 (5.23) | -71.0 (5.27) | -65.7 (5.02) | -59.3 (4.87)
  Week 40 | -75.1 (5.24) | -71.4 (5.28) | -65.9 (5.02) | -59.6 (4.87)
  Week 41: number analyzed (Participants) | 38 | 38 | 41 | 44
  Week 41 | -74.7 (5.17) | -70.8 (5.21) | -68.3 (5.05) | -62.3 (4.88)
  Week 42: number analyzed (Participants) | 38 | 37 | 41 | 43
  Week 42 | -75.8 (5.05) | -71.2 (5.15) | -67.0 (4.93) | -62.7 (4.82)
  Week 43: number analyzed (Participants) | 37 | 38 | 40 | 43
  Week 43 | -72.9 (5.08) | -73.0 (5.06) | -68.0 (4.96) | -62.1 (4.78)
  Week 44: number analyzed (Participants) | 37 | 37 | 40 | 43
  Week 44 | -75.6 (5.08) | -70.5 (5.15) | -67.8 (4.97) | -63.4 (4.80)
  Week 45: number analyzed (Participants) | 38 | 37 | 40 | 43
  Week 45 | -76.9 (4.92) | -73.7 (5.05) | -65.4 (4.86) | -62.8 (4.71)
  Week 46: number analyzed (Participants) | 38 | 38 | 40 | 43
  Week 46 | -76.0 (4.99) | -74.0 (5.02) | -65.2 (4.92) | -64.3 (4.76)
  Week 47: number analyzed (Participants) | 38 | 38 | 40 | 43
  Week 47 | -78.0 (5.09) | -72.4 (5.13) | -66.1 (5.02) | -65.2 (4.86)
  Week 48: number analyzed (Participants) | 38 | 37 | 39 | 44
  Week 48 | -77.6 (4.99) | -74.4 (5.09) | -66.8 (5.00) | -64.9 (4.71)
  Week 49: number analyzed (Participants) | 38 | 35 | 36 | 43
  Week 49 | -78.2 (5.15) | -73.8 (5.40) | -65.5 (5.37) | -67.3 (4.92)
  Week 50: number analyzed (Participants) | 36 | 35 | 36 | 39
  Week 50 | -78.7 (5.30) | -72.8 (5.40) | -68.8 (5.36) | -66.8 (5.16)
  Week 51: number analyzed (Participants) | 36 | 31 | 36 | 39
  Week 51 | -77.3 (5.23) | -75.7 (5.66) | -69.4 (5.25) | -64.6 (5.08)
  Week 52: number analyzed (Participants) | 36 | 30 | 36 | 40
  Week 52 | -79.1 (5.27) | -72.8 (5.76) | -64.8 (5.33) | -67.0 (5.08)
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -14.5, 95% CI 2-sided [-21.6 to -7.5], Standard Error of Mean 3.57
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p = 0.0368, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -7.5, 95% CI 2-sided [-14.5 to -0.5], Standard Error of Mean 3.56
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p = 0.1700, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -4.9, 95% CI 2-sided [-12.0 to 2.1], Standard Error of Mean 3.58
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -25.2, 95% CI 2-sided [-35.1 to -15.3], Standard Error of Mean 5.00
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0056, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.9, 95% CI 2-sided [-23.7 to -4.1], Standard Error of Mean 4.96
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0076, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.5, 95% CI 2-sided [-23.3 to -3.6], Standard Error of Mean 4.99
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -32.0, 95% CI 2-sided [-42.5 to -21.5], Standard Error of Mean 5.33
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p = 0.0014, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -17.2, 95% CI 2-sided [-27.7 to -6.7], Standard Error of Mean 5.32
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p = 0.0296, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -11.7, 95% CI 2-sided [-22.3 to -1.2], Standard Error of Mean 5.35
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -35.9, 95% CI 2-sided [-46.9 to -25.0], Standard Error of Mean 5.54
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -20.6, 95% CI 2-sided [-31.4 to -9.7], Standard Error of Mean 5.50
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.1652, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -7.7, 95% CI 2-sided [-18.6 to 3.2], Standard Error of Mean 5.53
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -38.2, 95% CI 2-sided [-49.1 to -27.3], Standard Error of Mean 5.52
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -24.5, 95% CI 2-sided [-35.3 to -13.7], Standard Error of Mean 5.47
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p = 0.0146, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.6, 95% CI 2-sided [-24.5 to -2.7], Standard Error of Mean 5.51
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -39.0, 95% CI 2-sided [-50.2 to -27.8], Standard Error of Mean 5.66
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -27.7, 95% CI 2-sided [-38.8 to -16.7], Standard Error of Mean 5.59
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p = 0.0022, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -17.5, 95% CI 2-sided [-28.5 to -6.4], Standard Error of Mean 5.62
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -39.1, 95% CI 2-sided [-50.8 to -27.4], Standard Error of Mean 5.92
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -30.3, 95% CI 2-sided [-41.8 to -18.8], Standard Error of Mean 5.84
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p = 0.0069, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -16.1, 95% CI 2-sided [-27.7 to -4.5], Standard Error of Mean 5.87
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -40.1, 95% CI 2-sided [-52.1 to -28.0], Standard Error of Mean 6.09
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -30.4, 95% CI 2-sided [-42.3 to -18.5], Standard Error of Mean 6.01
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0194, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -14.3, 95% CI 2-sided [-26.2 to -2.3], Standard Error of Mean 6.05
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -40.6, 95% CI 2-sided [-53.2 to -28.1], Standard Error of Mean 6.35
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -32.5, 95% CI 2-sided [-44.9 to -20.1], Standard Error of Mean 6.27
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p = 0.0054, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -17.8, 95% CI 2-sided [-30.2 to -5.3], Standard Error of Mean 6.30
Statistical Analysis 28: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -40.7, 95% CI 2-sided [-53.4 to -27.9], Standard Error of Mean 6.46
Statistical Analysis 29: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -35.1, 95% CI 2-sided [-47.8 to -22.5], Standard Error of Mean 6.41
Statistical Analysis 30: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p = 0.0009, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -21.8, 95% CI 2-sided [-34.4 to -9.1], Standard Error of Mean 6.42
Statistical Analysis 31: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -40.9, 95% CI 2-sided [-54.1 to -27.8], Standard Error of Mean 6.66
Statistical Analysis 32: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -35.2, 95% CI 2-sided [-48.3 to -22.1], Standard Error of Mean 6.64
Statistical Analysis 33: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p = 0.0067, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -18.2, 95% CI 2-sided [-31.2 to -5.1], Standard Error of Mean 6.61
Statistical Analysis 34: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -41.3, 95% CI 2-sided [-54.5 to -28.2], Standard Error of Mean 6.64
Statistical Analysis 35: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -32.2, 95% CI 2-sided [-45.3 to -19.1], Standard Error of Mean 6.63
Statistical Analysis 36: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0279, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -14.6, 95% CI 2-sided [-27.6 to -1.6], Standard Error of Mean 6.60
Statistical Analysis 37: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -38.7, 95% CI 2-sided [-51.9 to -25.4], Standard Error of Mean 6.70
Statistical Analysis 38: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -33.7, 95% CI 2-sided [-46.7 to -20.5], Standard Error of Mean 6.69
Statistical Analysis 39: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p = 0.0085, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -17.7, 95% CI 2-sided [-30.8 to -4.6], Standard Error of Mean 6.65
Statistical Analysis 40: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -41.9, 95% CI 2-sided [-55.4 to -28.4], Standard Error of Mean 6.85
Statistical Analysis 41: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -37.6, 95% CI 2-sided [-51.1 to -24.1], Standard Error of Mean 6.84
Statistical Analysis 42: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p = 0.0020, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -21.4, 95% CI 2-sided [-34.8 to -8.0], Standard Error of Mean 6.80
Statistical Analysis 43: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -42.7, 95% CI 2-sided [-55.9 to -29.4], Standard Error of Mean 6.72
Statistical Analysis 44: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -37.2, 95% CI 2-sided [-50.4 to -24.0], Standard Error of Mean 6.70
Statistical Analysis 45: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p = 0.0016, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -21.4, 95% CI 2-sided [-34.5 to -8.2], Standard Error of Mean 6.67
Statistical Analysis 46: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -41.6, 95% CI 2-sided [-55.0 to -28.3], Standard Error of Mean 6.77
Statistical Analysis 47: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -36.4, 95% CI 2-sided [-49.7 to -23.1], Standard Error of Mean 6.75
Statistical Analysis 48: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0067, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -18.4, 95% CI 2-sided [-31.7 to -5.2], Standard Error of Mean 6.72
Statistical Analysis 49: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -35.2, 95% CI 2-sided [-49.0 to -21.4], Standard Error of Mean 7.00
Statistical Analysis 50: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -32.1, 95% CI 2-sided [-46.0 to -18.1], Standard Error of Mean 7.07
Statistical Analysis 51: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p = 0.0111, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -17.9, 95% CI 2-sided [-31.7 to -4.1], Standard Error of Mean 6.98
Statistical Analysis 52: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -29.9, 95% CI 2-sided [-43.8 to -16.1], Standard Error of Mean 7.02
Statistical Analysis 53: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0003, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -26.6, 95% CI 2-sided [-40.6 to -12.5], Standard Error of Mean 7.12
Statistical Analysis 54: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0445, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -14.1, 95% CI 2-sided [-27.8 to -0.4], Standard Error of Mean 6.96
Statistical Analysis 55: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.0008, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -24.2, 95% CI 2-sided [-38.1 to -10.2], Standard Error of Mean 7.06
Statistical Analysis 56: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.0027, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -21.8, 95% CI 2-sided [-36.0 to -7.7], Standard Error of Mean 7.17
Statistical Analysis 57: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.0724, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.7, 95% CI 2-sided [-26.7 to 1.2], Standard Error of Mean 7.05
Statistical Analysis 58: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0028, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -21.6, 95% CI 2-sided [-35.7 to -7.6], Standard Error of Mean 7.11
Statistical Analysis 59: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0158, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -17.6, 95% CI 2-sided [-31.9 to -3.3], Standard Error of Mean 7.22
Statistical Analysis 60: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.1468, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -10.3, 95% CI 2-sided [-24.2 to 3.6], Standard Error of Mean 7.06
Statistical Analysis 61: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.0167, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -17.4, 95% CI 2-sided [-31.7 to -3.2], Standard Error of Mean 7.21
Statistical Analysis 62: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.0242, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -16.6, 95% CI 2-sided [-31.0 to -2.2], Standard Error of Mean 7.29
Statistical Analysis 63: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.2240, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -8.6, 95% CI 2-sided [-22.6 to 5.3], Standard Error of Mean 7.08
Statistical Analysis 64: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.0310, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -15.9, 95% CI 2-sided [-30.3 to -1.5], Standard Error of Mean 7.30
Statistical Analysis 65: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.0437, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -14.9, 95% CI 2-sided [-29.4 to -0.4], Standard Error of Mean 7.33
Statistical Analysis 66: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.4123, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -5.9, 95% CI 2-sided [-19.9 to 8.2], Standard Error of Mean 7.12
Statistical Analysis 67: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.0808, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.1, 95% CI 2-sided [-27.8 to 1.6], Standard Error of Mean 7.46
Statistical Analysis 68: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.1064, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.1, 95% CI 2-sided [-26.8 to 2.6], Standard Error of Mean 7.45
Statistical Analysis 69: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.4366, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -5.6, 95% CI 2-sided [-19.9 to 8.6], Standard Error of Mean 7.24
Statistical Analysis 70: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.0644, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.8, 95% CI 2-sided [-28.3 to 0.8], Standard Error of Mean 7.39
Statistical Analysis 71: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.0633, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.9, 95% CI 2-sided [-28.5 to 0.8], Standard Error of Mean 7.41
Statistical Analysis 72: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.4775, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -5.2, 95% CI 2-sided [-19.4 to 9.1], Standard Error of Mean 7.23
Statistical Analysis 73: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.1106, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -11.8, 95% CI 2-sided [-26.2 to 2.7], Standard Error of Mean 7.33
Statistical Analysis 74: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.1043, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.0, 95% CI 2-sided [-26.4 to 2.5], Standard Error of Mean 7.32
Statistical Analysis 75: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.5630, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -4.2, 95% CI 2-sided [-18.4 to 10.0], Standard Error of Mean 7.19
Statistical Analysis 76: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.0629, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.6, 95% CI 2-sided [-27.9 to 0.7], Standard Error of Mean 7.26
Statistical Analysis 77: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.0523, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -14.3, 95% CI 2-sided [-28.8 to 0.1], Standard Error of Mean 7.34
Statistical Analysis 78: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.4420, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -5.5, 95% CI 2-sided [-19.6 to 8.6], Standard Error of Mean 7.15
Statistical Analysis 79: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.0908, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.2, 95% CI 2-sided [-26.4 to 2.0], Standard Error of Mean 7.19
Statistical Analysis 80: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.0688, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.4, 95% CI 2-sided [-27.9 to 1.0], Standard Error of Mean 7.32
Statistical Analysis 81: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.2802, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -7.8, 95% CI 2-sided [-21.9 to 6.4], Standard Error of Mean 7.17
Statistical Analysis 82: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.0337, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -15.5, 95% CI 2-sided [-29.8 to -1.2], Standard Error of Mean 7.24
Statistical Analysis 83: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.0673, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.4, 95% CI 2-sided [-27.8 to 1.0], Standard Error of Mean 7.28
Statistical Analysis 84: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.3564, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -6.7, 95% CI 2-sided [-21.1 to 7.6], Standard Error of Mean 7.27
Statistical Analysis 85: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.0558, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.6, 95% CI 2-sided [-27.6 to 0.3], Standard Error of Mean 7.08
Statistical Analysis 86: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.0471, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -14.3, 95% CI 2-sided [-28.5 to -0.2], Standard Error of Mean 7.16
Statistical Analysis 87: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.4101, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -5.8, 95% CI 2-sided [-19.7 to 8.1], Standard Error of Mean 7.03
Statistical Analysis 88: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.0287, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -15.8, 95% CI 2-sided [-29.9 to -1.7], Standard Error of Mean 7.16
Statistical Analysis 89: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.0427, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -14.8, 95% CI 2-sided [-29.1 to -0.5], Standard Error of Mean 7.24
Statistical Analysis 90: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.2828, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -7.6, 95% CI 2-sided [-21.7 to 6.4], Standard Error of Mean 7.10
Statistical Analysis 91: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.0294, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -15.7, 95% CI 2-sided [-29.7 to -1.6], Standard Error of Mean 7.12
Statistical Analysis 92: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.0636, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.4, 95% CI 2-sided [-27.5 to 0.8], Standard Error of Mean 7.15
Statistical Analysis 93: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.3812, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -6.2, 95% CI 2-sided [-20.0 to 7.7], Standard Error of Mean 7.02
Statistical Analysis 94: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.0270, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -15.8, 95% CI 2-sided [-29.7 to -1.8], Standard Error of Mean 7.06
Statistical Analysis 95: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.0679, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.9, 95% CI 2-sided [-26.9 to 1.0], Standard Error of Mean 7.04
Statistical Analysis 96: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.4452, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -5.4, 95% CI 2-sided [-19.2 to 8.5], Standard Error of Mean 7.00
Statistical Analysis 97: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.0467, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -14.2, 95% CI 2-sided [-28.2 to -0.2], Standard Error of Mean 7.08
Statistical Analysis 98: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.0829, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.2, 95% CI 2-sided [-26.1 to 1.6], Standard Error of Mean 7.01
Statistical Analysis 99: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.5263, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -4.4, 95% CI 2-sided [-18.0 to 9.2], Standard Error of Mean 6.89
Statistical Analysis 100: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.0210, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -16.8, 95% CI 2-sided [-31.0 to -2.6], Standard Error of Mean 7.19
Statistical Analysis 101: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.0623, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.5, 95% CI 2-sided [-27.6 to 0.7], Standard Error of Mean 7.17
Statistical Analysis 102: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.4899, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -4.9, 95% CI 2-sided [-18.9 to 9.1], Standard Error of Mean 7.08
Statistical Analysis 103: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.0281, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -15.8, 95% CI 2-sided [-29.9 to -1.7], Standard Error of Mean 7.14
Statistical Analysis 104: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.1318, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -10.7, 95% CI 2-sided [-24.7 to 3.3], Standard Error of Mean 7.08
Statistical Analysis 105: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.4458, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -5.3, 95% CI 2-sided [-19.1 to 8.5], Standard Error of Mean 6.99
Statistical Analysis 106: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.0229, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -16.3, 95% CI 2-sided [-30.4 to -2.3], Standard Error of Mean 7.11
Statistical Analysis 107: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.0978, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -11.8, 95% CI 2-sided [-25.9 to 2.2], Standard Error of Mean 7.11
Statistical Analysis 108: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.3792, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -6.1, 95% CI 2-sided [-19.8 to 7.6], Standard Error of Mean 6.93
Statistical Analysis 109: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.0290, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -15.9, 95% CI 2-sided [-30.2 to -1.7], Standard Error of Mean 7.22
Statistical Analysis 110: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.1306, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -10.9, 95% CI 2-sided [-25.0 to 3.3], Standard Error of Mean 7.15
Statistical Analysis 111: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.3923, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -6.0, 95% CI 2-sided [-19.8 to 7.8], Standard Error of Mean 6.99
Statistical Analysis 112: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.0265, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -16.1, 95% CI 2-sided [-30.3 to -1.9], Standard Error of Mean 7.19
Statistical Analysis 113: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.1456, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -10.4, 95% CI 2-sided [-24.5 to 3.6], Standard Error of Mean 7.12
Statistical Analysis 114: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.5138, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -4.6, 95% CI 2-sided [-18.3 to 9.2], Standard Error of Mean 6.96
Statistical Analysis 115: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.0265, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -15.9, 95% CI 2-sided [-29.8 to -1.9], Standard Error of Mean 7.08
Statistical Analysis 116: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.0986, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -11.7, 95% CI 2-sided [-25.7 to 2.2], Standard Error of Mean 7.05
Statistical Analysis 117: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.3600, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -6.3, 95% CI 2-sided [-20.0 to 7.3], Standard Error of Mean 6.91
Statistical Analysis 118: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.0303, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -15.5, 95% CI 2-sided [-29.5 to -1.5], Standard Error of Mean 7.09
Statistical Analysis 119: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.0979, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -11.8, 95% CI 2-sided [-25.7 to 2.2], Standard Error of Mean 7.07
Statistical Analysis 120: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.3664, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -6.3, 95% CI 2-sided [-19.9 to 7.4], Standard Error of Mean 6.92
Statistical Analysis 121: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.0806, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.4, 95% CI 2-sided [-26.3 to 1.5], Standard Error of Mean 7.04
Statistical Analysis 122: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.2260, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -8.5, 95% CI 2-sided [-22.4 to 5.3], Standard Error of Mean 7.01
Statistical Analysis 123: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.3835, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -6.0, 95% CI 2-sided [-19.7 to 7.6], Standard Error of Mean 6.92
Statistical Analysis 124: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.0594, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -13.1, 95% CI 2-sided [-26.7 to 0.5], Standard Error of Mean 6.90
Statistical Analysis 125: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.2189, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -8.5, 95% CI 2-sided [-22.2 to 5.1], Standard Error of Mean 6.91
Statistical Analysis 126: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.5238, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -4.3, 95% CI 2-sided [-17.8 to 9.1], Standard Error of Mean 6.79
Statistical Analysis 127: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.1204, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -10.8, 95% CI 2-sided [-24.5 to 2.9], Standard Error of Mean 6.92
Statistical Analysis 128: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.1129, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -10.9, 95% CI 2-sided [-24.4 to 2.6], Standard Error of Mean 6.84
Statistical Analysis 129: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.3911, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -5.9, 95% CI 2-sided [-19.3 to 7.6], Standard Error of Mean 6.81
Statistical Analysis 130: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.0784, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.3, 95% CI 2-sided [-26.0 to 1.4], Standard Error of Mean 6.93
Statistical Analysis 131: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.3046, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -7.1, 95% CI 2-sided [-20.7 to 6.5], Standard Error of Mean 6.90
Statistical Analysis 132: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.5205, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -4.4, 95% CI 2-sided [-17.9 to 9.1], Standard Error of Mean 6.82
Statistical Analysis 133: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.0388, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -14.0, 95% CI 2-sided [-27.3 to -0.7], Standard Error of Mean 6.74
Statistical Analysis 134: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.1105, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -10.8, 95% CI 2-sided [-24.2 to 2.5], Standard Error of Mean 6.75
Statistical Analysis 135: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.7039, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.5, 95% CI 2-sided [-15.7 to 10.7], Standard Error of Mean 6.68
Statistical Analysis 136: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.0885, ANCOVA — [p-value comment as in outcome 28, analysis 1]; ls = -11.7, 95% CI 2-sided [-25.2 to 1.8], Standard Error of Mean 6.82
Statistical Analysis 137: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.1535, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -9.7, 95% CI 2-sided [-23.1 to 3.7], Standard Error of Mean 6.79
Statistical Analysis 138: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.8975, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-14.2 to 12.5], Standard Error of Mean 6.76
Statistical Analysis 139: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Superiority; p = 0.0674, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.8, 95% CI 2-sided [-26.6 to 0.9], Standard Error of Mean 6.96
Statistical Analysis 140: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Superiority; p = 0.3025, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -7.2, 95% CI 2-sided [-20.8 to 6.5], Standard Error of Mean 0.3025
Statistical Analysis 141: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Superiority; p = 0.8964, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-14.5 to 12.7], Standard Error of Mean 6.90
Statistical Analysis 142: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.0633, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.7, 95% CI 2-sided [-26.1 to 0.7], Standard Error of Mean 6.79
Statistical Analysis 143: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.1665, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -9.5, 95% CI 2-sided [-22.9 to 4.0], Standard Error of Mean 6.81
Statistical Analysis 144: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.7748, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-15.3 to 11.4], Standard Error of Mean 6.78
Statistical Analysis 145: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.1239, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -10.9, 95% CI 2-sided [-24.8 to 3.0], Standard Error of Mean 7.04
Statistical Analysis 146: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.3647, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -6.5, 95% CI 2-sided [-20.7 to 7.6], Standard Error of Mean 7.17
Statistical Analysis 147: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.8056, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = 1.8, 95% CI 2-sided [-12.5 to 16.0], Standard Error of Mean 7.20
Statistical Analysis 148: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.1079, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -11.9, 95% CI 2-sided [-26.4 to 2.6], Standard Error of Mean 7.35
Statistical Analysis 149: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.4174, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -6.0, 95% CI 2-sided [-20.6 to 8.6], Standard Error of Mean 7.37
Statistical Analysis 150: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.7815, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -2.1, 95% CI 2-sided [-16.7 to 12.6], Standard Error of Mean 7.39
Statistical Analysis 151: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.0802, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.7, 95% CI 2-sided [-27.0 to 1.6], Standard Error of Mean 7.22
Statistical Analysis 152: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.1386, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -11.1, 95% CI 2-sided [-25.9 to 3.6], Standard Error of Mean 7.48
Statistical Analysis 153: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.5101, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -4.8, 95% CI 2-sided [-19.2 to 9.6], Standard Error of Mean 7.26
Statistical Analysis 154: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.0972, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -12.1, 95% CI 2-sided [-26.5 to 2.2], Standard Error of Mean 7.25
Statistical Analysis 155: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.4454, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = -5.8, 95% CI 2-sided [-20.9 to 9.2], Standard Error of Mean 7.61
Statistical Analysis 156: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.7638, ANCOVA — [p-value comment as in outcome 28, analysis 1]; LS Mean Difference = 2.2, 95% CI 2-sided [-12.2 to 16.6], Standard Error of Mean 7.28

30. Secondary Outcome: Phase 2b: Percentage of Participants Achieving at Least a 6-Point Reduction From Baseline in Weekly Average WI-NRS Over Time
Description: as for outcome 2
Time Frame: Baseline, Weeks 1 through 52
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period. Non-responders imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage of participants
  Week 1 | 4.3 [0.5 to 14.5] | 0 [0.0 to 7.5] | 2.2 [0.1 to 11.5] | 2.1 [0.1 to 11.1]
  Week 2 | 12.8 [4.8 to 25.7] | 4.3 [0.5 to 14.5] | 8.7 [2.4 to 20.8] | 2.1 [0.1 to 11.1]
  Week 3 | 21.3 [10.7 to 35.7] | 2.1 [0.1 to 11.3] | 8.7 [2.4 to 20.8] | 2.1 [0.1 to 11.1]
  Week 4 | 27.7 [15.6 to 42.6] | 10.6 [3.5 to 23.1] | 6.5 [1.4 to 17.9] | 0 [0.0 to 7.4]
  Week 5 | 29.8 [17.3 to 44.9] | 10.6 [3.5 to 23.1] | 8.7 [2.4 to 20.8] | 2.1 [0.1 to 11.1]
  Week 6 | 27.7 [15.6 to 42.6] | 17.0 [7.6 to 30.8] | 8.7 [2.4 to 20.8] | 0 [0.0 to 7.4]
  Week 7 | 29.8 [17.3 to 44.9] | 21.3 [10.7 to 35.7] | 10.9 [3.6 to 23.6] | 0 [0.0 to 7.4]
  Week 8 | 34.0 [20.9 to 49.3] | 19.1 [9.1 to 33.3] | 6.5 [1.4 to 17.9] | 2.1 [0.1 to 11.1]
  Week 9 | 31.9 [19.1 to 47.1] | 21.3 [10.7 to 35.7] | 15.2 [6.3 to 28.9] | 4.2 [0.5 to 14.3]
  Week 10 | 38.3 [24.5 to 53.6] | 23.4 [12.3 to 38.0] | 19.6 [9.4 to 33.9] | 6.3 [1.3 to 17.2]
  Week 11 | 40.4 [26.4 to 55.7] | 25.5 [13.9 to 40.3] | 13.0 [4.9 to 26.3] | 4.2 [0.5 to 14.3]
  Week 12 | 36.2 [22.7 to 51.5] | 21.3 [10.7 to 35.7] | 10.9 [3.6 to 23.6] | 6.3 [1.3 to 17.2]
  Week 13 | 36.2 [22.7 to 51.5] | 31.9 [19.1 to 47.1] | 17.4 [7.8 to 31.4] | 6.3 [1.3 to 17.2]
  Week 14 | 42.6 [28.3 to 57.8] | 29.8 [17.3 to 44.9] | 19.6 [9.4 to 33.9] | 8.3 [2.3 to 20.0]
  Week 15 | 42.6 [28.3 to 57.8] | 27.7 [15.6 to 42.6] | 17.4 [7.8 to 31.4] | 6.3 [1.3 to 17.2]
  Week 16 | 42.6 [28.3 to 57.8] | 23.4 [12.3 to 38.0] | 17.4 [7.8 to 31.4] | 2.1 [0.1 to 11.1]
  Week 17 | 51.1 [35.8 to 66.3] | 34.9 [21.0 to 50.9] | 21.7 [10.9 to 36.4] | 13.0 [4.9 to 26.3]
  Week 18 | 53.3 [37.9 to 68.3] | 37.2 [23.0 to 53.3] | 28.3 [16.0 to 43.5] | 17.4 [7.8 to 31.4]
  Week 19 | 53.3 [37.9 to 68.3] | 41.9 [27.0 to 57.9] | 39.1 [25.1 to 54.6] | 23.9 [12.6 to 38.8]
  Week 20 | 55.6 [40.0 to 70.4] | 37.2 [23.0 to 53.3] | 34.8 [21.4 to 50.2] | 32.6 [19.5 to 48.0]
  Week 21 | 55.6 [40.0 to 70.4] | 55.8 [39.9 to 70.9] | 43.5 [28.9 to 58.9] | 32.6 [19.5 to 48.0]
  Week 22 | 51.1 [35.8 to 66.3] | 53.5 [37.7 to 68.8] | 37.0 [23.2 to 52.5] | 32.6 [19.5 to 48.0]
  Week 23 | 46.7 [31.7 to 62.1] | 51.2 [35.5 to 66.7] | 43.5 [28.9 to 58.9] | 43.5 [28.9 to 58.9]
  Week 24 | 46.7 [31.7 to 62.1] | 58.1 [42.1 to 73.0] | 47.8 [32.9 to 63.1] | 43.5 [28.9 to 58.9]
  Week 25 | 48.9 [33.7 to 64.2] | 53.5 [37.7 to 68.8] | 45.7 [30.9 to 61.0] | 47.8 [32.9 to 63.1]
  Week 26 | 48.9 [33.7 to 64.2] | 55.8 [39.9 to 70.9] | 45.7 [30.9 to 61.0] | 45.7 [30.9 to 61.0]
  Week 27 | 55.6 [40.0 to 70.4] | 55.8 [39.9 to 70.9] | 43.5 [28.9 to 58.9] | 47.8 [32.9 to 63.1]
  Week 28 | 53.3 [37.9 to 68.3] | 55.8 [39.9 to 70.9] | 41.3 [27.0 to 56.8] | 45.7 [30.9 to 61.0]
  Week 29 | 55.6 [40.0 to 70.4] | 58.1 [42.1 to 73.0] | 47.8 [32.9 to 63.1] | 47.8 [32.9 to 63.1]
  Week 30 | 57.8 [42.2 to 72.3] | 55.8 [39.9 to 70.9] | 45.7 [30.9 to 61.0] | 47.8 [32.9 to 63.1]
  Week 31 | 60.0 [44.3 to 74.3] | 55.8 [39.9 to 70.9] | 50.0 [34.9 to 65.1] | 47.8 [32.9 to 63.1]
  Week 32 | 53.3 [37.9 to 68.3] | 53.5 [37.7 to 68.8] | 45.7 [30.9 to 61.0] | 52.2 [36.9 to 67.1]
  Week 33 | 57.8 [42.2 to 72.3] | 62.8 [46.7 to 77.0] | 50.0 [34.9 to 65.1] | 50.0 [34.9 to 65.1]
  Week 34 | 60.0 [44.3 to 74.3] | 58.1 [42.1 to 73.0] | 47.8 [32.9 to 63.1] | 50.0 [34.9 to 65.1]
  Week 35 | 57.8 [42.2 to 72.3] | 55.8 [39.9 to 70.9] | 50.0 [34.9 to 65.1] | 50.0 [34.9 to 65.1]
  Week 36 | 57.8 [42.2 to 72.3] | 55.8 [39.9 to 70.9] | 58.7 [43.2 to 73.0] | 50.0 [34.9 to 65.1]
  Week 37 | 55.6 [40.0 to 70.4] | 58.1 [42.1 to 73.0] | 56.5 [41.1 to 71.1] | 47.8 [32.9 to 63.1]
  Week 38 | 55.6 [40.0 to 70.4] | 60.5 [44.4 to 75.0] | 54.3 [39.0 to 69.1] | 50.0 [34.9 to 65.1]
  Week 39 | 60.0 [44.3 to 74.3] | 60.5 [44.4 to 75.0] | 60.9 [45.4 to 74.9] | 52.2 [36.9 to 67.1]
  Week 40 | 51.1 [35.8 to 66.3] | 58.1 [42.1 to 73.0] | 60.9 [45.4 to 74.9] | 52.2 [36.9 to 67.1]
  Week 41 | 55.6 [40.0 to 70.4] | 58.1 [42.1 to 73.0] | 56.5 [41.1 to 71.1] | 54.3 [39.0 to 69.1]
  Week 42 | 53.3 [37.9 to 68.3] | 60.5 [44.4 to 75.0] | 58.7 [43.2 to 73.0] | 54.3 [39.0 to 69.1]
  Week 43 | 46.7 [31.7 to 62.1] | 62.8 [46.7 to 77.0] | 54.3 [39.0 to 69.1] | 52.2 [36.9 to 67.1]
  Week 44 | 51.1 [35.8 to 66.3] | 58.1 [42.1 to 73.0] | 58.7 [43.2 to 73.0] | 50.0 [34.9 to 65.1]
  Week 45 | 55.6 [40.0 to 70.4] | 65.1 [49.1 to 79.0] | 50.0 [34.9 to 65.1] | 52.2 [36.9 to 67.1]
  Week 46 | 55.6 [40.0 to 70.4] | 60.5 [44.4 to 75.0] | 47.8 [32.9 to 63.1] | 52.2 [36.9 to 67.1]
  Week 47 | 55.6 [40.0 to 70.4] | 60.5 [44.4 to 75.0] | 47.8 [32.9 to 63.1] | 54.3 [39.0 to 69.1]
  Week 48 | 55.6 [40.0 to 70.4] | 58.1 [42.1 to 73.0] | 58.7 [43.2 to 73.0] | 56.5 [41.1 to 71.1]
  Week 49 | 60.0 [44.3 to 74.3] | 55.8 [39.9 to 70.9] | 52.2 [36.9 to 67.1] | 58.7 [43.2 to 73.0]
  Week 50 | 60.0 [44.3 to 74.3] | 55.8 [39.9 to 70.9] | 54.3 [39.0 to 69.1] | 54.3 [39.0 to 69.1]
  Week 51 | 57.8 [42.2 to 72.3] | 53.5 [37.7 to 68.8] | 54.3 [39.0 to 69.1] | 52.2 [36.9 to 67.1]
  Week 52 | 60.0 [44.3 to 74.3] | 46.5 [31.2 to 62.3] | 47.8 [32.9 to 63.1] | 56.5 [41.1 to 71.1]
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p = 0.5673, Cochran-Mantel-Haenszel — Calculated from CMH tests adjusted by the randomization stratification variables: sex and years since the first nodule observed (>= 10 years vs. < 10 years); Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.18 to 20.86]
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p = 0.3173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p = 0.7668, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.08 to 29.41]
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0520, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 6.26, 95% CI 2-sided [0.76 to 51.82]
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.5457, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.17 to 28.14]
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.1053, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 6.77, 95% CI 2-sided [0.57 to 79.79]
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p = 0.0043, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 11.30, 95% CI 2-sided [1.45 to 88.33]
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.06 to 18.08]
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p = 0.1006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 6.81, 95% CI 2-sided [0.59 to 79.12]
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0193, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0463, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 15.95, 95% CI 2-sided [2.26 to 112.81]
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p = 0.0917, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 5.82, 95% CI 2-sided [0.62 to 54.99]
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p = 0.1006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 6.81, 95% CI 2-sided [0.59 to 79.12]
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p = 0.0035, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p = 0.0269, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p = 0.0098, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 28.79, 95% CI 2-sided [3.21 to 258.26]
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0074, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 10.16, 95% CI 2-sided [1.31 to 79.08]
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.2466, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 3.09, 95% CI 2-sided [0.37 to 26.06]
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 11.56, 95% CI 2-sided [2.37 to 56.49]
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p = 0.0140, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 6.06, 95% CI 2-sided [1.25 to 29.37]
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p = 0.0823, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 3.70, 95% CI 2-sided [0.76 to 18.07]
Statistical Analysis 28: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 9.38, 95% CI 2-sided [2.51 to 35.02]
Statistical Analysis 29: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p = 0.0197, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 4.65, 95% CI 2-sided [1.20 to 18.10]
Statistical Analysis 30: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p = 0.0392, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 3.94, 95% CI 2-sided [0.99 to 15.69]
Statistical Analysis 31: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 13.93, 95% CI 2-sided [3.18 to 61.09]
Statistical Analysis 32: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p = 0.0036, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 8.54, 95% CI 2-sided [1.72 to 42.37]
Statistical Analysis 33: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p = 0.0638, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 4.43, 95% CI 2-sided [0.81 to 24.23]
Statistical Analysis 34: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 8.56, 95% CI 2-sided [2.28 to 32.07]
Statistical Analysis 35: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0379, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 4.09, 95% CI 2-sided [1.03 to 16.19]
Statistical Analysis 36: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.3367, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.46 to 8.78]
Statistical Analysis 37: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 9.73, 95% CI 2-sided [2.46 to 38.51]
Statistical Analysis 38: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 6.72, 95% CI 2-sided [1.82 to 24.75]
Statistical Analysis 39: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p = 0.0831, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.93, 95% CI 2-sided [0.79 to 10.83]
Statistical Analysis 40: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 8.51, 95% CI 2-sided [2.58 to 28.06]
Statistical Analysis 41: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p = 0.0087, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 4.74, 95% CI 2-sided [1.41 to 15.94]
Statistical Analysis 42: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p = 0.1361, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.61, 95% CI 2-sided [0.73 to 9.37]
Statistical Analysis 43: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 11.72, 95% CI 2-sided [3.08 to 44.56]
Statistical Analysis 44: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p = 0.0058, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 5.74, 95% CI 2-sided [1.51 to 21.75]
Statistical Analysis 45: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p = 0.1036, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 3.16, 95% CI 2-sided [0.77 to 13.03]
Statistical Analysis 46: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 71.24, 95% CI 2-sided [5.35 to 948.31]
Statistical Analysis 47: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0019, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 11.62, 95% CI 2-sided [1.62 to 83.47]
Statistical Analysis 48: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0117, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 8.48, 95% CI 2-sided [1.14 to 68.26]
Statistical Analysis 49: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 6.97, 95% CI 2-sided [2.46 to 19.76]
Statistical Analysis 50: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p = 0.0173, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 3.64, 95% CI 2-sided [1.23 to 10.74]
Statistical Analysis 51: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p = 0.2598, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.63 to 6.00]
Statistical Analysis 52: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 5.09, 95% CI 2-sided [1.98 to 13.11]
Statistical Analysis 53: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0402, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.90, 95% CI 2-sided [1.05 to 8.02]
Statistical Analysis 54: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.2003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.70 to 5.51]
Statistical Analysis 55: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.0034, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 3.84, 95% CI 2-sided [1.52 to 9.67]
Statistical Analysis 56: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.0749, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.31, 95% CI 2-sided [0.92 to 5.80]
Statistical Analysis 57: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.1248, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.82 to 5.02]
Statistical Analysis 58: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0278, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.09 to 6.03]
Statistical Analysis 59: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.7001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.48 to 2.97]
Statistical Analysis 60: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.7844, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.46 to 2.84]
Statistical Analysis 61: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.0249, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.68, 95% CI 2-sided [1.12 to 6.44]
Statistical Analysis 62: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.0303, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.09 to 6.54]
Statistical Analysis 63: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.2601, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.69 to 4.12]
Statistical Analysis 64: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.0691, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.94 to 5.46]
Statistical Analysis 65: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.0538, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 2.32, 95% CI 2-sided [0.98 to 5.52]
Statistical Analysis 66: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.6258, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.52 to 2.94]
Statistical Analysis 67: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.7407, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.50 to 2.63]
Statistical Analysis 68: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.5218, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.57 to 3.06]
Statistical Analysis 69: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.9855, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.43 to 2.34]
Statistical Analysis 70: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.7407, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.50 to 2.68]
Statistical Analysis 71: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.1843, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.76 to 4.17]
Statistical Analysis 72: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.6364, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.54 to 2.77]
Statistical Analysis 73: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.9206, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.45 to 2.40]
Statistical Analysis 74: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.6473, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.52 to 2.87]
Statistical Analysis 75: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.8733, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.40 to 2.15]
Statistical Analysis 76: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.7380, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.50 to 2.68]
Statistical Analysis 77: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.3768, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.63 to 3.43]
Statistical Analysis 78: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.9363, Cochran-Mantel-Haenszel — [p-value comment as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.45 to 2.41]
Statistical Analysis 79: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.4558, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.60 to 3.18]
Statistical Analysis 80: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.4883, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.57 to 3.24]
Statistical Analysis 81: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.6970, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.36 to 1.96]
Statistical Analysis 82: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.4601, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.60 to 3.16]
Statistical Analysis 83: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.3758, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.63 to 3.51]
Statistical Analysis 84: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.7248, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.36 to 2.02]
Statistical Analysis 85: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.4550, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.60 to 3.11]
Statistical Analysis 86: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.3672, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.64 to 3.35]
Statistical Analysis 87: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.9120, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.47 to 2.35]
Statistical Analysis 88: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.3506, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.65 to 3.35]
Statistical Analysis 89: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.4969, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.58 to 3.16]
Statistical Analysis 90: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.9265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.42 to 2.19]
Statistical Analysis 91: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.2440, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.72 to 3.79]
Statistical Analysis 92: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.4829, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.59 to 3.15]
Statistical Analysis 93: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.7382, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.51 to 2.61]
Statistical Analysis 94: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.8833, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.47 to 2.41]
Statistical Analysis 95: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.9385, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.44 to 2.41]
Statistical Analysis 96: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.5975, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.35 to 1.82]
Statistical Analysis 97: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.4491, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.61 to 3.13]
Statistical Analysis 98: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.2348, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.72 to 4.05]
Statistical Analysis 99: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.9087, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.46 to 2.38]
Statistical Analysis 100: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.3349, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.66 to 3.42]
Statistical Analysis 101: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.4806, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.58 to 3.17]
Statistical Analysis 102: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.8998, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.42 to 2.15]
Statistical Analysis 103: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.4618, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.60 to 3.12]
Statistical Analysis 104: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.6154, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.53 to 2.93]
Statistical Analysis 105: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.9442, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.45 to 2.34]
Statistical Analysis 106: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.4580, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.60 to 3.08]
Statistical Analysis 107: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.6275, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.52 to 2.95]
Statistical Analysis 108: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.3558, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.65 to 3.36]
Statistical Analysis 109: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.4749, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.60 to 3.04]
Statistical Analysis 110: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.3672, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.64 to 3.46]
Statistical Analysis 111: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.3462, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.65 to 3.37]
Statistical Analysis 112: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.5856, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.56 to 2.82]
Statistical Analysis 113: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.3563, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.64 to 3.58]
Statistical Analysis 114: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.6165, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.54 to 2.82]
Statistical Analysis 115: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.4532, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.60 to 3.10]
Statistical Analysis 116: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.4691, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.58 to 3.27]
Statistical Analysis 117: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.3703, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.64 to 3.32]
Statistical Analysis 118: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.9319, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.43 to 2.15]
Statistical Analysis 119: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.6374, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.52 to 2.94]
Statistical Analysis 120: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.3457, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.65 to 3.42]
Statistical Analysis 121: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.8906, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.47 to 2.37]
Statistical Analysis 122: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.7882, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.47 to 2.68]
Statistical Analysis 123: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.7898, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.49 to 2.59]
Statistical Analysis 124: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.9521, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.44 to 2.18]
Statistical Analysis 125: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.6001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.53 to 3.05]
Statistical Analysis 126: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.6054, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.55 to 2.80]
Statistical Analysis 127: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.6042, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.36 to 1.81]
Statistical Analysis 128: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.3465, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.64 to 3.73]
Statistical Analysis 129: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.7427, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.50 to 2.64]
Statistical Analysis 130: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.9218, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.47 to 2.30]
Statistical Analysis 131: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.4909, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.57 to 3.30]
Statistical Analysis 132: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.3616, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.65 to 3.31]
Statistical Analysis 133: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.7578, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.51 to 2.55]
Statistical Analysis 134: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.2369, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.71 to 4.24]
Statistical Analysis 135: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.8774, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.41 to 2.12]
Statistical Analysis 136: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.7578, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.51 to 2.55]
Statistical Analysis 137: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.4691, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.58 to 3.33]
Statistical Analysis 138: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.7272, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.38 to 1.95]
Statistical Analysis 139: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Superiority; p = 0.9080, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.47 to 2.35]
Statistical Analysis 140: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Superiority; p = 0.6001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.53 to 3.05]
Statistical Analysis 141: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Superiority; p = 0.5599, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.35 to 1.76]
Statistical Analysis 142: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.9274, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.43 to 2.17]
Statistical Analysis 143: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.9333, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.44 to 2.47]
Statistical Analysis 144: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.7796, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.50 to 2.50]
Statistical Analysis 145: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.8861, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.46 to 2.44]
Statistical Analysis 146: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.7331, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.36 to 2.03]
Statistical Analysis 147: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.5686, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.35 to 1.78]
Statistical Analysis 148: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.6010, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.55 to 2.84]
Statistical Analysis 149: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.9732, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.43 to 2.40]
Statistical Analysis 150: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.9378, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.46 to 2.32]
Statistical Analysis 151: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.5799, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.55 to 2.92]
Statistical Analysis 152: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.9790, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.42 to 2.44]
Statistical Analysis 153: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.7299, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.51 to 2.64]
Statistical Analysis 154: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.7357, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.51 to 2.64]
Statistical Analysis 155: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.3243, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.28 to 1.51]
Statistical Analysis 156: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.4364, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.32 to 1.63]

31. Secondary Outcome: Phase 2b: Percentage of Participants Achieving at Least a 4-Point Reduction From Baseline in Weekly Average WI-NRS Over Time
Description: as for outcome 2
Time Frame: Baseline, Weeks 1 through 52
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage of participants
  Week 1 | 10.6 [3.5 to 23.1] | 4.3 [0.5 to 14.5] | 4.3 [0.5 to 14.5] | 2.1 [0.1 to 11.1]
  Week 2 | 25.5 [13.9 to 40.3] | 17.0 [7.6 to 30.8] | 17.0 [7.6 to 30.8] | 4.2 [0.5 to 14.3]
  Week 3 | 44.7 [30.2 to 59.9] | 17.0 [7.6 to 30.8] | 17.0 [7.6 to 30.8] | 4.2 [0.5 to 14.3]
  Week 4 | 53.2 [38.1 to 67.9] | 25.5 [13.9 to 40.3] | 10.6 [3.5 to 23.1] | 6.3 [1.3 to 17.2]
  Week 5 | 53.2 [38.1 to 67.9] | 29.8 [17.3 to 44.9] | 21.3 [10.7 to 35.7] | 2.1 [0.1 to 11.1]
  Week 6 | 53.2 [38.1 to 67.9] | 38.3 [24.5 to 53.6] | 27.7 [15.6 to 42.6] | 6.3 [1.3 to 17.2]
  Week 7 | 57.4 [42.2 to 71.7] | 38.3 [24.5 to 53.6] | 27.7 [15.6 to 42.6] | 8.3 [2.3 to 20.0]
  Week 8 | 57.4 [42.2 to 71.7] | 36.2 [22.7 to 51.5] | 27.7 [15.6 to 42.6] | 8.3 [2.3 to 20.0]
  Week 9 | 59.6 [44.3 to 73.6] | 51.1 [36.1 to 65.9] | 36.2 [22.7 to 51.5] | 8.3 [2.3 to 20.0]
  Week 10 | 66.0 [50.7 to 79.1] | 59.6 [44.3 to 73.6] | 38.3 [24.5 to 53.6] | 12.5 [4.7 to 25.2]
  Week 11 | 63.8 [48.5 to 77.3] | 55.3 [40.1 to 69.8] | 31.9 [19.1 to 47.1] | 16.7 [7.5 to 30.2]
  Week 12 | 61.7 [46.4 to 75.5] | 57.4 [42.2 to 71.7] | 29.8 [17.3 to 44.9] | 16.7 [7.5 to 30.2]
  Week 13 | 63.8 [48.5 to 77.3] | 59.6 [44.3 to 73.6] | 36.2 [22.7 to 51.5] | 14.6 [6.1 to 27.8]
  Week 14 | 68.1 [52.9 to 80.9] | 63.8 [48.5 to 77.3] | 38.3 [24.5 to 53.6] | 16.7 [7.5 to 30.2]
  Week 15 | 66.0 [50.7 to 79.1] | 59.6 [44.3 to 73.6] | 36.2 [22.7 to 51.5] | 14.6 [6.1 to 27.8]
  Week 16 | 66.0 [50.7 to 79.1] | 61.7 [46.4 to 75.5] | 29.8 [17.3 to 44.9] | 16.7 [7.5 to 30.2]
  Week 17 | 68.9 [53.4 to 81.8] | 72.1 [56.3 to 84.7] | 48.9 [34.1 to 63.9] | 21.7 [10.9 to 36.4]
  Week 18 | 66.7 [51.0 to 80.0] | 72.1 [56.3 to 84.7] | 46.8 [32.1 to 61.9] | 32.6 [19.5 to 48.0]
  Week 19 | 71.1 [55.7 to 83.6] | 72.1 [56.3 to 84.7] | 55.3 [40.1 to 69.8] | 43.5 [28.9 to 58.9]
  Week 20 | 71.1 [55.7 to 83.6] | 67.4 [51.5 to 80.9] | 57.4 [42.2 to 71.7] | 47.8 [32.9 to 63.1]
  Week 21 | 68.9 [53.4 to 81.8] | 72.1 [56.3 to 84.7] | 68.1 [52.9 to 80.9] | 52.2 [36.9 to 67.1]
  Week 22 | 66.7 [51.0 to 80.0] | 72.1 [56.3 to 84.7] | 61.7 [46.4 to 75.5] | 54.3 [39.0 to 69.1]
  Week 23 | 64.4 [48.8 to 78.1] | 76.7 [61.4 to 88.2] | 66.0 [50.7 to 79.1] | 56.5 [41.1 to 71.1]
  Week 24 | 68.9 [53.4 to 81.8] | 72.1 [56.3 to 84.7] | 68.1 [52.9 to 80.9] | 54.3 [39.0 to 69.1]
  Week 25 | 64.4 [48.8 to 78.1] | 74.4 [58.8 to 86.5] | 66.0 [50.7 to 79.1] | 56.5 [41.1 to 71.1]
  Week 26 | 66.7 [51.0 to 80.0] | 72.1 [56.3 to 84.7] | 70.2 [55.1 to 82.7] | 56.5 [41.1 to 71.1]
  Week 27 | 66.7 [51.0 to 80.0] | 72.1 [56.3 to 84.7] | 68.1 [52.9 to 80.9] | 60.9 [45.4 to 74.9]
  Week 28 | 68.9 [53.4 to 81.8] | 72.1 [56.3 to 84.7] | 61.7 [46.4 to 75.5] | 60.9 [45.4 to 74.9]
  Week 29 | 68.9 [53.4 to 81.8] | 72.1 [56.3 to 84.7] | 68.1 [52.9 to 80.9] | 65.2 [49.8 to 78.6]
  Week 30 | 68.9 [53.4 to 81.8] | 72.1 [56.3 to 84.7] | 68.1 [52.9 to 80.9] | 63.0 [47.5 to 76.8]
  Week 31 | 71.1 [55.7 to 83.6] | 72.1 [56.3 to 84.7] | 66.0 [50.7 to 79.1] | 63.0 [47.5 to 76.8]
  Week 32 | 68.9 [53.4 to 81.8] | 74.4 [58.8 to 86.5] | 61.7 [46.4 to 75.5] | 63.0 [47.5 to 76.8]
  Week 33 | 66.7 [51.0 to 80.0] | 76.7 [61.4 to 88.2] | 66.0 [50.7 to 79.1] | 67.4 [52.0 to 80.5]
  Week 34 | 71.1 [55.7 to 83.6] | 72.1 [56.3 to 84.7] | 66.0 [50.7 to 79.1] | 63.0 [47.5 to 76.8]
  Week 35 | 71.1 [55.7 to 83.6] | 67.4 [51.5 to 80.9] | 68.1 [52.9 to 80.9] | 67.4 [52.0 to 80.5]
  Week 36 | 71.1 [55.7 to 83.6] | 69.8 [53.9 to 82.8] | 72.3 [57.4 to 84.4] | 65.2 [49.8 to 78.6]
  Week 37 | 71.1 [55.7 to 83.6] | 74.4 [58.8 to 86.5] | 72.3 [57.4 to 84.4] | 69.6 [54.2 to 82.3]
  Week 38 | 75.6 [60.5 to 87.1] | 72.1 [56.3 to 84.7] | 72.3 [57.4 to 84.4] | 69.6 [54.2 to 82.3]
  Week 39 | 71.1 [55.7 to 83.6] | 72.1 [56.3 to 84.7] | 68.1 [52.9 to 80.9] | 71.7 [56.5 to 84.0]
  Week 40 | 73.3 [58.1 to 85.4] | 69.8 [53.9 to 82.8] | 68.1 [52.9 to 80.9] | 69.6 [54.2 to 82.3]
  Week 41 | 71.1 [55.7 to 83.6] | 72.1 [56.3 to 84.7] | 68.1 [52.9 to 80.9] | 71.7 [56.5 to 84.0]
  Week 42 | 71.1 [55.7 to 83.6] | 72.1 [56.3 to 84.7] | 68.1 [52.9 to 80.9] | 71.7 [56.5 to 84.0]
  Week 43 | 71.1 [55.7 to 83.6] | 74.4 [58.8 to 86.5] | 66.0 [50.7 to 79.1] | 69.6 [54.2 to 82.3]
  Week 44 | 73.3 [58.1 to 85.4] | 69.8 [53.9 to 82.8] | 66.0 [50.7 to 79.1] | 73.9 [58.9 to 85.7]
  Week 45 | 75.6 [60.5 to 87.1] | 69.8 [53.9 to 82.8] | 66.0 [50.7 to 79.1] | 69.6 [54.2 to 82.3]
  Week 46 | 75.6 [60.5 to 87.1] | 76.7 [61.4 to 88.2] | 68.1 [52.9 to 80.9] | 73.9 [58.9 to 85.7]
  Week 47 | 75.6 [60.5 to 87.1] | 72.1 [56.3 to 84.7] | 66.0 [50.7 to 79.1] | 73.9 [58.9 to 85.7]
  Week 48 | 75.6 [60.5 to 87.1] | 69.8 [53.9 to 82.8] | 63.8 [48.5 to 77.3] | 76.1 [61.2 to 87.4]
  Week 49 | 75.6 [60.5 to 87.1] | 67.4 [51.5 to 80.9] | 59.6 [44.3 to 73.6] | 73.9 [58.9 to 85.7]
  Week 50 | 71.1 [55.7 to 83.6] | 65.1 [49.1 to 79.0] | 61.7 [46.4 to 75.5] | 67.4 [52.0 to 80.5]
  Week 51 | 71.1 [55.7 to 83.6] | 60.5 [44.4 to 75.0] | 61.7 [46.4 to 75.5] | 65.2 [49.8 to 78.6]
  Week 52 | 71.1 [55.7 to 83.6] | 55.8 [39.9 to 70.9] | 57.4 [42.2 to 71.7] | 69.6 [54.2 to 82.3]
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p = 0.0957, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.18, 95% CI 2-sided [0.60 to 44.60]
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p = 0.5457, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.17 to 28.14]
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 1; Test type: Superiority; p = 0.3797, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.14, 95% CI 2-sided [0.24 to 41.51]
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0042, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 7.97, 95% CI 2-sided [1.64 to 38.75]
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0383, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.08, 95% CI 2-sided [0.99 to 26.09]
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0357, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.42, 95% CI 2-sided [1.02 to 28.92]
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 17.35, 95% CI 2-sided [3.86 to 77.91]
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p = 0.0408, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.04, 95% CI 2-sided [0.97 to 26.01]
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 3; Test type: Superiority; p = 0.0357, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.42, 95% CI 2-sided [1.02 to 28.92]
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 16.80, 95% CI 2-sided [4.51 to 62.54]
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0116, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.95, 95% CI 2-sided [1.31 to 18.78]
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.3738, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.43 to 8.82]
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 44.08, 95% CI 2-sided [6.06 to 320.77]
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 27.11, 95% CI 2-sided [2.73 to 268.93]
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 5; Test type: Superiority; p = 0.0029, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 17.02, 95% CI 2-sided [1.74 to 166.84]
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 17.84, 95% CI 2-sided [4.70 to 67.78]
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 9.86, 95% CI 2-sided [2.60 to 37.44]
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 6; Test type: Superiority; p = 0.0055, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.87, 95% CI 2-sided [1.53 to 22.53]
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 14.14, 95% CI 2-sided [4.37 to 45.75]
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 6.85, 95% CI 2-sided [2.11 to 22.25]
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 7; Test type: Superiority; p = 0.0160, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.24, 95% CI 2-sided [1.25 to 14.41]
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 14.14, 95% CI 2-sided [4.37 to 45.75]
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 6.26, 95% CI 2-sided [1.93 to 20.33]
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0151, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.19, 95% CI 2-sided [1.25 to 14.04]
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 19.23, 95% CI 2-sided [5.35 to 69.06]
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 11.51, 95% CI 2-sided [3.48 to 38.09]
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 9; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 6.12, 95% CI 2-sided [1.86 to 20.20]
Statistical Analysis 28: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 14.64, 95% CI 2-sided [4.89 to 43.82]
Statistical Analysis 29: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 9.59, 95% CI 2-sided [3.44 to 26.76]
Statistical Analysis 30: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 10; Test type: Superiority; p = 0.0049, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.20, 95% CI 2-sided [1.48 to 11.90]
Statistical Analysis 31: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 8.30, 95% CI 2-sided [3.17 to 21.77]
Statistical Analysis 32: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.53, 95% CI 2-sided [2.20 to 13.92]
Statistical Analysis 33: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 11; Test type: Superiority; p = 0.0939, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.85 to 5.86]
Statistical Analysis 34: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 7.68, 95% CI 2-sided [2.91 to 20.31]
Statistical Analysis 35: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 6.51, 95% CI 2-sided [2.51 to 16.93]
Statistical Analysis 36: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.1425, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.77 to 5.28]
Statistical Analysis 37: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 9.99, 95% CI 2-sided [3.61 to 27.64]
Statistical Analysis 38: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 8.31, 95% CI 2-sided [3.08 to 22.43]
Statistical Analysis 39: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 13; Test type: Superiority; p = 0.0194, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.17, 95% CI 2-sided [1.17 to 8.60]
Statistical Analysis 40: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 9.13, 95% CI 2-sided [3.50 to 23.77]
Statistical Analysis 41: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 8.02, 95% CI 2-sided [3.11 to 20.70]
Statistical Analysis 42: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 14; Test type: Superiority; p = 0.0266, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.96, 95% CI 2-sided [1.12 to 7.87]
Statistical Analysis 43: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 10.39, 95% CI 2-sided [3.85 to 28.00]
Statistical Analysis 44: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 8.15, 95% CI 2-sided [3.04 to 21.86]
Statistical Analysis 45: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 15; Test type: Superiority; p = 0.0172, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.36, 95% CI 2-sided [1.22 to 9.29]
Statistical Analysis 46: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 8.60, 95% CI 2-sided [3.34 to 22.14]
Statistical Analysis 47: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 7.60, 95% CI 2-sided [2.91 to 19.79]
Statistical Analysis 48: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.1252, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.14, 95% CI 2-sided [0.80 to 5.75]
Statistical Analysis 49: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 8.01, 95% CI 2-sided [3.09 to 20.75]
Statistical Analysis 50: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 8.60, 95% CI 2-sided [3.30 to 22.40]
Statistical Analysis 51: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 17; Test type: Superiority; p = 0.0074, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.39, 95% CI 2-sided [1.38 to 8.34]
Statistical Analysis 52: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0015, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.94, 95% CI 2-sided [1.66 to 9.33]
Statistical Analysis 53: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.03, 95% CI 2-sided [2.04 to 12.40]
Statistical Analysis 54: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.1667, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.78 to 4.23]
Statistical Analysis 55: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.0087, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.12, 95% CI 2-sided [1.31 to 7.41]
Statistical Analysis 56: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.0079, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.26, 95% CI 2-sided [1.35 to 7.87]
Statistical Analysis 57: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 19; Test type: Superiority; p = 0.2631, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.71 to 3.63]
Statistical Analysis 58: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0263, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.59, 95% CI 2-sided [1.11 to 6.05]
Statistical Analysis 59: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0643, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.96 to 5.46]
Statistical Analysis 60: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.3954, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.63 to 3.27]
Statistical Analysis 61: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.1083, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.86 to 4.61]
Statistical Analysis 62: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.0613, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.96 to 5.69]
Statistical Analysis 63: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 21; Test type: Superiority; p = 0.1354, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.92, 95% CI 2-sided [0.82 to 4.47]
Statistical Analysis 64: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.2362, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.72 to 3.82]
Statistical Analysis 65: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.0949, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.88 to 5.17]
Statistical Analysis 66: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 22; Test type: Superiority; p = 0.5013, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.58 to 3.04]
Statistical Analysis 67: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.4386, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.61 to 3.16]
Statistical Analysis 68: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.0504, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.49, 95% CI 2-sided [0.99 to 6.24]
Statistical Analysis 69: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 23; Test type: Superiority; p = 0.3781, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.64 to 3.32]
Statistical Analysis 70: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.1535, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.79 to 4.21]
Statistical Analysis 71: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.0925, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.09, 95% CI 2-sided [0.87 to 4.99]
Statistical Analysis 72: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 24; Test type: Superiority; p = 0.1948, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.75 to 4.07]
Statistical Analysis 73: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.4304, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.61 to 3.17]
Statistical Analysis 74: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.0873, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.17, 95% CI 2-sided [0.89 to 5.31]
Statistical Analysis 75: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 25; Test type: Superiority; p = 0.3683, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.64 to 3.38]
Statistical Analysis 76: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.3203, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.66 to 3.48]
Statistical Analysis 77: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.1284, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.82 to 4.98]
Statistical Analysis 78: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 26; Test type: Superiority; p = 0.1790, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.76 to 4.11]
Statistical Analysis 79: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.5470, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.56 to 2.91]
Statistical Analysis 80: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.2612, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.68 to 4.16]
Statistical Analysis 81: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 27; Test type: Superiority; p = 0.5071, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.57 to 3.11]
Statistical Analysis 82: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.4175, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.61 to 3.19]
Statistical Analysis 83: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.284, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.68 to 4.32]
Statistical Analysis 84: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 28; Test type: Superiority; p = 0.9281, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.46 to 2.33]
Statistical Analysis 85: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.6987, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.51 to 2.69]
Statistical Analysis 86: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.4794, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.56 to 3.41]
Statistical Analysis 87: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 29; Test type: Superiority; p = 0.8164, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.48 to 2.52]
Statistical Analysis 88: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.5484, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.56 to 2.93]
Statistical Analysis 89: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.3596, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.62 to 3.76]
Statistical Analysis 90: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 30; Test type: Superiority; p = 0.6414, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.53 to 2.78]
Statistical Analysis 91: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.4233, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.60 to 3.20]
Statistical Analysis 92: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.3632, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.62 to 3.70]
Statistical Analysis 93: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 31; Test type: Superiority; p = 0.8018, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.49 to 2.49]
Statistical Analysis 94: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.5465, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.55 to 3.02]
Statistical Analysis 95: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.2560, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.68 to 4.14]
Statistical Analysis 96: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.8810, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.42 to 2.10]
Statistical Analysis 97: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.9701, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.43 to 2.24]
Statistical Analysis 98: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.3331, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.62 to 3.96]
Statistical Analysis 99: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 33; Test type: Superiority; p = 0.8386, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.40 to 2.11]
Statistical Analysis 100: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.4091, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.61 to 3.28]
Statistical Analysis 101: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.3746, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.61 to 3.57]
Statistical Analysis 102: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 34; Test type: Superiority; p = 0.8018, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.49 to 2.49]
Statistical Analysis 103: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.6717, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.51 to 2.79]
Statistical Analysis 104: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.9850, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.41 to 2.41]
Statistical Analysis 105: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 35; Test type: Superiority; p = 0.9983, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.43 to 2.31]
Statistical Analysis 106: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.5311, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.56 to 3.02]
Statistical Analysis 107: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.6628, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.50 to 2.99]
Statistical Analysis 108: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 36; Test type: Superiority; p = 0.5208, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.56 to 3.09]
Statistical Analysis 109: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.8483, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.46 to 2.55]
Statistical Analysis 110: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.6232, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.50 to 3.20]
Statistical Analysis 111: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 37; Test type: Superiority; p = 0.8312, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.46 to 2.61]
Statistical Analysis 112: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.5083, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.55 to 3.30]
Statistical Analysis 113: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.8111, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.44 to 2.86]
Statistical Analysis 114: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 38; Test type: Superiority; p = 0.8089, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.46 to 2.68]
Statistical Analysis 115: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.9723, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.41 to 2.37]
Statistical Analysis 116: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.9883, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.39 to 2.58]
Statistical Analysis 117: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 39; Test type: Superiority; p = 0.6781, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.35 to 1.98]
Statistical Analysis 118: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.6924, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.50 to 2.86]
Statistical Analysis 119: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.9883, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.40 to 2.47]
Statistical Analysis 120: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 40; Test type: Superiority; p = 0.8581, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.39 to 2.18]
Statistical Analysis 121: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.9723, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.41 to 2.37]
Statistical Analysis 122: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.9937, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.38 to 2.63]
Statistical Analysis 123: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 41; Test type: Superiority; p = 0.6781, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.35 to 1.98]
Statistical Analysis 124: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.9723, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.41 to 2.37]
Statistical Analysis 125: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.9937, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.38 to 2.63]
Statistical Analysis 126: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 42; Test type: Superiority; p = 0.6781, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.35 to 1.98]
Statistical Analysis 127: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.8892, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.44 to 2.57]
Statistical Analysis 128: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.6296, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.50 to 3.21]
Statistical Analysis 129: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 43; Test type: Superiority; p = 0.7271, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.36 to 2.02]
Statistical Analysis 130: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.9636, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.40 to 2.42]
Statistical Analysis 131: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.6355, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.32 to 2.00]
Statistical Analysis 132: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 44; Test type: Superiority; p = 0.3901, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.28 to 1.64]
Statistical Analysis 133: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.5177, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.54 to 3.36]
Statistical Analysis 134: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.9910, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.40 to 2.49]
Statistical Analysis 135: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 45; Test type: Superiority; p = 0.7064, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.35 to 2.01]
Statistical Analysis 136: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.8373, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.44 to 2.77]
Statistical Analysis 137: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.7614, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.44 to 3.11]
Statistical Analysis 138: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 46; Test type: Superiority; p = 0.5301, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.31 to 1.83]
Statistical Analysis 139: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Superiority; p = 0.8248, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.44 to 2.80]
Statistical Analysis 140: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Superiority; p = 0.8374, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.35 to 2.32]
Statistical Analysis 141: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 47; Test type: Superiority; p = 0.4088, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.29 to 1.67]
Statistical Analysis 142: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.9745, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.39 to 2.50]
Statistical Analysis 143: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.4916, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.28 to 1.84]
Statistical Analysis 144: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.1854, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.23 to 1.35]
Statistical Analysis 145: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.8373, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.44 to 2.77]
Statistical Analysis 146: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.5051, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.29 to 1.83]
Statistical Analysis 147: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 49; Test type: Superiority; p = 0.1375, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.21 to 1.24]
Statistical Analysis 148: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.7180, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.49 to 2.82]
Statistical Analysis 149: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.7838, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.37 to 2.13]
Statistical Analysis 150: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 50; Test type: Superiority; p = 0.5795, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.34 to 1.83]
Statistical Analysis 151: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.5517, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.54 to 3.14]
Statistical Analysis 152: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.6060, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.34 to 1.89]
Statistical Analysis 153: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 51; Test type: Superiority; p = 0.7491, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.38 to 2.02]
Statistical Analysis 154: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.8593, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.45 to 2.63]
Statistical Analysis 155: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.1868, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.23 to 1.32]
Statistical Analysis 156: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.2436, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.26 to 1.41]

32. Secondary Outcome: Phase 2b: Percentage of Participants Achieving 0 or 1 in PN-IGA Over Time
Description: PN-IGA is a novel exploratory tool for the overall investigator assessment of PN disease severity based on the presence/absence of nodules and the size of the nodules as defined by their elevation. The IGA utilizes a 5-point scale that ranges from 0 (clear) to 4 (severe disease); 0 (clear) indicates no nodules and 1 (almost clear) indicates nodules are present, few of the nodules are moderately raised.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 18, 20, 32, 48, 52
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage of participants
  Week 2 | 6.4 [1.3 to 17.5] | 0.0 [0.0 to 7.5] | 2.1 [0.1 to 11.3] | 0 [0.0 to 7.4]
  Week 4 | 6.4 [1.3 to 17.5] | 4.3 [0.5 to 14.5] | 4.3 [0.5 to 14.5] | 2.1 [0.1 to 11.1]
  Week 8 | 23.4 [12.3 to 38.0] | 10.6 [3.5 to 23.1] | 2.1 [0.1 to 11.3] | 4.2 [0.5 to 14.3]
  Week 12 | 29.8 [17.3 to 44.9] | 25.5 [13.9 to 40.3] | 8.5 [2.4 to 20.4] | 10.4 [3.5 to 22.7]
  Week 16 | 38.3 [24.5 to 53.6] | 29.8 [17.3 to 44.9] | 14.9 [6.2 to 28.3] | 10.4 [3.5 to 22.7]
  Week 18 | 44.4 [29.6 to 60.0] | 34.9 [21.0 to 50.9] | 19.1 [9.1 to 33.3] | 10.9 [3.6 to 23.6]
  Week 20 | 53.3 [37.9 to 68.3] | 46.5 [31.2 to 62.3] | 25.5 [13.9 to 40.3] | 21.7 [10.9 to 36.4]
  Week 32 | 48.9 [33.7 to 64.2] | 46.5 [31.2 to 62.3] | 34.0 [20.9 to 49.3] | 41.3 [27.0 to 56.8]
  Week 48 | 51.1 [35.8 to 66.3] | 53.5 [37.7 to 68.8] | 36.2 [22.7 to 51.5] | 52.2 [36.9 to 67.1]
  Week 52 | 51.1 [35.8 to 66.3] | 51.2 [35.5 to 66.7] | 44.7 [30.2 to 59.9] | 56.5 [41.1 to 71.1]
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0841, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.3442, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.3083, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.22, 95% CI 2-sided [0.31 to 33.01]
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.4905, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.21 to 22.64]
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.6379, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.15 to 21.08]
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0073, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 7.37, 95% CI 2-sided [1.48 to 36.68]
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.2453, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.68, 95% CI 2-sided [0.49 to 14.66]
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.4853, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.04 to 4.90]
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0205, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.51, 95% CI 2-sided [1.15 to 10.68]
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0548, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.05, 95% CI 2-sided [0.95 to 9.78]
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.6853, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.19 to 2.96]
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.65, 95% CI 2-sided [1.83 to 17.47]
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0196, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.61, 95% CI 2-sided [1.19 to 10.99]
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.6213, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.40 to 4.69]
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 7.44, 95% CI 2-sided [2.33 to 23.73]
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0060, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.84, 95% CI 2-sided [1.50 to 15.58]
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.3432, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.54 to 6.07]
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0012, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.96, 95% CI 2-sided [1.84 to 13.37]
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0121, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.21, 95% CI 2-sided [1.27 to 8.11]
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.8315, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.41 to 3.08]
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.4161, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.61 to 3.35]
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.6277, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.54 to 2.82]
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.4128, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.29 to 1.64]
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.9726, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.42 to 2.30]
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.9070, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.46 to 2.39]
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.0944, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.21 to 1.14]
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.6513, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.37 to 1.88]
Statistical Analysis 28: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.5924, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.35 to 1.82]
Statistical Analysis 29: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.2313, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.27 to 1.38]

33. Secondary Outcome: Phase 2b: Percentage of Participants With at Least 2-Point Improvement From Baseline in PN-IGA Over Time
Description: PN-IGA is a novel exploratory tool for the overall investigator assessment of PN disease severity based on the size of the nodules as defined by their elevation. The IGA utilizes a 5-point scale that ranges from 0 (clear) to 4 (severe disease).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 18, 20, 32, 48, 52
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage of participants
  Week 2 | 6.4 [1.3 to 17.5] | 2 [0.5 to 14.5] | 6.4 [1.3 to 17.5] | 2.1 [0.1 to 11.1]
  Week 4 | 14.9 [6.2 to 28.3] | 10.6 [3.5 to 23.1] | 8.5 [2.4 to 20.4] | 2.1 [0.1 to 11.1]
  Week 8 | 27.7 [15.6 to 42.6] | 21.3 [10.7 to 35.7] | 8.5 [2.4 to 20.4] | 4.2 [0.5 to 14.3]
  Week 12 | 31.9 [19.1 to 47.1] | 31.9 [19.1 to 47.1] | 12.8 [4.8 to 25.7] | 12.5 [4.7 to 25.2]
  Week 16 | 38.3 [24.5 to 53.6] | 40.4 [26.4 to 55.7] | 25.5 [13.9 to 40.3] | 12.5 [4.7 to 25.2]
  Week 18 | 46.7 [31.7 to 62.1] | 48.8 [33.3 to 64.5] | 27.7 [15.6 to 42.6] | 17.4 [7.8 to 31.4]
  Week 20 | 57.8 [42.2 to 72.3] | 58.1 [42.1 to 73.0] | 34.0 [20.9 to 49.3] | 26.1 [14.3 to 41.1]
  Week 32 | 55.6 [40.0 to 70.4] | 58.1 [42.1 to 73.0] | 46.8 [32.1 to 61.9] | 54.3 [39.0 to 69.1]
  Week 48 | 57.8 [42.2 to 72.3] | 62.8 [46.7 to 77.0] | 40.4 [26.4 to 55.7] | 58.7 [43.2 to 73.0]
  Week 52 | 53.3 [37.9 to 68.3] | 58.1 [42.1 to 73.0] | 48.9 [34.1 to 63.9] | 58.7 [43.2 to 73.0]
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.3137, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.19, 95% CI 2-sided [0.31 to 33.17]
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.5982, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.16 to 25.75]
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.3244, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.80, 95% CI 2-sided [0.31 to 25.38]
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0266, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 7.58, 95% CI 2-sided [0.96 to 59.86]
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0892, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.20, 95% CI 2-sided [0.63 to 42.80]
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.1864, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.06, 95% CI 2-sided [0.44 to 37.67]
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0020, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 9.27, 95% CI 2-sided [1.89 to 45.55]
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0141, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 6.42, 95% CI 2-sided [1.28 to 32.22]
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.4485, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.34 to 10.89]
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0235, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.30, 95% CI 2-sided [1.14 to 9.55]
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0252, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.29, 95% CI 2-sided [1.13 to 9.59]
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.9062, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.27 to 3.14]
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0041, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.55, 95% CI 2-sided [1.57 to 13.19]
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0025, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.72, 95% CI 2-sided [1.66 to 13.39]
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.1632, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.73 to 6.76]
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0030, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.09, 95% CI 2-sided [1.57 to 10.65]
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0014, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.01, 95% CI 2-sided [1.80 to 13.91]
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.3017, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.62 to 4.82]
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0018, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.18, 95% CI 2-sided [1.67 to 10.48]
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.31, 95% CI 2-sided [1.69 to 10.99]
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.5365, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.52 to 3.55]
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.8774, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.46 to 2.46]
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.7261, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.50 to 2.70]
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.4195, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.31 to 1.63]
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.9759, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.42 to 2.31]
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.6857, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.51 to 2.81]
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.0633, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.19 to 1.04]
Statistical Analysis 28: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.6466, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.36 to 1.88]
Statistical Analysis 29: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.9298, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.41 to 2.23]
Statistical Analysis 30: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.3143, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.29 to 1.49]

34. Secondary Outcome: Phase 2b: Percentage of Participants Achieving 0 (Clear) or 1 (Almost Clear) in Investigator's Global Assessment for Prurigo Nodularis-Stage (IGA-CNPG-S) Over Time
Description: IGA-CNPG-S is a novel tool for the investigator assessment of PN disease severity based on the number of palpable nodules and utilizes a 5-point scale that ranges from 0 (clear) to 4 (severe); 0 (clear) indicates no nodules and 1 (almost clear) indicates rare palpable pruriginous nodules (approximately 1-5 nodules). A score is assigned based on the appearance of the disease at the time of the evaluation without referring to the baseline state.
Time Frame: Weeks 2, 4, 8, 12, 16, 18, 20, 32, 48, 52
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage of participants
  Week 2 | 4.3 [0.5 to 14.5] | 2.1 [0.1 to 11.3] | 2.1 [0.1 to 11.3] | 0 [0.0 to 7.4]
  Week 4 | 8.5 [2.4 to 20.4] | 4.3 [0.5 to 14.5] | 4.3 [0.5 to 14.5] | 2.1 [0.1 to 11.1]
  Week 8 | 14.9 [6.2 to 28.3] | 10.6 [3.5 to 23.1] | 2.1 [0.1 to 11.3] | 4.2 [0.5 to 14.3]
  Week 12 | 25.5 [13.9 to 40.3] | 17.0 [7.6 to 30.8] | 10.6 [3.5 to 23.1] | 10.4 [3.5 to 22.7]
  Week 16 | 34.0 [20.9 to 49.3] | 25.5 [13.9 to 40.3] | 14.9 [6.2 to 28.3] | 6.3 [1.3 to 17.2]
  Week 18 | 42.2 [27.7 to 57.8] | 34.9 [21.0 to 50.9] | 21.3 [10.7 to 35.7] | 10.9 [3.6 to 23.6]
  Week 20 | 42.2 [27.7 to 57.8] | 39.5 [25.0 to 55.6] | 21.3 [10.7 to 35.7] | 17.4 [7.8 to 31.4]
  Week 32 | 44.4 [29.6 to 60.0] | 41.9 [27.0 to 57.9] | 21.3 [10.7 to 35.7] | 34.8 [21.4 to 50.2]
  Week 48 | 48.9 [33.7 to 64.2] | 51.2 [35.5 to 66.7] | 29.8 [17.3 to 44.9] | 50.0 [34.9 to 65.1]
  Week 52 | 46.7 [31.7 to 62.1] | 48.8 [33.3 to 64.5] | 42.6 [28.3 to 57.8] | 50.0 [34.9 to 65.1]
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.1656, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.3026, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.3442, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.1641, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.60, 95% CI 2-sided [0.47 to 45.07]
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.5103, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.24, 95% CI 2-sided [0.20 to 25.61]
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.5457, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.19 to 22.02]
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0722, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.24, 95% CI 2-sided [0.80 to 22.44]
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.2215, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.85, 95% CI 2-sided [0.51 to 16.01]
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.4872, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.03 to 5.06]
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0550, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.03, 95% CI 2-sided [0.95 to 9.68]
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.3519, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.52 to 6.10]
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.8266, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.22 to 3.34]
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 7.99, 95% CI 2-sided [2.11 to 30.30]
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0116, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.93, 95% CI 2-sided [1.32 to 18.39]
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.2127, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.50, 95% CI 2-sided [0.59 to 10.60]
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 7.00, 95% CI 2-sided [2.17 to 22.61]
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0061, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.61, 95% CI 2-sided [1.47 to 14.43]
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.2317, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.62 to 6.90]
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0093, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.65, 95% CI 2-sided [1.36 to 9.81]
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0183, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.26, 95% CI 2-sided [1.21 to 8.80]
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.7648, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.40 to 3.45]
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.3370, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.65 to 3.68]
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.5054, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.57 to 3.16]
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.1341, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.19 to 1.24]
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.9628, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.43 to 2.25]
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.9185, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.46 to 2.39]
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.0496, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.18 to 1.00]
Statistical Analysis 28: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.7785, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.38 to 2.04]
Statistical Analysis 29: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.8857, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.42 to 2.13]
Statistical Analysis 30: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.4174, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.31 to 1.62]

35. Secondary Outcome: Phase 2b: Percentage of Participants With at Least 2-point Improvement From Baseline in IGA-CNPG-S Over Time
Description: IGA-CNPG-S, administered at designated visits, is a novel tool for the investigator assessment of PN disease severity based on the number of palpable nodules and utilizes a 5-point scale that ranges from 0 (clear) to 4 (severe). A score is assigned based on the appearance of the disease at the time of the evaluation without referring to the baseline state.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 18, 20, 32, 48, 52
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage of participants
  Week 2 | 4.3 [0.5 to 14.5] | 6.4 [1.3 to 17.5] | 4.3 [0.5 to 14.5] | 2.1 [0.1 to 11.1]
  Week 4 | 12.8 [4.8 to 25.7] | 10.6 [3.5 to 23.1] | 8.5 [2.4 to 20.4] | 2.1 [0.1 to 11.1]
  Week 8 | 19.1 [9.1 to 33.3] | 12.8 [4.8 to 25.7] | 8.5 [2.4 to 20.4] | 4.2 [0.5 to 14.3]
  Week 12 | 27.7 [15.6 to 42.6] | 25.5 [13.9 to 40.3] | 14.9 [6.2 to 28.3] | 12.5 [4.7 to 25.2]
  Week 16 | 34.0 [20.9 to 49.3] | 34.0 [20.9 to 49.3] | 25.5 [13.9 to 40.3] | 12.5 [4.7 to 25.2]
  Week 18 | 46.7 [31.7 to 62.1] | 41.9 [27.0 to 57.9] | 29.8 [17.3 to 44.9] | 19.6 [9.4 to 33.9]
  Week 20 | 44.4 [29.6 to 60.0] | 46.5 [31.2 to 62.3] | 31.9 [19.1 to 47.1] | 30.4 [17.7 to 45.8]
  Week 32 | 48.9 [33.7 to 64.2] | 51.2 [35.5 to 66.7] | 36.2 [22.7 to 51.5] | 52.2 [36.9 to 67.1]
  Week 48 | 53.3 [37.9 to 72.3] | 60.5 [44.4 to 75.0] | 38.3 [24.5 to 53.6] | 56.5 [41.1 to 71.1]
  Week 52 | 53.3 [37.9 to 68.3] | 55.8 [39.9 to 70.9] | 46.8 [32.1 to 61.9] | 60.9 [45.4 to 74.9]
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.5673, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.18 to 22.87]
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.3139, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.17, 95% CI 2-sided [0.31 to 32.21]
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.6197, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.16 to 22.83]
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0480, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 6.95, 95% CI 2-sided [0.80 to 60.25]
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0945, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.44, 95% CI 2-sided [0.62 to 48.12]
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.1745, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 4.29, 95% CI 2-sided [0.45 to 40.60]
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0233, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 5.49, 95% CI 2-sided [1.10 to 27.25]
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.1422, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.21, 95% CI 2-sided [0.63 to 16.53]
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.4810, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.92, 95% CI 2-sided [0.31 to 11.77]
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0628, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.83, 95% CI 2-sided [0.93 to 8.60]
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.1149, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.80 to 6.87]
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.9726, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.30 to 3.48]
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0134, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.76, 95% CI 2-sided [1.28 to 11.00]
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0148, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.31, 95% CI 2-sided [1.21 to 9.06]
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.1611, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.21, 95% CI 2-sided [0.73 to 6.71]
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0061, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 3.72, 95% CI 2-sided [1.44 to 9.60]
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0228, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 2.84, 95% CI 2-sided [1.13 to 7.18]
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.3331, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.61 to 4.37]
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.1718, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.78 to 4.38]
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.1219, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.83 to 4.66]
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.9755, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.40 to 2.45]
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.7579, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.38 to 2.02]
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.9213, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.42 to 2.19]
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.1001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.21 to 1.14]
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.7945, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.39 to 2.05]
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.7214, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.51 to 2.69]
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.0727, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.20 to 1.07]
Statistical Analysis 28: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.4871, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.32 to 1.72]
Statistical Analysis 29: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.6037, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.35 to 1.85]
Statistical Analysis 30: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.1323, Cochran-Mantel-Haenszel — [p-value comment as in outcome 25, analysis 1]; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.23 to 1.22]

36. Secondary Outcome: Phase 2b: Change From Baseline in Weekly Average of Sleep Loss VAS Over Time
Description: Participants rated intensity of their average sleeplessness over previous 3 days on 0-10 line scale (0=no sleeplessness, 10=worst imaginable sleeplessness). A score was set to missing after a participant received prohibited/rescue medication that potentially impact efficacy analyses prior to Week 16, and the participant's worst post baseline observation before the time of the medication usage was carried forward (WOCF) to impute missing endpoint value (for participants whose postbaseline values were all missing, the baseline was used to impute). The least squares mean (LSM) and LSM difference were rounded up or down to the nearest single decimal place.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 18, 20, 32, 48, 52
Population: mITT Analysis Set: All randomized participants who receive at least 1 dose of vixarelimab or placebo and have at least 1 post-baseline efficacy assessment in the double-blind treatment period; WOCF: Baseline through Week 52.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
units on a scale
  Week 2 | -2.9 (0.40) | -2.4 (0.39) | -1.5 (0.41) | -0.1 (0.38)
  Week 4 | -3.1 (0.34) | -2.1 (0.35) | -1.3 (0.36) | -0.1 (0.33)
  Week 8 | -3.2 (0.42) | -3.0 (0.41) | -1.9 (0.41) | -1.0 (0.41)
  Week 12 | -3.6 (0.43) | -3.2 (0.43) | -1.8 (0.45) | -1.1 (0.45)
  Week 16 | -3.5 (0.43) | -3.3 (0.44) | -2.1 (0.44) | -1.5 (0.44)
  Week 18 | -3.8 (0.43) | -3.6 (0.44) | -2.4 (0.45) | -2.3 (0.47)
  Week 20 | -3.9 (0.38) | -3.8 (0.39) | -2.7 (0.39) | -3.0 (0.39)
  Week 32 | -4.1 (0.38) | -4.1 (0.40) | -3.3 (0.40) | -3.5 (0.39)
  Week 48 | -4.5 (0.40) | -4.4 (0.40) | -3.7 (0.38) | -3.7 (0.39)
  Week 52 | -4.5 (0.41) | -4.4 (0.42) | -3.8 (0.42) | -3.9 (0.41)
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p < 0.0001, ANCOVA — Estimated from ANCOVA models with treatment and randomization stratification factors of sex and years since the first nodule observed (i.e., ≥10 vs. <10 years) as fixed effect factors, baseline as covariate; LS Mean Difference = -2.7, 95% CI 2-sided [-3.8 to -1.6], Standard Error of Mean 0.55
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -2.3, 95% CI 2-sided [-3.3 to -1.2], Standard Error of Mean 0.54
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0125, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.5 to -0.3], Standard Error of Mean 0.55
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -2.9, 95% CI 2-sided [-3.8 to -2.0], Standard Error of Mean 0.47
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -2.0, 95% CI 2-sided [-2.9 to -1.0], Standard Error of Mean 0.48
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0198, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -1.1, 95% CI 2-sided [-2.1 to -0.2], Standard Error of Mean 0.48
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -2.3, 95% CI 2-sided [-3.4 to -1.2], Standard Error of Mean 0.57
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0004, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -2.0, 95% CI 2-sided [-3.2 to -0.9], Standard Error of Mean 0.57
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0969, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.1 to 0.2], Standard Error of Mean 0.57
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -2.5, 95% CI 2-sided [-3.7 to -1.3], Standard Error of Mean 0.61
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0012, ANCOVA — [p-value comment as in outcome 36, analysis 1]; ls = -2.0, 95% CI 2-sided [-3.2 to -0.8], Standard Error of Mean 0.62
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.3212, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.9 to 0.6], Standard Error of Mean 0.63
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0011, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -2.0, 95% CI 2-sided [-3.2 to -0.8], Standard Error of Mean 0.61
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0044, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -1.8, 95% CI 2-sided [-3.0 to -0.6], Standard Error of Mean 0.61
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.3635, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.8 to 0.7], Standard Error of Mean 0.62
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0172, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -1.5, 95% CI 2-sided [-2.7 to -0.3], Standard Error of Mean 0.62
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0401, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-2.6 to -0.1], Standard Error of Mean 0.63
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.7627, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.4 to 1.1], Standard Error of Mean 0.63
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0827, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-2.0 to 0.1], Standard Error of Mean 0.54
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.1315, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-1.9 to 0.3], Standard Error of Mean 0.55
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.6133, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.8 to 1.4], Standard Error of Mean 0.54
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.3136, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.6 to 0.5], Standard Error of Mean 0.54
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.3218, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.6 to 0.5], Standard Error of Mean 0.55
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.6576, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.8 to 1.3], Standard Error of Mean 0.55
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.1565, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.8, 95% CI 2-sided [-1.9 to 0.3], Standard Error of Mean 0.55
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.2280, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.7 to 0.4], Standard Error of Mean 0.55
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.9400, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = 0.0, 95% CI 2-sided [-1.0 to 1.1], Standard Error of Mean 0.54
Statistical Analysis 28: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.2760, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.8 to 0.5], Standard Error of Mean 0.57
Statistical Analysis 29: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.4096, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.6 to 0.7], Standard Error of Mean 0.58
Statistical Analysis 30: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.8177, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-1.0 to 1.3], Standard Error of Mean 0.58

37. Secondary Outcome: Phase 2b: Percent Change From Baseline in Weekly Average of Sleep Loss VAS Over Time
Description: as for outcome 36
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 18, 20, 32, 48, 52
Population: as for outcome 36
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage change
  Week 2 | -63.6 (26.46) | -24.9 (25.73) | -28.5 (27.03) | 81.4 (25.30)
  Week 4 | -50.6 (10.74) | -30.2 (11.03) | -18.1 (11.34) | 25.2 (10.53)
  Week 8 | -36.7 (15.47) | -48.2 (15.12) | -25.3 (15.39) | 5.9 (15.22)
  Week 12 | -62.4 (19.30) | -46.1 (19.73) | -26.7 (20.58) | 25.6 (20.17)
  Week 16 | -57.4 (9.75) | -46.3 (10.02) | -28.6 (10.11) | -12.3 (9.98)
  Week 18 | -55.1 (11.14) | -44.7 (11.35) | -29.0 (11.90) | -22.4 (12.24)
  Week 20 | -64.9 (9.83) | -56.8 (10.36) | -37.0 (10.39) | -27.6 (10.30)
  Week 32 | -66.4 (10.57) | -56.5 (11.17) | -41.8 (11.14) | -38.3 (10.60)
  Week 48 | -71.2 (10.88) | -67.3 (11.19) | -49.9 (10.66) | -44.0 (10.75)
  Week 52 | -67.8 (10.85) | -65.4 (11.43) | -55.0 (11.41) | -49.3 (11.03)
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -145.0, 95% CI 2-sided [-216.6 to -73.3], Standard Error of Mean 36.24
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0035, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -106.4, 95% CI 2-sided [-177.2 to -35.5], Standard Error of Mean 35.82
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 2; Test type: Superiority; p = 0.0031, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -109.9, 95% CI 2-sided [-182.2 to -37.6]
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -75.8, 95% CI 2-sided [-105.2 to -46.4], Standard Error of Mean 14.90
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0003, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -55.4, 95% CI 2-sided [-85.3 to -25.5], Standard Error of Mean 15.14
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0053, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -43.3, 95% CI 2-sided [-73.5 to -13.1], Standard Error of Mean 0.0053
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0472, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -42.6, 95% CI 2-sided [-84.6 to -0.5], Standard Error of Mean 21.28
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0115, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -54.0, 95% CI 2-sided [-95.7 to -12.3], Standard Error of Mean 21.11
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.1453, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -31.1, 95% CI 2-sided [-73.2 to 10.9], Standard Error of Mean 21.28
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0017, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -88.1, 95% CI 2-sided [-142.5 to -33.6], Standard Error of Mean 27.58
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0110, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -71.7, 95% CI 2-sided [-126.8 to -16.7], Standard Error of Mean 27.87
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0681, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -52.3, 95% CI 2-sided [-108.5 to 3.9], Standard Error of Mean 28.46
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0013, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -45.0, 95% CI 2-sided [-72.3 to -17.8], Standard Error of Mean 13.79
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0161, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -34.0, 95% CI 2-sided [-61.5 to -6.4], Standard Error of Mean 13.96
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.2466, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -16.3, 95% CI 2-sided [-44.0 to 11.4], Standard Error of Mean 14.02
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0451, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -32.7, 95% CI 2-sided [-64.6 to -0.7], Standard Error of Mean 16.17
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.1770, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -22.3, 95% CI 2-sided [-54.8 to 10.2], Standard Error of Mean 16.43
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.6893, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -6.6, 95% CI 2-sided [-39.3 to 26.1], Standard Error of Mean 16.54
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0087, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -37.3, 95% CI 2-sided [-65.0 to -9.6], Standard Error of Mean 14.02
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0439, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -29.3, 95% CI 2-sided [-57.7 to -0.8], Standard Error of Mean 14.40
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.5110, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -9.4, 95% CI 2-sided [-37.8 to 18.9], Standard Error of Mean 14.33
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.0592, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -28.1, 95% CI 2-sided [-57.2 to 1.1], Standard Error of Mean 14.76
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.2327, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -18.2, 95% CI 2-sided [-48.3 to 11.8], Standard Error of Mean 15.21
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.8173, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -3.5, 95% CI 2-sided [-33.5 to 26.4], Standard Error of Mean 15.16
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.0725, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -27.3, 95% CI 2-sided [-57.1 to 2.5], Standard Error of Mean 15.06
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.1285, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -23.3, 95% CI 2-sided [-53.5 to 6.8], Standard Error of Mean 15.25
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.6911, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -5.9, 95% CI 2-sided [-35.2 to 23.4], Standard Error of Mean 14.82
Statistical Analysis 28: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.2283, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -18.4, 95% CI 2-sided [-48.6 to 11.7], Standard Error of Mean 15.24
Statistical Analysis 29: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.3049, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -16.1, 95% CI 2-sided [-46.9 to 14.8], Standard Error of Mean 15.60
Statistical Analysis 30: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.7172, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -5.7, 95% CI 2-sided [-36.6 to 25.2], Standard Error of Mean 15.62

38. Secondary Outcome: Phase 2b: Change From Baseline in ItchyQoL Over Time
Description: as for outcome 20
Time Frame: Baseline, Weeks 4, 8, 12, 16, 18, 20, 32, 48, 52
Population: as for outcome 36
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
score on a scale
  Week 4 | -19.7 (2.19) | -13.4 (2.23) | -11.5 (2.26) | -1.7 (2.15)
  Week 8 | -26.1 (2.57) | -17.4 (2.52) | -12.1 (2.54) | -5.1 (2.54)
  Week 12 | -27.0 (2.93) | -22.7 (2.96) | -15.4 (3.09) | -6.4 (3.07)
  Week 16 | -28.8 (2.78) | -23.4 (2.83) | -18.2 (2.87) | -7.8 (2.87)
  Week 18 | -30.6 (2.93) | -27.7 (2.98) | -22.5 (3.07) | -17.9 (3.22)
  Week 20 | -31.0 (2.85) | -28.3 (2.96) | -25.1 (2.99) | -23.7 (3.00)
  Week 32 | -33.9 (3.09) | -29.4 (3.21) | -27.8 (3.22) | -26.0 (3.11)
  Week 48 | -34.8 (3.24) | -30.6 (3.27) | -27.9 (3.15) | -30.4 (3.20)
  Week 52 | -34.7 (3.22) | -34.0 (3.32) | -31.1 (3.30) | -29.8 (3.27)
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -18.0, 95% CI 2-sided [-24.1 to -12.0], Standard Error of Mean 3.05
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -11.7, 95% CI 2-sided [-17.8 to -5.6], Standard Error of Mean 3.08
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0017, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -9.9, 95% CI 2-sided [-15.9 to -3.8], Standard Error of Mean 3.08
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -21.0, 95% CI 2-sided [-28.0 to -13.9], Standard Error of Mean 3.56
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0006, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -12.3, 95% CI 2-sided [-19.3 to -5.4], Standard Error of Mean 3.52
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0497, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -7.0, 95% CI 2-sided [-13.9 to 0.0], Standard Error of Mean 3.53
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -20.6, 95% CI 2-sided [-28.9 to -12.3], Standard Error of Mean 4.20
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -16.3, 95% CI 2-sided [-24.6 to -8.0], Standard Error of Mean 4.21
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0362, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -9.1, 95% CI 2-sided [-17.5 to -0.6], Standard Error of Mean 4.29
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -21.0, 95% CI 2-sided [-28.8 to -13.2], Standard Error of Mean 3.96
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -15.6, 95% CI 2-sided [-23.5 to -7.7], Standard Error of Mean 3.98
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0100, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -10.4, 95% CI 2-sided [-18.3 to -2.5], Standard Error of Mean 4.00
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0035, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -12.7, 95% CI 2-sided [-21.1 to -4.3], Standard Error of Mean 4.27
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0255, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -9.8, 95% CI 2-sided [-18.3 to -1.2], Standard Error of Mean 4.33
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.2869, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -4.6, 95% CI 2-sided [-13.1 to 3.9], Standard Error of Mean 4.31
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0760, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -7.3, 95% CI 2-sided [-15.4 to 0.8], Standard Error of Mean 4.09
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.2673, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -4.6, 95% CI 2-sided [-12.8 to 3.6], Standard Error of Mean 4.15
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.7320, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-9.6 to 6.8], Standard Error of Mean 4.14
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.0726, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -7.9, 95% CI 2-sided [-16.4 to 0.7], Standard Error of Mean 4.34
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.4475, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -3.4, 95% CI 2-sided [-12.1 to 5.4], Standard Error of Mean 4.41
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.6854, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -1.8, 95% CI 2-sided [-10.5 to 6.9], Standard Error of Mean 4.41
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.3287, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -4.4, 95% CI 2-sided [-13.3 to 4.5], Standard Error of Mean 4.50
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.9752, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-9.0 to 8.7], Standard Error of Mean 4.49
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.5761, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = 2.5, 95% CI 2-sided [-6.2 to 11.2], Standard Error of Mean 4.40
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.2817, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -4.9, 95% CI 2-sided [-13.9 to 4.1], Standard Error of Mean 4.54
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.3554, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -4.2, 95% CI 2-sided [-13.3 to 4.8], Standard Error of Mean 4.56
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.7713, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -1.3, 95% CI 2-sided [-10.4 to 7.7], Standard Error of Mean 4.57

39. Secondary Outcome: Phase 2b: Percent Change From Baseline in ItchyQoL Over Time
Description: as for outcome 20
Time Frame: Baseline, Weeks 4, 8, 12, 16, 18, 20, 32, 48, 52
Population: as for outcome 36
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE)
Number analyzed (Participants) | 47 | 47 | 47 | 48
percentage change
  Week 4 | -25.4 (2.88) | -17.2 (2.93) | -13.8 (2.97) | -0.6 (2.83)
  Week 8 | -32.8 (3.18) | -21.8 (3.11) | -13.6 (3.14) | -5.0 (3.14)
  Week 12 | -34.0 (3.66) | -28.4 (3.70) | -17.7 (3.87) | -6.5 (3.84)
  Week 16 | -36.4 (3.45) | -29.5 (3.51) | -21.1 (3.56) | -8.3 (3.55)
  Week 18 | -39.3 (3.69) | -34.8 (3.76) | -26.7 (3.87) | -20.3 (4.06)
  Week 20 | -39.9 (3.60) | -35.8 (3.74) | -30.3 (3.77) | -28.2 (3.79)
  Week 32 | -43.5 (4.04) | -36.4 (4.20) | -33.5 (4.21) | -31.3 (4.07)
  Week 48 | -44.4 (4.16) | -38.3 (4.20) | -34.4 (4.04) | -36.2 (4.11)
  Week 52 | -44.5 (4.19) | -43.0 (4.31) | -37.7 (4.30) | -36.3 (4.26)
Statistical Analysis 1: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -24.8, 95% CI 2-sided [-32.8 to -16.9], Standard Error of Mean 4.01
Statistical Analysis 2: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -16.6, 95% CI 2-sided [-24.6 to -8.6], Standard Error of Mean 4.04
Statistical Analysis 3: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 4; Test type: Superiority; p = 0.0013, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -13.3, 95% CI 2-sided [-21.2 to -5.3], Standard Error of Mean 4.05
Statistical Analysis 4: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -27.8, 95% CI 2-sided [-36.5 to -19.1], Standard Error of Mean 4.40
Statistical Analysis 5: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -16.8, 95% CI 2-sided [-25.4 to -8.2], Standard Error of Mean 4.35
Statistical Analysis 6: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 8; Test type: Superiority; p = 0.0511, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -8.6, 95% CI 2-sided [-17.2 to 0.0], Standard Error of Mean 4.36
Statistical Analysis 7: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -27.5, 95% CI 2-sided [-37.8 to -17.1], Standard Error of Mean 5.26
Statistical Analysis 8: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -21.9, 95% CI 2-sided [-32.3 to -11.5], Standard Error of Mean 5.26
Statistical Analysis 9: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 12; Test type: Superiority; p = 0.0386, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -11.2, 95% CI 2-sided [-21.8 to -0.6], Standard Error of Mean 5.37
Statistical Analysis 10: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -28.1, 95% CI 2-sided [-37.8 to -18.4], Standard Error of Mean 4.90
Statistical Analysis 11: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -21.2, 95% CI 2-sided [-31.0 to -11.5], Standard Error of Mean 4.93
Statistical Analysis 12: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 16; Test type: Superiority; p = 0.0108, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -12.8, 95% CI 2-sided [-22.5 to -3.0], Standard Error of Mean 4.95
Statistical Analysis 13: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0006, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -19.0, 95% CI 2-sided [-29.6 to -8.4], Standard Error of Mean 5.39
Statistical Analysis 14: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.0084, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -14.6, 95% CI 2-sided [-25.3 to -3.8], Standard Error of Mean 5.45
Statistical Analysis 15: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 18; Test type: Superiority; p = 0.2422, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -6.4, 95% CI 2-sided [-17.1 to 4.4], Standard Error of Mean 5.43
Statistical Analysis 16: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.0249, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -11.7, 95% CI 2-sided [-21.9 to -1.5], Standard Error of Mean 5.17
Statistical Analysis 17: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.1497, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -7.6, 95% CI 2-sided [-17.9 to 2.8], Standard Error of Mean 5.24
Statistical Analysis 18: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 20; Test type: Superiority; p = 0.6910, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -2.1, 95% CI 2-sided [-12.4 to 8.2], Standard Error of Mean 5.23
Statistical Analysis 19: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.0331, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -12.2, 95% CI 2-sided [-23.4 to -1.0], Standard Error of Mean 5.68
Statistical Analysis 20: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.3709, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -5.2, 95% CI 2-sided [-16.6 to 6.2], Standard Error of Mean 5.77
Statistical Analysis 21: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 32; Test type: Superiority; p = 0.6924, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -2.3, 95% CI 2-sided [-13.7 to 9.1], Standard Error of Mean 5.77
Statistical Analysis 22: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.1583, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -8.2, 95% CI 2-sided [-19.6 to 3.2], Standard Error of Mean 5.78
Statistical Analysis 23: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.7193, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -2.1, 95% CI 2-sided [-13.5 to 9.3], Standard Error of Mean 5.77
Statistical Analysis 24: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 48; Test type: Superiority; p = 0.7589, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = 1.7, 95% CI 2-sided [-9.4 to 12.9], Standard Error of Mean 5.64
Statistical Analysis 25: Comparison: Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.1642, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -8.3, 95% CI 2-sided [-20.0 to 3.4], Standard Error of Mean 5.91
Statistical Analysis 26: Comparison: Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.2611, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -6.7, 95% CI 2-sided [-18.4 to 5.0], Standard Error of Mean 5.94
Statistical Analysis 27: Comparison: Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) vs Phase 2b - Placebo SC, Q4W (DBL), Then Vixarelimab (OLE); Week 52; Test type: Superiority; p = 0.8076, ANCOVA — [p-value comment as in outcome 36, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-13.2 to 10.3], Standard Error of Mean 5.94

ADVERSE EVENTS:
Time Frame: Phase 2a: From the Screening Visit through end of study (EOS) Visit (Week 24). Phase 2b: Double-blind (DBL) period: after signing the informed consent form (ICF) until Week 16; Open-label extension (OLE) period: End of Week 16 until Week 52.
Groups:
- Phase 2b - Vixarelimab 540 mg SC Q4W (DBL): Vixarelimab 540 mg SC, every 4 weeks (Q4W) for 16 weeks during the double-blind (DBL) period.
- Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL): Vixarelimab 360 mg SC, Q4W for 16 weeks during the double-blind (DBL) period.
- Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL): Vixarelimab 120 mg SC, Q4W for 16 weeks during the double-blind (DBL) period.
- Phase 2b - Placebo SC, Q4W (DBL): Placebo SC, Q4W for 16 weeks during the double-blind (DBL) period.
- Phase 2b - Vixarelimab 360 mg SC, Q2W (OLE Period): Vixarelimab 360 mg SC, every 2 weeks (Q2W) for 36 weeks during the open-label extension (OLE) period.
Arm/Group | Phase 2a - Vixarelimab 360 mg SC QW | Phase 2a - Placebo SC QW | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) | Phase 2b - Placebo SC, Q4W (DBL) | Phase 2b - Vixarelimab 360 mg SC, Q2W (OLE Period)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26 | 0/47 | 0/47 | 0/47 | 0/48 | 0/181
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26 | 3/47 | 0/47 | 1/47 | 3/48 | 8/181
Other Adverse Events (participants affected / at risk) | 17/23 | 14/26 | 18/47 | 13/47 | 10/47 | 14/48 | 77/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2a - Vixarelimab 360 mg SC QW (N=23) | Phase 2a - Placebo SC QW (N=26) | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) (N=47) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) (N=47) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) (N=47) | Phase 2b - Placebo SC, Q4W (DBL) (N=48) | Phase 2b - Vixarelimab 360 mg SC, Q2W (OLE Period) (N=181)
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal fusion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2a - Vixarelimab 360 mg SC QW (N=23) | Phase 2a - Placebo SC QW (N=26) | Phase 2b - Vixarelimab 540 mg SC Q4W (DBL) (N=47) | Phase 2b - Vixarelimab 360 mg SC, Q4W (DBL) (N=47) | Phase 2b - Vixarelimab 120 mg SC, Q4W (DBL) (N=47) | Phase 2b - Placebo SC, Q4W (DBL) (N=48) | Phase 2b - Vixarelimab 360 mg SC, Q2W (OLE Period) (N=181)
Fatigue (General disorders) | 0 | 0 | 5 | 1 | 1 | 1 | 3
COVID-19 (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 4 | 28
Nasopharyngitis (Infections and infestations) | 3 | 4 | 4 | 1 | 1 | 2 | 14
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 1 | 2 | 0 | 2 | 16
Urinary tract infection (Infections and infestations) | 0 | 4 | 1 | 0 | 1 | 0 | 6
Procedural headache (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 3 | 4 | 2 | 3 | 0 | 6
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 10
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 2 | 1 | 1 | 14
Eczema nummular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 1 | 0 | 6
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 4
Hypertension (Vascular disorders) | 1 | 1 | 2 | 0 | 2 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the first right to publish study results. PI may publish study results after Sponsor publishes the study results or 18 months after study completion at all participating sites, whichever comes first, provided that Sponsor may embargo such publication for up to 60 days for purposes of identifying confidential information that must be removed and up to an additional 60 days to prepare a patent application if there is patentable subject matter in the PI's proposed publication.

DOCUMENTS (4):
  • Study Protocol: Phase 2a Protocol (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT03816891/Prot_000.pdf
  • Study Protocol: Phase 2b Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03816891/Prot_001.pdf
  • Statistical Analysis Plan: Phase 2a SAP (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT03816891/SAP_002.pdf
  • Statistical Analysis Plan: Phase 2b SAP (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT03816891/SAP_003.pdf